CLINICAL TRIAL: NCT00005129
Title: The Bogalusa Heart Study
Brief Title: Bogalusa Heart Study
Acronym: BHS
Status: Active, not recruiting | Type: Observational
Sponsor: Tulane University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institute on Aging (NIA) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Lydia A. Bazzano, Professor, Tulane University
Other Study IDs: 908; R01AG041200 (NIH); R01HD069587 (NIH); R01ES021724 (NIH); 2R01AG016592 (NIH); R01HL121230 (NIH); R21AG057983 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Atherosclerosis; Cardiovascular Diseases; Heart Diseases; Coronary Disease; Hypertension
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Heart Diseases; Coronary Disease; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples were collected at each examination for biochemical cardiovascular risk factors, as well as genomic and DNA methylation analyses. No biospecimens are available from prior to 2005.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To determine the natural history of atherosclerosis, coronary artery disease, and hypertension in children and adults from birth through mid-life in a total biracial community.

DETAILED DESCRIPTION:
BACKGROUND:

The Bogalusa Heart Study has been a long-term epidemiologic study. The investigators have identified and followed black and white participants for nearly 40 years, and have described the incidence and prevalence of biologic and behavioral cardiovascular disease risk factors from childhood through adulthood. Their participation has enabled the study to not only document differences between males and females, but also between blacks and whites. The results from the Bogalusa Heart Study have clearly documented that the genesis of atherosclerosis has its basis in childhood, and that prevention can and must begin at the early ages.

The Bogalusa Heart Study had been funded over the years by the Specialized Centers of Research (SCOR) Program. The SCOR program was initiated by NHLBI in 1970 to expedite the development and application of new knowledge essential for improved diagnosis, treatment, and prevention of arteriosclerosis, hypertension, pulmonary disease, and thrombosis. In 1984 a Demonstration and Education Component was added to the parent SCOR of the Bogalusa Heart Study in order to translate the experience gained in epidemiological studies into an intervention study designed to retard the development of cardiovascular risk factors in children. Beginning in 1987, the Bogalusa Heart Study was supported by a regular research grant. Beginning in 1997, the study is supported by the cooperative agreement mechanism.

DESIGN :

The initial survey in 1973-1974 was restricted to children ages 2 1/2 to 14. A physical examination was conducted and information was collected on anthropometric data, hemoglobin, blood pressure, serum lipids, and health history. Over 3,500 children participated. The second cross-sectional survey of 1976-1977 and subsequent surveys expanded the eligible population to include all children ages 5-17 years. The second survey of over 4,000 children also included information on salt intake, smoking, health beliefs, and attitudes, and for girls ages 8-17, menstrual history and oral contraceptive use. The third survey of over 3,500 participants in 1978-1979 also collected anthropometric measurements on skinfold thickness and two measurements of heart rate. The fourth survey of over 3,300 participants in 1981-1982 added data on alcohol use, Type A behavior, peer networks and dieting habits.

The Bogalusa Heart Study continued to use a cross-sectional and longitudinal design with the general cross-sectional survey of approximately 3,700 Bogalusa children ages five to seventeen in 1988-1989 in the sixth screen and additional longitudinal studies to recall children in defined subgroups for more intensive evaluation. Half of the 12,000 participants screened since 1973 had been studied three or more times. There were several other cohort groups and studies. The Newborn-Infant Cohort Study was designed to describe distributions, inter-relationships, and trends through time for blood pressure, serum lipid and lipoprotein concentrations, dietary intake patterns, and anthropometric measurements. Four hundred and forty infants born between January 1, 1974 through June 30, 1975 were examined at birth, at six months, and yearly at ages one through four and at seven, ten and thirteen years for cardiovascular risk factor variables. The Post High School Study examined young adults ages 21 through 30 who previously were examined as children ages five through fourteen in the first Bogalusa Heart Study screening in 1973-1974. The population included approximately 4,603 young adults originally screened and any other children or adolescents examined for the first time in any subsequent surveys.

The fifth screening began in 1988 and extended through December 1991. The Pediatric Pathology Risk Factor Program, which began in 1978, documented the relationship of cardiovascular disease risk factors to anatomic and pathologic changes. A local information system was established to obtain family or coroner's consent to autopsy any deceased resident between the ages of three and 26 in the Bogalusa area. Autopsy specimens were collected from over 100 deceased children and young adults, of whom approximately forty percent had been previously examined in the Bogalusa Heart Study.

Major activity during 1988-1991 involved 24-hour dietary recall collections on all the 1963, 1966, and 1968 birth cohorts attending the Post High School Study. A food frequency questionnaire was also self-administered to all the Post High School Study participants. The use of these two dietary methodologies, 24-hour dietary recall and food frequency questionnaire, provided data to assess the nutrient composition of diets of young adults, assess the weekly consumption of individual foods, compare nutrient composition data with food frequency data, and compare dietary intakes at the post high school age with those of school age. Several substudies were conducted using the Bogalusa Heart Study population. Among them were the impact of childhood obesity on risk factors, the relationship of apolipoproteins A-I and B in children to parental myocardial infarction and the relationship between left ventricular size as demonstrated by echocardiography and blood pressure distribution.

The study was renewed in Fiscal Year 1992 in order to follow-up the previously examined young adults for development of abnormal levels of cardiovascular risk factors and even clinical disease.

In 1997, the study was renewed and extended through 2002, and from 2002-2010, and again in 2012 in order to study the impact of genetic factors on the evolution from childhood cardiovascular risk factors to subclinical and clinical morbidity in an adult population, ages 20 to 43, who had been followed over a long period of time. The study also seeks to study the association of risk factor phenotypes to anatomic changes in the cardiovascular system as seen by necropsy. The population for genotype-phenotype studies includes approximately 1,400 siblings derived from longitudinal birth cohorts.

The cardiovascular phenotypes include obesity, blood pressure, lipids, lipoproteins, apoproteins, homocysteine, glucose-insulin, fibrinogen, plasminogen activator inhibitor-1 and von Willebrand Factor. Environmental risk factors consist of sociodemographic characteristics, tobacco and alcohol use, oral contraception, physical activity, cognitive and physical function, and quality of sleep and diet. Subclinical morbidity includes echo-Doppler measurements of cardiac-carotid structure and function. Using robust sibling pair linkage methods, a genome-wide search involving 391 markers with spacing of 10 centimorgans is conducted for genes which influence quantitative traits. This is supplemented with 41 highly polymorphic markers located in or near candidate genes likely to be related to obesity, lipoprotein metabolism, blood pressure, insulin resistance, diabetes, atherogenesis and thrombosis.

Approximately 75 percent of the dollars of a Specialized Center of Research (SCOR) in Arteriosclerosis (P50HL14103) were used to support the Bogalusa Heart Study from 1972 through 1986.

Since 2002, the study has been supported by the National Institute on Aging (NIA), the National Heart, Lung, and Blood Institute (NHLBI), the National Institute of Environmental Health Sciences (NIEHS), and the National Institute of Child Health and Human Development (NICHD).

ELIGIBILITY:
Index individuals were identified as those living in Bogalusa, Louisiana between 1972 and 2000 who attended Bogalusa City Schools in childhood. The families of index individuals were eligible to participate in certain sub-studies e.g. sibling and parent studies. After 2000, only previously examined individuals and, in limited circumstances, their offspring, were eligible for participation in on-going follow-up of heart disease risk factors and related outcomes.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 12,000 individuals have ever been examined at least once. Approximately 6,000 have more than one examination constituting a dynamic cohort. Between 2014 and 2019, 3,550 were contacted for CV events follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 11737 (Actual)
Dates: Start 1973-08 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2029-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Lydia Bazzano, MD, PhD, MPH, Principal Investigator — Tulane University; Wei Chen, MD, PhD, Principal Investigator — Tulane University; Emily Harville, PhD, Principal Investigator — Tulane University; Tanika Kelly, PhD, Principal Investigator — Tulane Universtiy
Locations (1):
- Tulane University, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Biolink

REFERENCES:
- [Background] Donker GA, Labarthe DR, Harrist RB, Selwyn BJ, Srinivasan SR, Wattigney W, Berenson GS. Low birth weight and serum lipid concentrations at age 7-11 years in a biracial sample. Am J Epidemiol. 1997 Mar 1;145(5):398-407. doi: 10.1093/oxfordjournals.aje.a009121. PMID 9048513
- [Background] Greenlund KJ, Johnson C, Wattigney W, Bao W, Webber LS, Berenson GS. Trends in cigarette smoking among children in a southern community, 1976-1994: the Bogalusa Heart Study. Ann Epidemiol. 1996 Nov;6(6):476-82. doi: 10.1016/s1047-2797(96)00069-5. PMID 8978877
- [Background] Farber HJ, Wattigney W, Berenson G. Trends in asthma prevalence: the Bogalusa Heart Study. Ann Allergy Asthma Immunol. 1997 Mar;78(3):265-9. doi: 10.1016/S1081-1206(10)63179-1. PMID 9087150
- [Background] Greenlund KJ, Valdez R, Bao W, Wattigney WA, Srinivasan SR, Berenson GS. Verification of parental history of coronary artery disease and associations with adult offspring risk factors in a community sample: the Bogalusa Heart Study. Am J Med Sci. 1997 Apr;313(4):220-7. doi: 10.1097/00000441-199704000-00005. PMID 9099152
- [Background] Madhavan M, Wattigney WA, Srinivasan SR, Berenson GS. Serum bilirubin distribution and its relation to cardiovascular risk in children and young adults. Atherosclerosis. 1997 May;131(1):107-13. doi: 10.1016/s0021-9150(97)06088-7. PMID 9180251
- [Background] Jiang X, Srinivasan SR, Dalferes ER Jr, Berenson GS. Plasma insulin-like growth factor 1 distribution and its relation to blood pressure in adolescents: the Bogalusa Heart Study. Am J Hypertens. 1997 Jul;10(7 Pt 1):714-9. doi: 10.1016/s0895-7061(97)00065-4. PMID 9234824
- [Background] Chen W, Srinivasan SR, Bao W, Wattigney WA, Berenson GS. The relationship of conjoint traits of dyslipidemias between young offspring and their parents in a community-based sample. Prev Med. 1997 Sep-Oct;26(5 Pt 1):717-23. doi: 10.1006/pmed.1997.0197. PMID 9327482
- [Background] Bao W, Srinivasan SR, Valdez R, Greenlund KJ, Wattigney WA, Berenson GS. Longitudinal changes in cardiovascular risk from childhood to young adulthood in offspring of parents with coronary artery disease: the Bogalusa Heart Study. JAMA. 1997 Dec 3;278(21):1749-54. PMID 9388151
- [Background] Greenlund KJ, Webber LS, Srinivasan S, Wattigney W, Johnson C, Berenson GS. Associations of oral contraceptive use with serum lipids and lipoproteins in young women: the Bogalusa Heart Study. Ann Epidemiol. 1997 Nov;7(8):561-7. doi: 10.1016/s1047-2797(97)00119-1. PMID 9408552
- [Background] Chen W, Srinivasan SR, Bao W, Wattigney WA, Berenson GS. Sibling aggregation of low- and high-density lipoprotein cholesterol and apolipoproteins B and A-I levels in black and white children: the Bogalusa Heart Study. Ethn Dis. 1997 Autumn;7(3):241-9. PMID 9467707
- [Background] Berenson GS. The control of hypertension in African-American children: the Bogalusa Heart Study. J Natl Med Assoc. 1995 Aug;87(8 Suppl):614-7. No abstract available. PMID 7674355
- [Background] Myers L, Coughlin SS, Webber LS, Srinivasan SR, Berenson GS. Prediction of adult cardiovascular multifactorial risk status from childhood risk factor levels. The Bogalusa Heart Study. Am J Epidemiol. 1995 Nov 1;142(9):918-24. doi: 10.1093/oxfordjournals.aje.a117739. PMID 7572972
- [Background] Nicklas TA. Dietary studies of children and young adults (1973-1988): the Bogalusa Heart Study. Am J Med Sci. 1995 Dec;310 Suppl 1:S101-8. doi: 10.1097/00000441-199512000-00018. PMID 7503111
- [Background] Bronfin DR, Urbina EM. The role of the pediatrician in the promotion of cardiovascular health. Am J Med Sci. 1995 Dec;310 Suppl 1:S42-7. doi: 10.1097/00000441-199512000-00008. PMID 7503123
- [Background] Spencer HC. Perspectives of public health and prevention. Am J Med Sci. 1995 Dec;310 Suppl 1:S83-5. doi: 10.1097/00000441-199512000-00015. PMID 7503131
- [Background] Hammond IW, Urbina EM, Wattigney WA, Bao W, Steinmann WC, Berenson GS. Comparison of fourth and fifth Korotkoff diastolic blood pressures in 5 to 30 year old individuals. The Bogalusa Heart Study. Am J Hypertens. 1995 Nov;8(11):1083-9. doi: 10.1016/0895-7061(95)00230-M. PMID 8554731
- [Background] Nicklas TA, Myers L, Berenson GS. Total nutrient intake and ready-to-eat cereal consumption of children and young adults in the Bogalusa Heart Study. Nutr Rev. 1995 Sep;53(9 Pt 2):S39-45. No abstract available. PMID 8577417
- [Background] Jiang X, Srinivasan SR, Radhakrishnamurthy B, Dalferes ER, Berenson GS. Racial (black-white) differences in insulin secretion and clearance in adolescents: the Bogalusa heart study. Pediatrics. 1996 Mar;97(3):357-60. PMID 8604270
- [Background] Wattigney WA, Webber LS, Srinivasan SR, Berenson GS. The emergence of clinically abnormal levels of cardiovascular disease risk factor variables among young adults: the Bogalusa Heart Study. Prev Med. 1995 Nov;24(6):617-26. doi: 10.1006/pmed.1995.1097. PMID 8610086
- [Background] Wattigney WA, Webber LS, Lawrence MD, Berenson GS. Utility of an automatic instrument for blood pressure measurement in children. The Bogalusa Heart Study. Am J Hypertens. 1996 Mar;9(3):256-62. doi: 10.1016/0895-7061(95)00334-7. PMID 8695025
- [Background] Nicklas TA. Dietary studies of children: the Bogalusa Heart Study experience. J Am Diet Assoc. 1995 Oct;95(10):1127-33. doi: 10.1016/S0002-8223(95)00305-3. PMID 7560684
- [Background] Nicklas TA, Myers L, Farris RP, Srinivasan SR, Berenson GS. Nutritional quality of a high carbohydrate diet as consumed by children: The Bogalusa Heart Study. J Nutr. 1996 May;126(5):1382-8. doi: 10.1093/jn/126.5.1382. PMID 8618134
- [Background] Zive MM, Nicklas TA, Busch EC, Myers L, Berenson GS. Marginal vitamin and mineral intakes of young adults: the Bogalusa Heart Study. J Adolesc Health. 1996 Jul;19(1):39-47. doi: 10.1016/1054-139X(96)00022-5. PMID 8842859
- [Background] Myers L, Strikmiller PK, Webber LS, Berenson GS. Physical and sedentary activity in school children grades 5-8: the Bogalusa Heart Study. Med Sci Sports Exerc. 1996 Jul;28(7):852-9. doi: 10.1097/00005768-199607000-00012. PMID 8832539
- [Background] Berenson GS, Wattigney WA, Webber LS. Epidemiology of hypertension from childhood to young adulthood in black, white, and Hispanic population samples. Public Health Rep. 1996;111 Suppl 2(Suppl 2):3-6. PMID 8898760
- [Background] Freedman DS, Srinivasan SR, Valdez RA, Williamson DF, Berenson GS. Secular increases in relative weight and adiposity among children over two decades: the Bogalusa Heart Study. Pediatrics. 1997 Mar;99(3):420-6. doi: 10.1542/peds.99.3.420. PMID 9041299
- [Background] Srinivasan SR, Ehnholm C, Wattigney WA, Berenson GS. Influence of apolipoprotein E polymorphism on the tracking of childhood levels of serum lipids and apolipoproteins over a 6-year period. The Bogalusa Heart Study. Atherosclerosis. 1996 Nov 15;127(1):73-9. doi: 10.1016/s0021-9150(96)05937-0. PMID 9006807
- [Background] Berenson GS, Srinivasan SR, Bao W. Precursors of cardiovascular risk in young adults from a biracial (black-white) population: the Bogalusa Heart Study. Ann N Y Acad Sci. 1997 May 28;817:189-98. doi: 10.1111/j.1749-6632.1997.tb48206.x. PMID 9239188
- [Background] Greenlund KJ, Johnson CC, Webber LS, Berenson GS. Cigarette smoking attitudes and first use among third- through sixth-grade students: the Bogalusa Heart Study. Am J Public Health. 1997 Aug;87(8):1345-8. doi: 10.2105/ajph.87.8.1345. PMID 9279273
- [Background] Burke GL, Freedman DS, Webber LS, Berenson GS. Persistence of high diastolic blood pressure in thin children. The Bogalusa Heart Study. Hypertension. 1986 Jan;8(1):24-9. doi: 10.1161/01.hyp.8.1.24. PMID 3484724
- [Background] Parker FC, Croft JB, Supik JD, Webber LS, Hunter SM, Berenson GS. Factors associated with adolescent participation in a cardiovascular risk factor assessment program. J Sch Health. 1986 Jan;56(1):23-8. doi: 10.1111/j.1746-1561.1986.tb05677.x. PMID 3633357
- [Background] Croft JB, Foster TA, Parker FC, Cresanta JL, Hunter SM, Webber LS, Srinivasan SR, Berenson GS. Transitions of cardiovascular risk from adolescence to young adulthood--the Bogalusa Heart Study: I. Effects of alterations in lifestyle. J Chronic Dis. 1986;39(2):81-90. doi: 10.1016/0021-9681(86)90064-0. PMID 3944230
- [Background] Webber LS, Cresanta JL, Croft JB, Srinivasan SR, Berenson GS. Transitions of cardiovascular risk from adolescence to young adulthood--the Bogalusa Heart Study: II. Alterations in anthropometric blood pressure and serum lipoprotein variables. J Chronic Dis. 1986;39(2):91-103. doi: 10.1016/0021-9681(86)90065-2. PMID 3944231
- [Background] Shear CL, Webber LS, Freedman DS, Srinivasan SR, Berenson GS. The relationship between parental history of vascular disease and cardiovascular disease risk factors in children: the Bogalusa Heart Study. Am J Epidemiol. 1985 Nov;122(5):762-71. doi: 10.1093/oxfordjournals.aje.a114159. PMID 3876762
- [Background] Burke GL, Cresanta JL, Shear CL, Miner MH, Berenson GS. Cardiovascular risk factors and their modification in children. Cardiol Clin. 1986 Feb;4(1):33-46. PMID 3518933
- [Background] Hunter SM, Croft JB, Burke GL, Parker FC, Webber LS, Berenson GS. Longitudinal patterns of cigarette smoking and smokeless tobacco use in youth: the Bogalusa Heart Study. Am J Public Health. 1986 Feb;76(2):193-5. doi: 10.2105/ajph.76.2.193. PMID 3484908
- [Background] Burke GL, Webber LS, Srinivasan SR, Radhakrishnamurthy B, Freedman DS, Berenson GS. Fasting plasma glucose and insulin levels and their relationship to cardiovascular risk factors in children: Bogalusa Heart Study. Metabolism. 1986 May;35(5):441-6. doi: 10.1016/0026-0495(86)90135-6. PMID 3517558
- [Background] Srinivasan SR, Amos C, Albares R, Bhandaru RR, Dalferes ER Jr, Webber LS, Berenson GS. Influence of serum lipoproteins and carbohydrate metabolism on erythrocyte membrane composition in children: Bogalusa Heart Study. Metabolism. 1986 May;35(5):466-71. doi: 10.1016/0026-0495(86)90139-3. PMID 3517559
- [Background] Farris RP, Cresanta JL, Croft JB, Webber LS, Frank GC, Berenson GS. Macronutrient intakes of 10-year-old children, 1973 to 1982. J Am Diet Assoc. 1986 Jun;86(6):765-70. PMID 3711557
- [Background] Freedman DS, Srinivasan SR, Shear CL, Hunter SM, Croft JB, Webber LS, Berenson GS. Cigarette smoking initiation and longitudinal changes in serum lipids and lipoproteins in early adulthood: the Bogalusa Heart Study. Am J Epidemiol. 1986 Aug;124(2):207-19. doi: 10.1093/oxfordjournals.aje.a114379. PMID 3728437
- [Background] Hunter SM, Croft JB, Burke GL, Vizelberg IA, Berenson GS: Social Influences and Longitudinal Patterns of Smokeless Tobacco Use. In: Health Implications of Smokeless Tobacco, NIH Consensus Development Conference, January 13-15, p. 32-37, 1986
- [Background] Cresanta JL, Burke GL, Downey AM, Freedman DS, Berenson GS. Prevention of atherosclerosis in childhood. Pediatr Clin North Am. 1986 Aug;33(4):835-58. doi: 10.1016/s0031-3955(16)36076-x. PMID 3737258
- [Background] Shear CL, Burke GL, Freedman DS, Berenson GS. Value of childhood blood pressure measurements and family history in predicting future blood pressure status: results from 8 years of follow-up in the Bogalusa Heart Study. Pediatrics. 1986 Jun;77(6):862-9. PMID 3714379
- [Background] Srinivasan SR, Freedman DS, Sharma C, Webber LS, Berenson GS. Serum apolipoproteins A-I and B in 2,854 children from a biracial community: Bogalusa Heart Study. Pediatrics. 1986 Aug;78(2):189-200. PMID 3090510
- [Background] Freedman DS, Newman WP III, Gard PD, Cresanta JL, Srinivasan SR, Tracy RE, Berenson GS: Atherosclerosis in Early Life - The Bogalusa Heart Study. Cardiol Board Rev, 3:26-40, 1986
- [Background] Amos CI, Wilson AF, Rosenbaum PA, Srinivasan SR, Webber LS, Elston RC, Berenson GS. An approach to the multivariate analysis of high-density-lipoprotein cholesterol in a large kindred: the Bogalusa Heart Study. Genet Epidemiol. 1986;3(4):255-67. doi: 10.1002/gepi.1370030406. PMID 3744022
- [Background] Rosenbaum PA, Amos CI, Shear CL, Elston RC, Sellers TA, Srinivasan SR, Berenson GS. Description of a large pedigree with an adverse lipoprotein cholesterol phenotype: the Bogalusa Heart Study. Genet Epidemiol. 1986;3(4):241-53. doi: 10.1002/gepi.1370030405. PMID 3744021
- [Background] Cohen JC, Buonagura K, Bickers J, Berenson GS, Rothschild H: Familial Clustering of Malignancies: Distribution of Ha-ras Restriction Fragment Length Polymorphisms in Normal and High Risk Populations. In: Proceedings of UCLA Symposia on Molecular and Cellular Biology, Vol 40 (Harris CC, Eds). New York: Alan R. Liss, Inc, p. 397-400, 1986
- [Background] Riley WA, Freedman DS, Higgs NA, Barnes RW, Zinkgraf SA, Berenson GS. Decreased arterial elasticity associated with cardiovascular disease risk factors in the young. Bogalusa Heart Study. Arteriosclerosis. 1986 Jul-Aug;6(4):378-86. doi: 10.1161/01.atv.6.4.378. PMID 3524521
- [Background] Srinivasan SR, Freedman DS, Sundaram GS, Webber LS, Berenson GS. Racial (black-white) comparisons of the relationship of levels of endogenous sex hormones to serum lipoproteins during male adolescence: the Bogalusa Heart Study. Circulation. 1986 Dec;74(6):1226-34. doi: 10.1161/01.cir.74.6.1226. PMID 2946492
- [Background] Webber LS, Cresanta JL, Voors AW, Berenson GS. Tracking of cardiovascular disease risk factor variables in school-age children. J Chronic Dis. 1983;36(9):647-60. doi: 10.1016/0021-9681(83)90081-4. PMID 6619260
- [Background] Webber LS, Freedman DS: Interrelationships of Coronary Heart Disease Risk Factors in Children. In: Causation of Cardiovascular Risk Factors in Children (Berenson GS, Ed). New York: Raven Press, 1986
- [Background] Freedman DS, Srinivasan SR, Shear CL, Franklin FA, Webber LS, Berenson GS. The relation of apolipoproteins A-I and B in children to parental myocardial infarction. N Engl J Med. 1986 Sep 18;315(12):721-6. doi: 10.1056/NEJM198609183151202. PMID 3092050
- [Background] Tracy RE, Mercante DE, Moncada A, Berenson G. Quantitation of hypertensive nephrosclerosis on an objective rational scale of measure in adults and children. Am J Clin Pathol. 1986 Mar;85(3):312-8. doi: 10.1093/ajcp/85.3.312. PMID 3751980
- [Background] Fox MH, Webber LS, Thurmon TF, Berenson GS. ABO blood group associations with cardiovascular risk factor variables. II. Blood pressure, obesity, and their anthropometric covariables. The Bogalusa Heart Study. Hum Biol. 1986 Aug;58(4):549-84. No abstract available. PMID 3759056
- [Background] Amos CI, Hunter SM, Zinkgraf SA, Miner MH, Berenson GS. Characterization of a comprehensive type A measure for children in a biracial community: the Bogalusa Heart Study. J Behav Med. 1987 Oct;10(5):425-39. doi: 10.1007/BF00846142. PMID 3430586
- [Background] Burke GL, Webber LS, Shear CL, Zinkgraf SA, Smoak CG, Berenson GS. Sources of error in measurement of children's blood pressure in a large epidemiologic study: Bogalusa Heart Study. J Chronic Dis. 1987;40(1):83-9. doi: 10.1016/0021-9681(87)90099-3. PMID 3805236
- [Background] Foster TA, Berenson GS. Measurement error and reliability in four pediatric cross-sectional surveys of cardiovascular disease risk factor variables--the Bogalusa Heart Study. J Chronic Dis. 1987;40(1):13-21. doi: 10.1016/0021-9681(87)90092-0. PMID 3492509
- [Background] Shear CL, Burke GL, Freedman DS, Webber LS, Berenson GS. Designation of children with high blood pressure--considerations on percentile cut points and subsequent high blood pressure: the Bogalusa Heart Study. Am J Epidemiol. 1987 Jan;125(1):73-84. doi: 10.1093/oxfordjournals.aje.a114513. PMID 3788956
- [Background] Parker FC, Croft JB, Cresanta JL, Freedman DS, Burke GL, Webber LS, Berenson GS. The association between cardiovascular response tasks and future blood pressure levels in children: Bogalusa Heart Study. Am Heart J. 1987 May;113(5):1174-9. doi: 10.1016/0002-8703(87)90931-8. PMID 3495163
- [Background] Berenson GS, Srinivasan SR, Freedman DS, Radhakrishnamurthy B, Dalferes ER Jr. Atherosclerosis and its evolution in childhood. Am J Med Sci. 1987 Dec;294(6):429-40. doi: 10.1097/00000441-198712000-00008. PMID 3321985
- [Background] Cresanta JL, Croft JB, Webber LS, Nicklas TA, Berenson GS. Racial difference in hemoglobin concentration of young adults. Prev Med. 1987 Sep;16(5):659-69. doi: 10.1016/0091-7435(87)90049-1. PMID 3500469
- [Background] Rosenbaum PA, Elston RC, Srinivasan SR, Webber LS, Berenson GS. Cardiovascular risk factors from birth to 7 years of age: the Bogalusa Heart Study. Predictive value of parental measures in determining cardiovascular risk factor variables in early life. Pediatrics. 1987 Nov;80(5 Pt 2):807-16. PMID 3670991
- [Background] Nicklas TA, Farris RP, Major C, Frank GC, Webber LS, Cresanta JL, Berenson GS. Cardiovascular risk factors from birth to 7 years of age: the Bogalusa Heart Study. Dietary intakes. Pediatrics. 1987 Nov;80(5 Pt 2):797-806. PMID 3670990
- [Background] Freedman DS, Srinivasan SR, Cresanta JL, Webber LS, Berenson GS. Cardiovascular risk factors from birth to 7 years of age: the Bogalusa Heart Study. Serum lipids and lipoproteins. Pediatrics. 1987 Nov;80(5 Pt 2):789-96. PMID 3478647
- [Background] Burke GL, Voors AW, Shear CL, Webber LS, Smoak CG, Cresanta JL, Berenson GS. Cardiovascular risk factors from birth to 7 years of age: the Bogalusa Heart Study. Blood pressure. Pediatrics. 1987 Nov;80(5 Pt 2):784-8. PMID 3670989
- [Background] Harsha DW, Smoak CG, Nicklas TA, Webber LS, Berenson GS. Cardiovascular risk factors from birth to 7 years of age: the Bogalusa Heart Study. Tracking of body composition variables. Pediatrics. 1987 Nov;80(5 Pt 2):779-83. PMID 3670988
- [Background] Webber LS, Frank GC, Smoak CG, Freedman DS, Berenson GS. Cardiovascular risk factors from birth to 7 years of age: the Bogalusa Heart Study. Design and participation. Pediatrics. 1987 Nov;80(5 Pt 2):767-78. PMID 3670987
- [Background] Amos CI, Elston RC, Srinivasan SR, Wilson AF, Cresanta JL, Ward LJ, Berenson GS. Linkage and segregation analyses of apolipoproteins A1 and B, and lipoprotein cholesterol levels in a large pedigree with excess coronary heart disease: the Bogalusa Heart Study. Genet Epidemiol. 1987;4(2):115-28. doi: 10.1002/gepi.1370040206. PMID 3108069
- [Background] Freedman DS, Shear CL, Burke GL, Srinivasan SR, Webber LS, Harsha DW, Berenson GS. Persistence of juvenile-onset obesity over eight years: the Bogalusa Heart Study. Am J Public Health. 1987 May;77(5):588-92. doi: 10.2105/ajph.77.5.588. PMID 3565653
- [Background] Shear CL, Freedman DS, Burke GL, Harsha DW, Berenson GS. Body fat patterning and blood pressure in children and young adults. The Bogalusa Heart Study. Hypertension. 1987 Mar;9(3):236-44. doi: 10.1161/01.hyp.9.3.236. PMID 3818021
- [Background] Smoak CG, Burke GL, Webber LS, Harsha DW, Srinivasan SR, Berenson GS. Relation of obesity to clustering of cardiovascular disease risk factors in children and young adults. The Bogalusa Heart Study. Am J Epidemiol. 1987 Mar;125(3):364-72. doi: 10.1093/oxfordjournals.aje.a114543. PMID 3544817
- [Background] Srinivasan SR, Freedman DS, Webber LS, Berenson GS. Black-white differences in cholesterol levels of serum high-density lipoprotein subclasses among children: the Bogalusa Heart Study. Circulation. 1987 Aug;76(2):272-9. doi: 10.1161/01.cir.76.2.272. PMID 3608116
- [Background] Freedman DS, Srinivasan SR, Shear CL, Webber LS, Chiang YK, Berenson GS. Correlates of high density lipoprotein cholesterol and apolipoprotein A-I levels in children. The Bogalusa Heart Study. Arteriosclerosis. 1987 Jul-Aug;7(4):354-60. doi: 10.1161/01.atv.7.4.354. PMID 3300617
- [Background] Freedman DS, Srinivasan SR, Webber LS, Berenson GS. Divergent levels of high density lipoprotein cholesterol and apolipoprotein A-I in children. The Bogalusa Heart Study. Arteriosclerosis. 1987 Jul-Aug;7(4):347-53. doi: 10.1161/01.atv.7.4.347. PMID 3606462
- [Background] Croft JB, Freedman DS, Cresanta JL, Srinivasan SR, Burke GL, Hunter SM, Webber LS, Smoak CG, Berenson GS. Adverse influences of alcohol, tobacco, and oral contraceptive use on cardiovascular risk factors during transition to adulthood. Am J Epidemiol. 1987 Aug;126(2):202-13. doi: 10.1093/aje/126.2.202. PMID 3605049
- [Background] George VT, Elston RC, Amos CI, Ward LJ, Berenson GS. Association between polymorphic blood markers and risk factors for cardiovascular disease in a large pedigree. Genet Epidemiol. 1987;4(4):267-75. doi: 10.1002/gepi.1370040405. PMID 3478281
- [Background] Hunter SM, Croft JB, Vizelberg IA, Berenson GS; Centers for Disease Control (CDC). Psychosocial influences on cigarette smoking among youth in a southern community: the Bogalusa Heart Study. MMWR Suppl. 1987 Sep 4;36(4):17S-23S. No abstract available. PMID 3116392
- [Background] Nicklas TA, Frank GC, Webber LS, Zinkgraf SA, Cresanta JL, Gatewood LC, Berenson GS. Racial contrasts in hemoglobin levels and dietary patterns related to hematopoiesis in children: the Bogalusa Heart Study. Am J Public Health. 1987 Oct;77(10):1320-3. doi: 10.2105/ajph.77.10.1320. PMID 3631367
- [Background] Freedman DS, Srinivasan SR, Burke GL, Shear CL, Smoak CG, Harsha DW, Webber LS, Berenson GS. Relation of body fat distribution to hyperinsulinemia in children and adolescents: the Bogalusa Heart Study. Am J Clin Nutr. 1987 Sep;46(3):403-10. doi: 10.1093/ajcn/46.3.403. PMID 3307372
- [Background] Burke GL, Arcilla RA, Culpepper WS, Webber LS, Chiang YK, Berenson GS. Blood pressure and echocardiographic measures in children: the Bogalusa Heart Study. Circulation. 1987 Jan;75(1):106-14. doi: 10.1161/01.cir.75.1.106. PMID 2947739
- [Background] Freedman DS, Srinivasan SR, Webber LS, Burke GL, Berenson GS. Black-white differences in serum lipoproteins during sexual maturation: the Bogalusa Heart Study. J Chronic Dis. 1987;40(4):309-18. doi: 10.1016/0021-9681(87)90046-4. PMID 3558707
- [Background] Freedman DS, Srinivasan SR, Shear CL, Franklin FA, Webber LS, Berenson GS: Apolipoproteins A-I and B in Relation to Parental Myocardial Infarction - The Bogalusa Heart Study. Cardiol Board Rev, March:1-24, 1987
- [Background] Johnson CC, Nicklas TA, Arbeit ML, Franklin FA, Cresanta JL, Harsha DW, Berenson GS. Cardiovascular risk in parents of children with elevated blood pressure. "Heart Smart"--family health promotion. J Clin Hypertens. 1987 Dec;3(4):559-66. PMID 3453389
- [Background] Manning DT, Balson PM, Hunter SM, Berenson GS, Willis AS. Comparison of the prevalence of type A behavior in boys and girls from two contrasting socioeconomic status groups. J Human Stress. 1987 Fall;13(3):116-20. doi: 10.1080/0097840X.1987.9936803. PMID 3655358
- [Background] Berenson GS, Srinivasan SR, Shear CL, Webber LS: The Epidemiology of Coronary Artery Disease in Childhood. In: Cardiovascular Risk Factors in Childhood: Epidemiology and Prevention (Hetzel BS, Berenson GS, Eds). Amsterdam: Elsevier Science Publishers, B.V., p. 3-20, 1987
- [Background] Freedman DS, Newman WP III, Tracy RE, Strong JP, Cresanta JL, Berenson GS: Pathology of Atherosclerosis in Childhood. In: Cardiovascular Risk Factors in Childhood: Epidemiology and Prevention (Hetzel BS, Berenson GS, Eds). Amsterdam: Elsevier Science Publishers, B.V., p. 83-99, 1987
- [Background] Asamoah A, Wilson AF, Elston RC, Dalferes E Jr, Berenson GS. Segregation and linkage analyses of dopamine-beta-hydroxylase activity in a six-generation pedigree. Am J Med Genet. 1987 Jul;27(3):613-21. doi: 10.1002/ajmg.1320270314. PMID 3631133
- [Background] Downey AM, Frank GC, Webber LS, Harsha DW, Virgilio SJ, Franklin FA, Berenson GS. Implementation of "Heart Smart:" a cardiovascular school health promotion program. J Sch Health. 1987 Mar;57(3):98-104. doi: 10.1111/j.1746-1561.1987.tb05378.x. PMID 3645182
- [Background] Thompson B, Butcher AH, Berenson GS: Children's Beliefs About Sources of Health: A Reliability and Validity Study. Measure Eval Guid Develop, 20(20:80-88, 1987
- [Background] Nicklas TA, Arbeit ML, Franklin FA, Johnson CC, Berenson GS: A Family Approach to Cardiovascular Risk Reduction Through Diet. J Nutr Educ GEM, 19:302A, 1987
- [Background] Srinivasan SR, Freedman DS, Berenson GA: Are Plasma Apolipoproteins Helpful as Markers of Coronary Artery Disease? Int Med, 8:195-201, 1987
- [Background] Butcher AH, Frank GC, Harsha DW, Serpas DC, Little SD, Nicklas TA, Hunter SM, Berenson GS. Heart Smart: a school health program meeting the 1990 Objectives for the Nation. Health Educ Q. 1988 Spring;15(1):17-34. doi: 10.1177/109019818801500103. PMID 3366584
- [Background] Croft JB, Cresanta JL, Webber LS, Srinivasan SR, Freedman DS, Burke GL, Berenson GS. Cardiovascular risk in parents of children with extreme lipoprotein cholesterol levels: the Bogalusa Heart Study. South Med J. 1988 Mar;81(3):341-9, 353. doi: 10.1097/00007611-198803000-00014. PMID 3279532
- [Background] Arbeit ML, Nicklas TA, Frank GC, Webber LS, Miner MH, Berenson GS. Caffeine intakes of children from a biracial population: the Bogalusa Heart Study. J Am Diet Assoc. 1988 Apr;88(4):466-71. PMID 3351166
- [Background] Downey AM, Virgilio SJ, Serpas DC, Nicklas TA, Arbeit ML, Berenson GS. "Heart Smart"--a staff development model for a school-based cardiovascular health intervention. Health Educ. 1988 Apr-May;19(2):12-20. No abstract available. PMID 3152217
- [Background] Johnson CC, Nicklas TA, Arbeit ML, Franklin FA, Berenson GS: A Comprehensive Model for Maintenance of Family Health Behaviors; The 'Heart Smart' Family Health Promotion Program. Family Commun Hlth, 11:1-7, 1988
- [Background] Nicklas TA, Farris RP, Smoak CG, Frank GC, Srinivasan SR, Webber LS, Berenson GS. Dietary factors relate to cardiovascular risk factors in early life. Bogalusa Heart Study. Arteriosclerosis. 1988 Mar-Apr;8(2):193-9. doi: 10.1161/01.atv.8.2.193. PMID 3348759
- [Background] Frank GC, Webber LS, Nicklas TA, Berenson GS. Sodium, potassium, calcium, magnesium, and phosphorus intakes of infants and children: Bogalusa Heart Study. J Am Diet Assoc. 1988 Jul;88(7):801-7. PMID 3385103
- [Background] Freedman DS, Newman WP 3rd, Tracy RE, Voors AE, Srinivasan SR, Webber LS, Restrepo C, Strong JP, Berenson GS. Black-white differences in aortic fatty streaks in adolescence and early adulthood: the Bogalusa Heart Study. Circulation. 1988 Apr;77(4):856-64. doi: 10.1161/01.cir.77.4.856. PMID 3258194
- [Background] Nicklas TA, Arbeit ML, Johnson CC, Franklin FA, Berenson GS: Intervention on Family Eating Behavior for Children at High Risk: Heart Smart Program. J Nutr Educ, 20:128-132, 1988
- [Background] Cresanta JL, Farris RP, Croft JB, Webber LS, Frank GC, Berenson GS. Trends in fatty acid intakes of 10-year-old children, 1973 to 1982. J Am Diet Assoc. 1988 Feb;88(2):178-84. PMID 3339204
- [Background] Shear CL, Freedman DS, Burke GL, Harsha DW, Webber LS, Berenson GS. Secular trends of obesity in early life: the Bogalusa Heart Study. Am J Public Health. 1988 Jan;78(1):75-7. doi: 10.2105/ajph.78.1.75. PMID 3337310
- [Background] Berenson GS, Srinivasan SR, Nicklas TA, Webber LS. Cardiovascular risk factors in children and early prevention of heart disease. Clin Chem. 1988;34(8B):B115-22. PMID 3042194
- [Background] Sharma C, Dalferes ER Jr, Freedman DS, Asamoah A, Berenson GS. Use of 86Rb and 22Na in assaying active and cotransport activities in human erythrocytes in a biracial population. Clin Chim Acta. 1988 Aug 31;176(2):133-42. doi: 10.1016/0009-8981(88)90200-8. PMID 3180461
- [Background] Bao W, Threefoot SA, Srinivasan SR, Berenson GS. Essential hypertension predicted by tracking of elevated blood pressure from childhood to adulthood: the Bogalusa Heart Study. Am J Hypertens. 1995 Jul;8(7):657-65. doi: 10.1016/0895-7061(95)00116-7. PMID 7546488
- [Background] Tracy RE, Newman WP 3rd, Wattigney WA, Srinivasan SR, Strong JP, Berenson GS. Histologic features of atherosclerosis and hypertension from autopsies of young individuals in a defined geographic population: the Bogalusa Heart Study. Atherosclerosis. 1995 Aug;116(2):163-79. doi: 10.1016/0021-9150(95)05525-2. PMID 7575772
- [Background] Berenson GS, Pickoff AS. Preventive cardiology and its potential influence on the early natural history of adult heart diseases: the Bogalusa Heart Study and the Heart Smart Program. Am J Med Sci. 1995 Dec;310 Suppl 1:S133-8. doi: 10.1097/00000441-199512000-00024. PMID 7503117
- [Background] Berenson GS, Wattigney WA, Bao W, Srinivasan SR, Radhakrishnamurthy B. Rationale to study the early natural history of heart disease: the Bogalusa Heart Study. Am J Med Sci. 1995 Dec;310 Suppl 1:S22-8. doi: 10.1097/00000441-199512000-00005. PMID 7503119
- [Background] Webber LS, Wattigney WA, Srinivasan SR, Berenson GS. Obesity studies in Bogalusa. Am J Med Sci. 1995 Dec;310 Suppl 1:S53-61. doi: 10.1097/00000441-199512000-00010. PMID 7503125
- [Background] Srinivasan SR, Berenson GS. Childhood lipoprotein profiles and implications for adult coronary artery disease: the Bogalusa Heart Study. Am J Med Sci. 1995 Dec;310 Suppl 1:S62-7. doi: 10.1097/00000441-199512000-00011. PMID 7503126
- [Background] Berenson GS, Radhakrishnamurthy B, Bao W, Srinivasan SR. Does adult-onset diabetes mellitus begin in childhood?: the Bogalusa Heart Study. Am J Med Sci. 1995 Dec;310 Suppl 1:S77-82. doi: 10.1097/00000441-199512000-00014. PMID 7503129
- [Background] Gidding SS, Bao W, Srinivasan SR, Berenson GS. Effects of secular trends in obesity on coronary risk factors in children: the Bogalusa Heart Study. J Pediatr. 1995 Dec;127(6):868-74. doi: 10.1016/s0022-3476(95)70020-x. PMID 8523181
- [Background] Srinivasan SR, Bao W, Wattigney WA, Berenson GS. Adolescent overweight is associated with adult overweight and related multiple cardiovascular risk factors: the Bogalusa Heart Study. Metabolism. 1996 Feb;45(2):235-40. doi: 10.1016/s0026-0495(96)90060-8. PMID 8596496
- [Background] Bao W, Srinivasan SR, Berenson GS. Persistent elevation of plasma insulin levels is associated with increased cardiovascular risk in children and young adults. The Bogalusa Heart Study. Circulation. 1996 Jan 1;93(1):54-9. doi: 10.1161/01.cir.93.1.54. PMID 8616941
- [Background] Bao W, Srinivasan SR, Wattigney WA, Bao W, Berenson GS. Usefulness of childhood low-density lipoprotein cholesterol level in predicting adult dyslipidemia and other cardiovascular risks. The Bogalusa Heart Study. Arch Intern Med. 1996 Jun 24;156(12):1315-20. PMID 8651840
- [Background] Agirbasli M, Radhakrishnamurthy B, Jiang X, Bao W, Berenson GS. Urinary N-acetyl-beta-D-glucosaminidase changes in relation to age, sex, race, and diastolic and systolic blood pressure in a young adult biracial population. The Bogalusa Heart Study. Am J Hypertens. 1996 Feb;9(2):157-61. doi: 10.1016/0895-7061(95)00336-3. PMID 8924265
- [Background] Valdez R, Greenlund KJ, Wattigney WA, Bao W, Berenson GS. Use of weight-for-height indices in children to predict adult overweight: the Bogalusa Heart Study. Int J Obes Relat Metab Disord. 1996 Aug;20(8):715-21. PMID 8856393
- [Background] Berenson GS, Bao W, Srinivasan SR. Abnormal characteristics in young offspring of parents with non-insulin-dependent diabetes mellitus. The Bogalusa Heart Study. Am J Epidemiol. 1996 Nov 15;144(10):962-7. doi: 10.1093/oxfordjournals.aje.a008866. PMID 8916507
- [Background] Berenson GS, Turner M, O'Meallie LP, Puyau FA, Pargaonkar PS, Srinivasan S, Hall RJ. A study of serum lipoproteins and angiographic evidence of coronary artery disease. South Med J. 1975 Dec;68(12):1513-9. doi: 10.1097/00007611-197512000-00014. PMID 173025
- [Background] Fox MH, Dessauer HC, Srinivasan SR, Thurmon TF, Berenson GS. Variability of polymorphic cellular enzymes in medical students with different serum lipid levels: a preliminary survey. Clin Chim Acta. 1975 Sep 1;63(2):149-55. doi: 10.1016/0009-8981(75)90157-6. PMID 170024
- [Background] Voors AW. Cuff bladder size in a blood pressure survey of children. Am J Epidemiol. 1975 Jun;101(6):489-94. doi: 10.1093/oxfordjournals.aje.a112119. PMID 1155428
- [Background] Berenson GS, Srinivasan SR, Frerichs RR. Not-so-hyper hyperlipo-proteinemia and coronary artery disease. Postgrad Med. 1976 Apr;59(4):173-8. doi: 10.1080/00325481.1976.11714336. PMID 177963
- [Background] Frerichs RR, Srinivasan SR, Webber LS, Berenson GR. Serum cholesterol and triglyceride levels in 3,446 children from a biracial community: the Bogalusa Heart Study. Circulation. 1976 Aug;54(2):302-9. doi: 10.1161/01.cir.54.2.302. PMID 939028
- [Background] Voors AW, Foster TA, Frerichs RR, Webber LS, Berenson GS. Studies of blood pressures in children, ages 5-14 years, in a total biracial community: the Bogalusa Heart Study. Circulation. 1976 Aug;54(2):319-27. doi: 10.1161/01.cir.54.2.319. PMID 939029
- [Background] Srinivasan SR, Frerichs RR, Webber LS, Berenson GS. Serum lipoprotein profile in children from a biracial community: the Bogalusa Heart Study. Circulation. 1976 Aug;54(2):309-18. doi: 10.1161/01.cir.54.2.309. PMID 181171
- [Background] Frank GC, Berenson GS, Schilling PE, Moore MC. Adapting the 24-hr. recall for epidemiologic studies of school children. J Am Diet Assoc. 1977 Jul;71(1):26-31. PMID 864159
- [Background] Frank GC, Voors AW, Schilling PE, Berenson GS. Dietary studies of rural school children in a cardiovascular survey. J Am Diet Assoc. 1977 Jul;71(1):31-5. No abstract available. PMID 864160
- [Background] Foster TA, Voors AW, Webber LS, Frerichs RR, Berenson GS. Anthropometric and maturation measurements of children, ages 5 to 14 years, in a biracial community--the Bogalusa Heart Study. Am J Clin Nutr. 1977 Apr;30(4):582-91. doi: 10.1093/ajcn/30.4.582. PMID 851088
- [Background] Voors AW, Webber LS, Berenson GS: A Consideration of Essential Hypertension in the Pediatric Age. Practical Cardiol, 3:29, 1977
- [Background] Frerichs RR, Srinivasan SR, Webber LS, Berenson GS: Serum Cholesterol and Triglyceride Levels in Children From a Biracial Community - The Bogalusa Heart Study. International Workshop-Conference on Atherosclerosis, London, Ontario, Canada, September 1975. Atherosclerosis. (G.W. Manning and M.D. Haust Eds.) Plenum Publ. Corp, New York, p. 204, 1977
- [Background] Voors AW, Webber LS, Frerichs RR, Berenson GS. Body height and body mass as determinants of basal blood pressure in children--The Bogalusa Heart Study. Am J Epidemiol. 1977 Aug;106(2):101-8. doi: 10.1093/oxfordjournals.aje.a112439. PMID 888812
- [Background] Frerichs RR, Webber LS, Srinivasan SR, Berenson GS. Hemoglobin levels in children from a biracial southern community. Am J Public Health. 1977 Sep;67(9):841-5. doi: 10.2105/ajph.67.9.841. PMID 900323
- [Background] Webber LS, Voors AW, Foster TA, Berenson GS. A study of instruments in preparation for a blood pressure survey of children. Circulation. 1977 Oct;56(4 Pt 1):651-6. doi: 10.1161/01.cir.56.4.651. PMID 902391
- [Background] Berenson GS: Risk Factors in Children - the Early Natural History of Arteriosclerosis. Tokyo. In: Atherosclerosis IV, (G Schettler, Goto Y, Hata G, Klose, Eds.) Springer-Verlag, Berlin, Heidelberg, p. 489, 1977
- [Background] Frank GC, Berenson GS, Webber LS. Dietary studies and the relationship of diet to cardiovascular disease risk factor variables in 10-year-old children--The Bogalusa Heart Study. Am J Clin Nutr. 1978 Feb;31(2):328-40. doi: 10.1093/ajcn/31.2.328. PMID 623054
- [Background] Voors AW, Webber LS, Berenson GS. Epidemiology of essential hypertension in youth--implications for clinical practice. Pediatr Clin North Am. 1978 Feb;25(1):15-27. doi: 10.1016/s0031-3955(16)33528-3. PMID 628561
- [Background] Berenson GS, Foster TA, Frank GC, Frerichs RR, Srinivasan SR, Voors AW, Webber LS. Cardiovascular disease risk factor variables at the preschool age. The Bogalusa heart study. Circulation. 1978 Mar;57(3):603-12. doi: 10.1161/01.cir.57.3.603. No abstract available. PMID 624172
- [Background] Berenson GS, Voors AW, Webber LS, Frerichs RR. Blood pressure in children and its interpretation. Pediatrics. 1978 Feb;61(2):333-6. No abstract available. PMID 634708
- [Background] Voors AW, Webber LS, Berenson GS. Blood pressure of children, ages 2 1/2-5 1/2 years, in a total community--the Bogalusa heart study. Am J Epidemiol. 1978 May;107(5):403-11. doi: 10.1093/oxfordjournals.aje.a112558. PMID 665656
- [Background] Shear CL, Frerichs RR, Weinberg R, Berenson GS. Childhood sibling aggregation of coronary artery disease risk factor variables in a biracial community. Am J Epidemiol. 1978 Jun;107(6):522-8. doi: 10.1093/oxfordjournals.aje.a112571. PMID 665666
- [Background] Frerichs RR, Srinivasan SR, Webber LS, Rieth MC, Berenson GS. Serum lipids and lipoproteins at birth in a biracial population: the Bogalusa heart study. Pediatr Res. 1978 Aug;12(8):858-63. doi: 10.1203/00006450-197808000-00011. PMID 210440
- [Background] Voors AW, Webber LS, Berenson GS: Relationship of Blood Pressure Levels to Height and Weight in Children. Cardiovasc Med, 3:911, 1978
- [Background] Frank GC, Farris RP, Berenson GS: Dietitians' Response to Knowledge of Their Own Cardiovascular Risk. J Nutr Ed, 10:105, 1978
- [Background] Berenson GS, Webber LS, Srinivasan SR, Frerichs RR, Voors AW: Interrelationship and Persistence of Risk Factor Variables at High Levels in Children - The Bogalusa Heart Study The 5th International Conference on Atherosclerosis, Milan, Italy, November 1977, (L. A. Carlson, R. Paoletti, C. R. Sirtori, and G. Weber, Eds.) Raven Press, New York, p. 357, 1978
- [Background] Srinivasan SR, Berenson GS, Frerichs RR: Serum Lipids and Lipoproteins in Children. In: Atherosclerosis: Its Pediatric Aspects (W. B. Strong, Ed.) Grune and Stratton, New York, p. 85, 1978
- [Background] Berenson GS: Children, the Next Generation of Patients with Myocardial Infarction. Proceedings of the International Kronberg Symposium, Frankfurt, Germany, May 1977. Changes in the Medical Panorama, (G. Schettler, J. Drews, and H. Greten, Eds.) Georg Thieme Publishers, Stuttgart, Germany, p. 75, 1978
- [Background] Harsha DW, Frerichs RR, Berenson GS. Densitometry and anthropometry of black and white children. Hum Biol. 1978 Sep;50(3):261-80. No abstract available. PMID 721084
- [Background] Frerichs RR, Webber LS, Srinivasan SR, Berenson GS. Relation of serum lipids and lipoproteins to obesity and sexual maturity in white and black children. Am J Epidemiol. 1978 Dec;108(6):486-96. doi: 10.1093/oxfordjournals.aje.a112647. PMID 216263
- [Background] Harsha DW, Frerichs RR, Berenson GS. A simple and complete densitometric technique for underwater weighing. J Sports Med Phys Fitness. 1978 Sep;18(3):253-62. No abstract available. PMID 732300
- [Background] Srinivasan SR, Foster TA, Berenson GS. Efficacy of a simplified primary screening procedure for detection of hyperlipoproteinemias in a pediatric population. Clin Chem. 1979 Feb;25(2):242-6. PMID 215345
- [Background] Berenson GS, Srinivasan SR, Frerichs RR, Webber LS. Serum high density lipoprotein and its relationship to cardiovascular disease risk factor variables in children--the Bogalusa heart study. Lipids. 1979 Jan;14(1):91-8. doi: 10.1007/BF02533576. PMID 218070
- [Background] Voors AW, Webber LS, Berenson GS. Time course studies of blood pressure in children--the Bogalusa Heart Study. Am J Epidemiol. 1979 Mar;109(3):320-34. doi: 10.1093/oxfordjournals.aje.a112685. PMID 453169
- [Background] Frerichs RR, Harsha DW, Berenson GS. Equations for estimating percentage of body fat in children 10--14 years old. Pediatr Res. 1979 Mar;13(3):170-4. doi: 10.1203/00006450-197903000-00007. PMID 471571
- [Background] Blonde CV, Frerichs RR, Foster TA, Webber LS, Berenson GS. Physician-diagnosed abnormalities in black and white children in a total community. Public Health Rep. 1979 Mar-Apr;94(2):124-9. No abstract available. PMID 432404
- [Background] Frerichs RR, Webber LS, Voors AW, Srinivasan SR, Berenson GS. Cardiovascular disease risk factor variables in children at two successive years--the Bogalusa heart study. J Chronic Dis. 1979;32(3):251-62. doi: 10.1016/0021-9681(79)90071-7. No abstract available. PMID 218982
- [Background] Webber LS, Voors AW, Srinivasan SR, Frerichs RR, Berenson GS. Occurrence in children of multiple risk factors for coronary artery disease: the Bogalusa heart study. Prev Med. 1979 May;8(3):407-18. doi: 10.1016/0091-7435(79)90018-5. No abstract available. PMID 471959
- [Background] Berenson GS, Voors AW, Dalferes ER Jr, Webber LS, Shuler SE. Creatinine clearance, electrolytes, and plasma renin activity related to the blood pressure of white and black children--the Bogalusa Heart Study. J Lab Clin Med. 1979 Apr;93(4):535-48. No abstract available. PMID 429858
- [Background] Voors AW, Berenson GS, Dalferes ER, Webber LS, Shuler SE. Racial differences in blood pressure control. Science. 1979 Jun 8;204(4397):1091-4. doi: 10.1126/science.451554.
- [Background] Hunter SM, Frerichs RR, Webber LS, Berenson GS. Social status and cardiovascular disease risk factor variables in children: the Bogalusa Heart Study. J Chronic Dis. 1979;32(6):441-9. doi: 10.1016/0021-9681(79)90104-8. No abstract available. PMID 222792
- [Background] Berenson GS, Blonde CV, Farris RP, Foster TA, Frank GC, Srinivasan SR, Voors AW, Webber LS. Cardiovascular disease risk factor variables during the first year of life. Am J Dis Child. 1979 Oct;133(10):1049-57. doi: 10.1001/archpedi.1979.02130100073015. PMID 495597
- [Background] Voors AW, Webber LS, Berenson GS. A choice of diastolic Korotkoff phases in mercury sphygmomanometry of children. Prev Med. 1979 Jul;8(4):492-9. doi: 10.1016/0091-7435(79)90323-2. No abstract available. PMID 471964
- [Background] Berenson GS, Voors AW, Webber LS, Dalferes ER Jr, Harsha DW. Racial differences of parameters associated with blood pressure levels in children--the Bogalusa heart study. Metabolism. 1979 Dec;28(12):1218-28. doi: 10.1016/0026-0495(79)90134-3. PMID 514082
- [Background] Berenson GS, Voors AW, Webber LS: Blood Pressure Levels in Black and White Children Related to the Early Onset of Essential Hypertension. Proceedings, VIII World Congress of Cardiology, Tokyo. (S. Hayase and S. Murae, Eds.) Excerpta Medica, Amsterdam, p. 406-413, 1979
- [Background] Berenson GS, Srinivasan SR, Webber LS: Prognostic Significance of Lipid Profiles in Children. In: Childhood Prevention of Atherosclerosis and Hypertension, (R.M. Lauer, and R.B. Shekelle, Eds.) Raven Press, New York, p. 75-86, 1980
- [Background] Harsha DW, Voors AW, Berenson GS. Racial differences in subcutaneous fat patterns in children aged 7--15 years. Am J Phys Anthropol. 1980 Sep;53(3):333-7. doi: 10.1002/ajpa.1330530303. PMID 7468776
- [Background] Berenson GS, Srinivasan SR, Voors AW, Webber LS: Clues to Mechanisms of Cardiovascular Disease From an Epidemiologic Study of Children - The Bogalusa Heart Study. In: Atherosclerosis V (Gotto AM Jr, Smith LC, Allen B, Eds). New York: Springer-Verlag, p. 272-277, 1980
- [Background] Hunter SM, Webber LS, Berenson GS. Cigarette smoking and tobacco usage behavior in children with adolescents: Bogalusa Heart Study. Prev Med. 1980 Nov;9(6):701-12. doi: 10.1016/0091-7435(80)90015-8. No abstract available. PMID 7454695
- [Background] Webber LS, Srinivasan SR, Voors AW, Berenson GS. Persistence of levels for risk factor variables during the first year of life: the Bogalusa Heart Study. J Chronic Dis. 1980;33(3):157-67. doi: 10.1016/0021-9681(80)90015-6. No abstract available. PMID 7354104
- [Background] Foster TA, Webber LS, Srinivasan SR, Voors AW, Berenson GS. Measurement error of risk factor variables in an epidemiologic study of children-the Bogalusa heart study. J Chronic Dis. 1980;33(10):661-72. doi: 10.1016/0021-9681(80)90009-0. No abstract available. PMID 6967874
- [Background] Voors AW, Webber LS, Berenson GS. Time course study of blood pressure in children over a three-year period. Bogalusa Heart Study. Hypertension. 1980 Jul-Aug;2(4 Pt 2):102-8. PMID 7399641
- [Background] Srinivasan SR, Foster TA, Berenson GS. Comparability of results by simplified methods for measuring serum lipoprotein cholesterol in a pediatric population. Clin Chem. 1980 Oct;26(11):1548-53. PMID 7418200
- [Background] Voors AW, Berenson GS, Shuler SE, Webber LS: Blood Pressure, Electrolyte Clearance, and Plasma Renin Activity in Children Sampled From an Entire Community J Appl Biochem, 2:87-99, 1980
- [Background] Voors AW, Webber LS, Berenson GS. Racial contrasts in cardiovascular response tests for children from a total community. Hypertension. 1980 Sep-Oct;2(5):686-94. doi: 10.1161/01.hyp.2.5.686. PMID 7419269
- [Background] Voors AW, Webber LS, Berenson GS: Epidemiologia de la Hipertension Arterial en Ninos Estadunidenses. In: Hipertension Arterial 1980. First Interamerican Course on Hypertension, Mexico City, Feb. 1979 (Gonzalez Caamano A, Alcocer DB, L, Eds). Mexico City: Ediciones Medicas Actualizadas, SA, p.91-102, 1980
- [Background] Voors AW, Webber LS, Berenson GS: Epidemiologia de la Hipertension Arterial an Adolescentes Estadunidenses. In: Hipertension Arterial 1980, First Interamerican Course on Hypertension, Mexico City, Feb. 1979 (Gonzalez Caamano A, Alcocer DB, L, Eds). Mexico City: Ediciones Medicas Actualizadas, SA, p. 103-115, 1980
- [Background] Berenson GS, Voors AW, Webber LS: Importance of Blood Pressures in Children - Distribution and Measurable Determinants. In: Epidemiology of Arterial Blood Pressure (Kesteloot H, Joossens JV Eds). The Hague, Netherlands: Martinus Nijhoff Publishers, p. 71-97, 1980
- [Background] Voors AW, Webber LS, Harsha DW, Frank GC, Berenson GS: Obesity: Determinants and Consequences in Children of An Entire Biracial Population - The Bogalusa Heart Study. J Chron Dis Ther Res, 4:169-191, 1980
- [Background] Berenson GS, Srinivasan SR, Cresanta JL, Foster TA, Webber LS. Dynamic changes of serum lipoproteins in children during adolescence and sexual maturation. Am J Epidemiol. 1981 Feb;113(2):157-70. doi: 10.1093/oxfordjournals.aje.a113080. PMID 7468573
- [Background] Voors AW, Frank GC, Srinivasan SR, Webber LS, Berenson GS. Hemoglobin levels and dietary iron in pubescent children in a biracial community. Public Health Rep. 1981 Jan-Feb;96(1):45-9. PMID 7454955
- [Background] Voors AW, Harsha DW, Webber LS, Berenson GS. Obesity and external sexual maturation---the Bogalusa Heart Study. Prev Med. 1981 Jan;10(1):50-61. doi: 10.1016/0091-7435(81)90005-0. No abstract available. PMID 6972036
- [Background] Blonde CV, Webber LS, Foster TA, Berenson GS. Parental history and cardiovascular disease risk factor variables in children. Prev Med. 1981 Jan;10(1):25-37. doi: 10.1016/0091-7435(81)90003-7. No abstract available. PMID 6972035
- [Background] Berenson GS, Voors AW, Webber LS: Hypertension in the Young - Measurement and Criteria. In: Phasic Pressor Mechanisms: Hypertension in the Young and the Old (Onesti G, Kim KE, Eds). New York: Grune and Stratton, p. 3-10, 1981
- [Background] Voors AW, Berenson GS: Search for the Determinants of the Early Onset of Essential Hypertension. In: Phasic Pressor Mechanisms: Hypertension in the Young and the Old (Onesti G, Kim KE, Eds). New York: Grune and Stratton, p. 43-55, 1981
- [Background] Berenson GS, Voors AW, Webber LS: Epidemiology in a Biracial Community in the Rural South of the United States. In: Phasic Pressor Mechanisms: Hypertension in the Young and Old (Onesti G, Kim KE, Eds). New York: Grune and Stratton, p. 183-190, 1981
- [Background] Voors AW, Radhakrishnamurthy B, Srinivasan SR, Webber LS, Berenson GS. Plasma glucose level related to blood pressure in 272 children, ages 7-15 years, sampled from a total biracial population. Am J Epidemiol. 1981 Apr;113(4):347-56. doi: 10.1093/oxfordjournals.aje.a113103. PMID 7211820
- [Background] Berenson GS, Srinivasan SR, Frank GC, Webber LS. Serum lipid and lipoprotein in infants and children and their relationship with diet. Prog Clin Biol Res. 1981;61:73-94. PMID 6976578
- [Background] Berenson GS, Radhakrishnamurthy B, Srinivasan SR, Voors AW, Foster TA, Dalferes ER Jr, Webber LS. Plasma glucose and insulin levels in relation to cardiovascular risk factors in children from a biracial population-the Bogalusa Heart Study. J Chronic Dis. 1981;34(8):379-91. doi: 10.1016/0021-9681(81)90037-0. No abstract available. PMID 7021577
- [Background] Wolf TM, Hunter SM, Webber LS, Berenson GS. Self-concept, locus of control, goal blockage, and coronary-prone behavior pattern in children and adolescents: Bogalusa heart study. J Gen Psychol. 1981 Jul;105(1st Half):13-26. doi: 10.1080/00221309.1981.9921056. PMID 7264614
- [Background] Fox MH, Weyer SM, Thurmon TF, Berenson GS. Genetically controlled enzymatic variation in a southern, biracial, semi-rural community: the Bogalusa heart study. Hum Hered. 1981;31(3):138-51. doi: 10.1159/000153196. PMID 7262887
- [Background] Fox MH, Webber LS, Srinivasan SR, Thurmon TF, Berenson GS. ABO blood group associations with cardiovascular risk factor variables. I. Serum lipids and lipoproteins. The Bogalusa heart study. Hum Biol. 1981 Sep;53(3):411-37. No abstract available. PMID 7309026
- [Background] Sklov MC, Srinivasan SR, Webber LS, Berenson GS. Variability of total cholesterol concentrations in serum by repeated measurements in a large pediatric population--limitations of quality controls for laboratory analyses. Clin Chem. 1981 Dec;27(12):1988-92. PMID 7307251
- [Background] Berenson GS, Voors AW, Webber LS: Blood Pressure in Children and Factors Predisposing to Hypertensive Disease in Adults. In: Paediatric Cardiology, Vol 4 (Godman MJ, Ed). Edinburgh: Churchill Livingstone, p. 591-600, 1981
- [Background] Cresanta JL, Srinivasan SR, Foster TA, Webber LS, Berenson GS. Serum lipoprotein levels in children: epidemiologic and clinical implications. J Chronic Dis. 1982;35(1):41-51. doi: 10.1016/0021-9681(82)90028-5. No abstract available. PMID 7068801
- [Background] Wolf TM, Sklov MC, Wenzl PA, Hunter SM, Berenson GS. Validation of a measure of type A behavior pattern in children: Bogalusa heart study. Child Dev. 1982 Feb;53(1):126-35. PMID 7060417
- [Background] Farris RP, Frank GC, Webber LS, Srinivasan SR, Berenson GS. Influence of milk source on serum lipids and lipoproteins during the first year of life, Bogalusa heart study. Am J Clin Nutr. 1982 Jan;35(1):42-9. doi: 10.1093/ajcn/35.1.42. PMID 7064877
- [Background] Webber LS, Hunter SM, Baugh JG, Srinivasan SR, Sklov MC, Berenson GS. The interaction of cigarette smoking, oral contraceptive use, and cardiovascular risk factor variables in children: the Bogalusa Heart Study. Am J Public Health. 1982 Mar;72(3):266-74. doi: 10.2105/ajph.72.3.266. PMID 7058967
- [Background] Berenson GS, Webber LS, Voors AW: Diagnostic Challenge: Diagnosing Hypertension in Children. J Cardiovasc Med, 7:273-279, 1982
- [Background] Voors AW, Sklov MC, Halperin H, Webber LS, Berenson GS. Comparison of two automatic blood pressure recorders and the mercury sphygomomanometer. Hypertension. 1982 Mar-Apr;4(2):329-36. doi: 10.1161/01.hyp.4.2.329. PMID 7068191
- [Background] Voors AW, Srinivasan SR, Hunter SM, Webber LS, Sklov MC, Berenson GS. Smoking, oral contraceptives, and serum lipid and lipoprotein levels in youths. Prev Med. 1982 Jan;11(1):1-12. doi: 10.1016/0091-7435(82)90001-9. No abstract available. PMID 7079241
- [Background] Hunter SM, Baugh JG, Webber LS, Sklov MC, Berenson GS. Social learning effects on trial and adoption of cigarette smoking in children: The Bogalusa heart study. Prev Med. 1982 Jan;11(1):29-42. doi: 10.1016/0091-7435(82)90003-2. No abstract available. PMID 7079245
- [Background] Wolf TM, Sklov MC, Hunter SM, Berenson GS: Factor Analytic Study of the Children's Nowicki-Strickland Locus of Control Scale. Educ Psychol Measure, 42:333-337, 1982
- [Background] Voors AW, Sklov MC, Wolf TM, Hunter SM, Berenson GS: Cardiovascular Risk Factors in Children and Coronary Related Behavior. In: Promoting Adolescent Health: A Dialogue on Research and Practice (Coates T, Petersen A, Perry C, Eds). New York: Academic Press, p. 281-304, 1982
- [Background] Frank GC, Berenson GS, Webber LS: Dietary Studies of Infants and Children. In: Promoting Adolescent Health: A Dialogue on Research and Practice (Coates T, Petersen A, Perry C, Eds). New York: Academic Press, p. 329-354, 1982
- [Background] Voors AW, Harsha DW, Webber LS, Berenson GS. Relation of blood pressure to stature in healthy young adults. Am J Epidemiol. 1982 Jun;115(6):833-40. doi: 10.1093/oxfordjournals.aje.a113370. No abstract available. PMID 7091142
- [Background] Frank GC, Webber LS, Berenson GS: Dietary Studies of 10-Year-Old Children in the Bogalusa Heart Study. In: Nutrition and Heart Disease (Naito HK, Ed). Jamaica, New York: Spectrum Publications, p. 91-110, 1982
- [Background] Berenson GS, Voors AW, Frank GC, Webber LS: Studies of Blood Pressure and Dietary Sodium Intake in Children in Semirural Southern United States: The Bogalusa Heart Study. In: The Role of Salt in Cardiovascular Hypertension (Fregly MJ, Kare MR, Eds). New York: Academic Press, p. 49-62, 1982
- [Background] Hunter SM, Wolf TM, Sklov MC, Webber LS, Watson RM, Berenson GS. Type A coronary-prone behavior pattern and cardiovascular risk factor variables in children and adolescents: the Bogalusa Heart Study. J Chronic Dis. 1982;35(8):613-21. doi: 10.1016/0021-9681(82)90013-3. PMID 7096525
- [Background] Berenson GS, Webber LS, Srinivasan SR, Voors AW, Harsha DW, Dalferes ER Jr. Biochemical and anthropometric determinants of serum beta- and pre-beta-lipoproteins in children. Bogalusa Heart Study. Arteriosclerosis. 1982 Jul-Aug;2(4):325-34. doi: 10.1161/01.atv.2.4.325. PMID 6981403
- [Background] Voors AW, Harsha DW, Webber LS, Radhakrishnamurthy B, Srinivasan SR, Berenson GS. Clustering of anthropometric parameters, glucose tolerance, and serum lipids in children with high and low beta- and pre-beta-lipoproteins. Bogalusa Heart Study. Arteriosclerosis. 1982 Jul-Aug;2(4):346-55. doi: 10.1161/01.atv.2.4.346. PMID 7052036
- [Background] Weinberg R, Webber LS, Berenson GS. Hereditary and environmental influences on cardiovascular risk factors for children: the Bogalusa Heart Study. Am J Epidemiol. 1982 Aug;116(2):385-93. doi: 10.1093/oxfordjournals.aje.a113422. PMID 7114047
- [Background] Voors AW, Webber LS, Berenson GS. Resting heart rate and pressure-rate product of children in a total biracial community: the Bogalusa Heart Study. Am J Epidemiol. 1982 Aug;116(2):276-86. doi: 10.1093/oxfordjournals.aje.a113412. PMID 7114038
- [Background] Baugh JG, Hunter SM, Webber LS, Berenson GS. Development trends of first cigarette smoking experience of children: the Bogalusa heart study. Am J Public Health. 1982 Oct;72(10):1161-4. doi: 10.2105/ajph.72.10.1161. PMID 7114342
- [Background] Berenson GS, Frank GC, Hunter SM, Srinivasan SR, Voors AW, Webber LS. Cardiovascular risk factors in children. Should they concern the pediatrician? Am J Dis Child. 1982 Sep;136(9):855-62. doi: 10.1001/archpedi.1982.03970450097024. PMID 7051814
- [Background] Srinivasan SR, Webber LS, Berenson GS. Lipid composition and interrelationships of major serum lipoproteins. Observations in children with different lipoprotein profiles. Bogalusa Heart Study. Arteriosclerosis. 1982 Jul-Aug;2(4):335-45. doi: 10.1161/01.atv.2.4.335. No abstract available. PMID 6956268
- [Background] Berenson GS, Voors AW, Frank G, Webber LS. Adolescent hypertension: a new dimension. N Y State J Med. 1982 Oct;82(11):1571-5. No abstract available. PMID 6959005
- [Background] Akman D, Berenson GS, Blonde CV, Webber LS, Stopa AR. Heart disease in a total population of children: the Bogalusa Heart Study. South Med J. 1982 Oct;75(10):1177-81. doi: 10.1097/00007611-198210000-00006. PMID 6981850
- [Background] Wolf TM, Sklov MC, Hunter SM, Webber LS, Berenson GS. Factor analytic study of the Piers-Harris Children's Self-Concept Scale. J Pers Assess. 1982 Oct;46(5):511-3. doi: 10.1207/s15327752jpa4605_11. PMID 16367632
- [Background] Frank GC, Farris RP, Ditmarsen P, Voors AW, Berenson GS. An approach to primary preventive treatment for children with high blood pressure in a total community. J Am Coll Nutr. 1982;1(4):357-74. doi: 10.1080/07315724.1982.10719006. PMID 7185868
- [Background] Srinivasan SR, Webber LS, Whitaker CF, Berenson GS. Quantification of lipoprotein cholesterol in serum from children with different lipoprotein profiles: heparin-calcium precipitation and ultracentrifugation compared. Clin Chem. 1983 Mar;29(3):481-5. PMID 6572114
- [Background] Berenson GS, Voors AW, Webber LS, Frank GC, Farris RP, Tobian L, Aristimuno GG. A model of intervention for prevention of early essential hypertension in the 1980s. Hypertension. 1983 Jan-Feb;5(1):41-54. doi: 10.1161/01.hyp.5.1.41. PMID 6848468
- [Background] Voors AW, Dalferes ER Jr, Frank GC, Aristimuno GG, Berenson GS. Relation between ingested potassium and sodium balance in young Blacks and whites. Am J Clin Nutr. 1983 Apr;37(4):583-94. doi: 10.1093/ajcn/37.4.583. PMID 6837493
- [Background] Berenson GS: Racial Differences in Hypertension. In: Hypertension: Prevention, Diet, and Treatment in Infancy and Childhood, (Blumenthal S, Chairman and Ed). Proceedings from a Symposium Sponsored by Wyeth Laboratories, Bethesda, MD, May 25, 1983. Library of Congress No. 83-072205, p. 24-28, 1983
- [Background] Cresanta JL, Srinivasan SR, Foster TA, Webber LS, Berenson GS. Distributions of serum lipoproteins in children by repeated measurements. Prev Med. 1983 Jul;12(4):554-68. doi: 10.1016/0091-7435(83)90209-8. PMID 6604913
- [Background] Frank GC, Nicolich J, Voors AW, Webber LS, Berenson GS. A simplified inventory method for quantitating dietary sodium, potassium, and energy. Am J Clin Nutr. 1983 Sep;38(3):474-80. doi: 10.1093/ajcn/38.3.474. PMID 6613917
- [Background] Berenson GS, Voors AW, Gard P, Newman WP III, Tracy RE: Clinical and Anatomic Correlates of Cardiovascular Disease in Children from the Bogalusa Heart Study. In: Atherosclerosis VI (Schettler FG, Gotto AM Jr, Middlehoff G, Habenicht AGR, Jurutke KR, Eds). New York: Springer-Verlag, p. 60-65, 1983
- [Background] Conference on Blood Lipids in Children: optimal levels for early prevention of coronary artery disease. Workshop report: Epidemiologic Section. April 18 and 19, 1983, American Health Foundation. Prev Med. 1983 Nov;12(6):741-97. doi: 10.1016/0091-7435(83)90259-1. No abstract available. PMID 6374648
- [Background] Srinivasan SR, Berenson GS: Serum Lipoproteins in Children and Methods for Study. In: CRC Handbook of Electrophoresis (Lipoproteins), Vol III (Lewis LA, Opplt JJ, Eds). Boca Raton, Florida: CRC Press, p. 185-203, 1983
- [Background] Berenson GS, Webber LS, Frank GC, Farris RP: Management of the Mildly Hypertensive Youth: Can Adult Hypertensive Disease be Prevented? In NHLBI Workshop on Juvenile Hypertension (Loggie JMH, Horan MJ, Gruskin AB, Hohn AR, Dunbar JB, Havlik RJ, Eds). New York: Biomedical Information Corp., p. 387-407, 1984
- [Background] Berenson GS, Cresanta JL, Webber LS. High blood pressure in the young. Annu Rev Med. 1984;35:535-60. doi: 10.1146/annurev.me.35.020184.002535. PMID 6372671
- [Background] Farris RP, Cresanta JL, Frank GC, Webber LS, Berenson GS. Dietary studies of children from a biracial population: intakes of fat and fatty acids in 10- and 13-year olds. Am J Clin Nutr. 1984 Jan;39(1):114-28. doi: 10.1093/ajcn/39.1.114. PMID 6606974
- [Background] Cresanta JL, Srinivasan SR, Webber LS, Berenson GS. Serum lipid and lipoprotein cholesterol grids for cardiovascular risk screening of children. Am J Dis Child. 1984 Apr;138(4):379-87. doi: 10.1001/archpedi.1984.02140420045016. PMID 6702791
- [Background] Aristimuno GG, Foster TA, Voors AW, Srinivasan SR, Berenson GS. Influence of persistent obesity in children on cardiovascular risk factors: the Bogalusa Heart Study. Circulation. 1984 May;69(5):895-904. doi: 10.1161/01.cir.69.5.895. PMID 6705165
- [Background] Frank GC, Farris RP, Berenson GS. Comparison of dietary intake by 2 computerized analysis systems. J Am Diet Assoc. 1984 Jul;84(7):818-20. PMID 6736511
- [Background] Berenson GS, Webber LS, Srinivasan SR, Cresanta JL, Frank GC, Farris RP. Black-white contrasts as determinants of cardiovascular risk in childhood: precursors of coronary artery and primary hypertensive diseases. Am Heart J. 1984 Sep;108(3 Pt 2):672-83. doi: 10.1016/0002-8703(84)90654-9. PMID 6382995
- [Background] Wynder EL, Berenson GS. Preventive strategies for reducing hyperlipidemia in childhood. Prev Med. 1984 May;13(3):327-9. doi: 10.1016/0091-7435(84)90089-6. No abstract available. PMID 6494113
- [Background] Croft JB, Webber LS, Parker FC, Berenson GS. Recruitment and participation of children in a long-term study of cardiovascular disease: The Bogalusa Heart Study, 1973-1982. Am J Epidemiol. 1984 Sep;120(3):436-48. doi: 10.1093/oxfordjournals.aje.a113908. PMID 6332531
- [Background] Farris RP, Frank GC, Webber LS, Berenson GS: Quality Controls for Processing Dietary Data. J Diet Software, 1:3-4, 1984
- [Background] Farris RP, Frank GC, Berenson GS: Halt the Salt. J Nutr Ed, 16:174a, 1984
- [Background] Frank GC, Hollatz AT, Webber LS, Berenson GS. Effect of interviewer recording practices on nutrient intake--Bogalusa Heart Study. J Am Diet Assoc. 1984 Dec;84(12):1432-6, 1439. PMID 6501751
- [Background] Aristimuno GG, Foster TA, Berenson GS, Akman D. Subtle electrocardiographic changes in children with high levels of blood pressure. Am J Cardiol. 1984 Dec 1;54(10):1272-6. doi: 10.1016/s0002-9149(84)80079-x. PMID 6239535
- [Background] Farris RP, Frank GC, Webber LS, Berenson GS. A nutrition curriculum for families with high blood pressure. J Sch Health. 1985 Mar;55(3):110-2. doi: 10.1111/j.1746-1561.1985.tb04092.x. PMID 3845257
- [Background] Freedman DS, Srinivasan SR, Voors AW, Webber LS, Berenson GS. High density lipoprotein and coronary artery disease risk factors in children with different lipoprotein profiles: Bogalusa Heart Study. J Chronic Dis. 1985;38(4):327-38. doi: 10.1016/0021-9681(85)90079-7. PMID 3923013
- [Background] Borecki IB, Elston RC, Rosenbaum PA, Srinivasan SR, Berenson GS. ABO associations with blood pressure, serum lipids and lipoproteins, and anthropometric measures. Hum Hered. 1985;35(3):161-70. doi: 10.1159/000153537. PMID 3997161
- [Background] Freedman DS, Cresanta JL, Srinivasan SR, Webber LS, Berenson GS. Longitudinal serum lipoprotein changes in white males during adolescence: the Bogalusa Heart Study. Metabolism. 1985 Apr;34(4):396-403. doi: 10.1016/0026-0495(85)90231-8. PMID 3872400
- [Background] Hunter SM, Rosenbaum PA, Borecki IB, Elston RC, Berenson GS. A method to assess the environment for genetic studies: the Common Environment Index and the Household Relationships Interview. Am J Med Genet. 1985 Jun;21(2):325-35. doi: 10.1002/ajmg.1320210215. PMID 4014314
- [Background] Croft JB, Hunter SM, Webber LS, Watson RB, Berenson GS. Cigarette smoking behavioral distinctions between experimental nonadopters and adopters in children and adolescents--a consideration of transitional smoking experience: the Bogalusa Heart Study. Prev Med. 1985 Jan;14(1):109-22. doi: 10.1016/0091-7435(85)90026-x. PMID 3875850
- [Background] Frank GC, Farris RP, Cresanta JL, Webber LS, Berenson GS. Dietary trends of 10- and 13-year-old children in a biracial community--the Bogalusa Heart Study. Prev Med. 1985 Jan;14(1):123-39. doi: 10.1016/0091-7435(85)90027-1. PMID 3875851
- [Background] Webber LS, Berenson GS. Racial contrasts of blood pressure levels in two southern, rural communities. Prev Med. 1985 Jan;14(1):140-51. doi: 10.1016/0091-7435(85)90028-3. PMID 3875852
- [Background] Freedman DS, Burke GL, Harsha DW, Srinivasan SR, Cresanta JL, Webber LS, Berenson GS. Relationship of changes in obesity to serum lipid and lipoprotein changes in childhood and adolescence. JAMA. 1985 Jul 26;254(4):515-20. PMID 3859672
- [Background] Farris RP, Cresanta JL, Frank GC, Webber LS, Berenson GS. Dietary studies of children from a biracial population: intakes of carbohydrate and fiber in 10- and 13-year-olds. J Am Coll Nutr. 1985;4(4):421-35. doi: 10.1080/07315724.1985.10720085. PMID 2995472
- [Background] Farris RP, Frank GC, Webber LS, Berenson GS. A group method for obtaining dietary recalls of children. J Am Diet Assoc. 1985 Oct;85(10):1315-20. PMID 4045073
- [Background] Freedman DS, Shear CL, Srinivasan SR, Webber LS, Berenson GS. Tracking of serum lipids and lipoproteins in children over an 8-year period: the Bogalusa Heart Study. Prev Med. 1985 Mar;14(2):203-16. doi: 10.1016/0091-7435(85)90036-2. PMID 4048083
- [Background] Berenson GS. Epidemiologic investigations of cardiovascular risk factor variables in childhood--an overview. Acta Paediatr Scand Suppl. 1985;318:7-9. doi: 10.1111/j.1651-2227.1985.tb10078.x. No abstract available. PMID 3879094
- [Background] Farris RP, Cresanta JL, Webber LS, Frank GC, Berenson GS. Dietary studies of children from a biracial population: intakes of vitamins in 10- and 13-year-olds. J Am Coll Nutr. 1985;4(5):539-52. doi: 10.1080/07315724.1985.10720096. PMID 4056238
- [Background] Srinivasan SR, Hatano S, Matsuzaki T, Hollatz A, Webber LS, Berenson GS. Studies of serum lipoproteins of adolescent Japanese and U.S. (Bogalusa) children using a common laboratory. Prev Med. 1985 Sep;14(5):597-606. doi: 10.1016/0091-7435(85)90080-5. PMID 4070191
- [Background] Hunter SM, Parker FC, Williamson GD, Downey AM, Webber LS, Berenson GS. Measurement assessment of the type A coronary prone behavior pattern and hyperactivity/problem behaviors in children: are they related? The Bogalusa Heart Study. J Human Stress. 1985 Winter;11(4):177-83. doi: 10.1080/0097840X.1985.9936756. PMID 3843121
- [Background] Parker FC, Harsha DW, Farris RP, Webber LS, Frank GC, Berenson GS: Reducing the Risk of Cardiovascular Disease in Children. In: Self-Management of Chronic Disease (Holroyd K, Creer T, Eds). Orlando, FL: Academic Press, 1986
- [Background] Berenson GS, Frank GC: Racial (Black-White) Differences in Blood Pressure in Children. In: Potassium in Cardiovascular and Renal Medicine: Arrhythmias, Myocardial Infarction, and Hypertension (Whelton PK, Whelton A, Walker WG, Eds). New York: Marcel Dekker, Inc., p. 365-380, 1986
- [Background] Newman WP 3rd, Freedman DS, Voors AW, Gard PD, Srinivasan SR, Cresanta JL, Williamson GD, Webber LS, Berenson GS. Relation of serum lipoprotein levels and systolic blood pressure to early atherosclerosis. The Bogalusa Heart Study. N Engl J Med. 1986 Jan 16;314(3):138-44. doi: 10.1056/NEJM198601163140302. PMID 3455748
- [Background] Nicklas TA, Johnson CC, Arbeit ML, Franklin FA, Berenson GS. A dynamic family approach for the prevention of cardiovascular disease. J Am Diet Assoc. 1988 Nov;88(11):1438-40. PMID 3183267
- [Background] Berenson GS, Wattigney W, Newman WP III, Tracy RE, Srinivasan SR, Webber LS: Relationship of Atherosclerosis and Risk Factors in Young Adults: Racial, Sex, and Anatomic Contrasts. The Bogalusa Heart Study. Symposium on Hypertension and Atherosclerosis CIC. Edizioni Internazionali, 1988
- [Background] Burke GL, Hunter SM, Croft JB, Cresanta JL, Berenson GS. The interaction of alcohol and tobacco use in adolescents and young adults: Bogalusa Heart Study. Addict Behav. 1988;13(4):387-93. doi: 10.1016/0306-4603(88)90046-9. PMID 3239471
- [Background] Soto LF, Kikuchi DA, Arcilla RA, Savage DD, Berenson GS. Echocardiographic functions and blood pressure levels in children and young adults from a biracial population: the Bogalusa Heart Study. Am J Med Sci. 1989 May;297(5):271-9. doi: 10.1097/00000441-198905000-00001. PMID 2719054
- [Background] Nicklas TA, Webber LS, Thompson B, Berenson GS. A multivariate model for assessing eating patterns and their relationship to cardiovascular risk factors: the Bogalusa Heart Study. Am J Clin Nutr. 1989 Jun;49(6):1320-7. doi: 10.1093/ajcn/49.6.1320. PMID 2729171
- [Background] Chiang YK, Srinivasan SR, Webber LS, Berenson GS. Relationship between change in height and changes in serum lipid and lipoprotein levels in adolescent males: the Bogalusa Heart Study. J Clin Epidemiol. 1989;42(5):409-15. doi: 10.1016/0895-4356(89)90129-7. PMID 2786556
- [Background] Johnson CC, Hunter SM, Amos CI, Elder ST, Berenson GS. Cigarette smoking, alcohol, and oral contraceptive use by type A adolescent--the Bogalusa Heart Study. J Behav Med. 1989 Feb;12(1):13-24. doi: 10.1007/BF00844746. PMID 2746640
- [Background] Srinivasan SR, Wattigney W, Webber LS, Berenson GS. Relation of cholesterol to apolipoprotein B in low density lipoproteins of children. The Bogalusa Heart Study. Arteriosclerosis. 1989 Jul-Aug;9(4):493-500. doi: 10.1161/01.atv.9.4.493. PMID 2751478
- [Background] Dennison BA, Kikuchi DA, Srinivasan SR, Webber LS, Berenson GS. Parental history of cardiovascular disease as an indication for screening for lipoprotein abnormalities in children. J Pediatr. 1989 Aug;115(2):186-94. doi: 10.1016/s0022-3476(89)80063-0. PMID 2754548
- [Background] Berenson GS, Srinivasan SR, Wattigney W, Webber LS, Newman WP 3rd, Tracy RE. Insight into a bad omen for white men: coronary artery disease--the Bogalusa Heart Study. Am J Cardiol. 1989 Aug 2;64(6):32C-39C. doi: 10.1016/0002-9149(89)90681-4. PMID 2756897
- [Background] Berenson GS, Lawrence M, Soto L. The heart and hypertension in childhood. Semin Nephrol. 1989 Sep;9(3):236-46. No abstract available. PMID 2675242
- [Background] Downey AM, Cresanta JL, Berenson GS. Cardiovascular health promotion in children: "Heart Smart" and the changing role of physicians. Am J Prev Med. 1989 Sep-Oct;5(5):279-95. PMID 2675942
- [Background] Berenson GS, Srinivasan SR, Hunter SM, Nicklas TA, Freedman DS, Shear CL, Webber LS. Risk factors in early life as predictors of adult heart disease: the Bogalusa Heart Study. Am J Med Sci. 1989 Sep;298(3):141-51. doi: 10.1097/00000441-198909000-00001. PMID 2679086
- [Background] Amos CI, Cohen JC, Srinivasan SR, Freedman DS, Elston RC, Berenson GS. Polymorphism in the 5'-flanking region of the insulin gene and its potential relation to cardiovascular disease risk: observations in a biracial community. The Bogalusa Heart Study. Atherosclerosis. 1989 Sep;79(1):51-7. doi: 10.1016/0021-9150(89)90033-6. PMID 2679572
- [Background] Freedman DS, Srinivasan SR, Harsha DW, Webber LS, Berenson GS. Relation of body fat patterning to lipid and lipoprotein concentrations in children and adolescents: the Bogalusa Heart Study. Am J Clin Nutr. 1989 Nov;50(5):930-9. doi: 10.1093/ajcn/50.5.930. PMID 2816800
- [Background] Srinivasan SR, Wattigney W, Webber LS, Berenson GS. Serum apolipoprotein E in children and adolescents: the Bogalusa Heart Study. Metabolism. 1989 Dec;38(12):1173-8. doi: 10.1016/0026-0495(89)90155-8. PMID 2593831
- [Background] Berenson GS, Webber LS, Srinivasan SR. Pathogenesis of hypertension in black and white children. Clin Cardiol. 1989 Dec;12(12 Suppl 4):IV3-8. doi: 10.1002/clc.4960121303. PMID 2620471
- [Background] Berenson GS, Shear CL, Chiang YK, Webber LS, Voors AW. Combined low-dose medication and primary intervention over a 30-month period for sustained high blood pressure in childhood. Am J Med Sci. 1990 Feb;299(2):79-86. doi: 10.1097/00000441-199002000-00001. PMID 2301454
- [Background] Dennison BA, Kikuchi DA, Srinivasan SR, Webber LS, Berenson GS. Serum total cholesterol screening for the detection of elevated low-density lipoprotein in children and adolescents: the Bogalusa Heart Study. Pediatrics. 1990 Apr;85(4):472-9. PMID 2314959
- [Background] Berenson GS, Srinivasan SR, Nicklas TA, Johnson CC. Prevention of adult heart disease beginning in the pediatric age. Cardiovasc Clin. 1990;20(3):21-45. PMID 2186863
- [Background] Dennison BA, Kikuchi DA, Srinivasan SR, Webber LS, Berenson GS. Measurement of apolipoprotein B as a screening test for identifying children with elevated levels of low-density lipoprotein cholesterol. J Pediatr. 1990 Sep;117(3):358-63. doi: 10.1016/s0022-3476(05)81073-x. PMID 2391590
- [Background] Agamah ES, Webber LS, Lawrence M, Wattigney W, Berenson GS. Serum creatinine and its relation to cardiovascular disease risk variables in children and young adults from a biracial community. The Bogalusa Heart Study. J Lab Clin Med. 1990 Sep;116(3):327-34. PMID 2401847
- [Background] Cardiovascular Profile of 15,000 Children of School Age in Three Communities, 1971-1975. National Heart, Lung, and Blood Institute DHEW Publication No. (NIH) 78-1472, 1978
- [Background] Berenson GS, McMahan CA, Voors AW, Webber LS, Srinivasan SR, Frank GC, Foster TA, Blonde CV: Cardiovascular Risk Factors in Children - The Early Natural History of Atherosclerosis and Essential Hypertension (editorial assistance: C. Andrews and H.E. Hester) New York, Oxford Univ. Press, p. 450, 1980
- [Background] Berenson GS, Blonde CV, Webber LS (Eds): Monograph. Cardiovascular-Profile of Preschool Children in a Biracial Community (Bogalusa, Louisiana) - Bogalusa Heart Study, 1974. New Orleans: Louisiana State University Specialized Center of Research - Arteriosclerosis (SCOR-A). Library of Congress No. 81-52250, 1981
- [Background] Berenson GS (Eds): Causation of Cardiovascular Risk Factors in Children: Perspectives on Cardiovascular Risk in Early Life. New York: Raven Press, p. 408, 1986
- [Background] Frank GC, Webber LS, Farris RP, Berenson GS (Eds): Dietary Data Book: Quantifying Dietary Intakes of Infants, Children and Adolescents - The Bogalusa Heart Study, 1973-1983. From the Nutrition Core and Planning and Analysis Core Components of the National Research and Demonstration Center - Arteriosclerosis (NRDC-A). New Orleans: Louisiana State University Medical Center. Library of Congress Catalog Card No. 86-51215, 1986
- [Background] Farris RP, Frank GC, Ditmarsen P, Berenson GS: Sodium Sense Curriculum: A Dietary Alteration Program Trial (ADAPT). New Orleans: LSU Medical Center. Library of Congress Catalog Card No. 86-82603, 1986
- [Background] Hetzel BS, Berenson GS (Eds): Cardiovascular Risk Factors in Childhood: Epidemiology and Prevention. Amsterdam: Elsevier Science Publishers, B.V., 1987
- [Background] Srinivasan SR, Webber LS, Berenson GS: Factors Influencing Serum Lipoprotein Levels in Children. In: Atherosclerosis: A Pediatric Perspective, (Subbiah MTR, Ed). CRC Press, Inc., 1989.
- [Background] Srinivasan SR, Dahlen GH, Jarpa RA, Webber LS, Berenson GS. Racial (black-white) differences in serum lipoprotein (a) distribution and its relation to parental myocardial infarction in children. Bogalusa Heart Study. Circulation. 1991 Jul;84(1):160-7. doi: 10.1161/01.cir.84.1.160. PMID 1829398
- [Background] Srinivasan SR, Wattigney W, Webber LS, Berenson GS. Race and gender differences in serum lipoproteins of children, adolescents, and young adults--emergence of an adverse lipoprotein pattern in white males: the Bogalusa Heart Study. Prev Med. 1991 Nov;20(6):671-84. doi: 10.1016/0091-7435(91)90063-a. PMID 1766940
- [Background] Wattigney WA, Harsha DW, Srinivasan SR, Webber LS, Berenson GS. Increasing impact of obesity on serum lipids and lipoproteins in young adults. The Bogalusa Heart Study. Arch Intern Med. 1991 Oct;151(10):2017-22. PMID 1929690
- [Background] Agamah ES, Srinivasan SR, Webber LS, Berenson GS. Serum uric acid and its relation to cardiovascular disease risk factors in children and young adults from a biracial community: the Bogalusa Heart Study. J Lab Clin Med. 1991 Sep;118(3):241-9. PMID 1919297
- [Background] Lawrence M, Arbeit M, Johnson CC, Berenson GS. Prevention of adult heart disease beginning in childhood: intervention programs. Cardiovasc Clin. 1991;21(3):249-62. PMID 2044108
- [Background] Strong JP. The natural history of atherosclerosis in childhood. Ann N Y Acad Sci. 1991;623:9-15. doi: 10.1111/j.1749-6632.1991.tb43714.x. No abstract available. PMID 2042878
- [Background] Newman WP 3rd, Wattigney W, Berenson GS. Autopsy studies in United States children and adolescents. Relationship of risk factors to atherosclerotic lesions. Ann N Y Acad Sci. 1991;623:16-25. doi: 10.1111/j.1749-6632.1991.tb43715.x. No abstract available. PMID 2042824
- [Background] Webber LS, Hunter SM, Johnson CC, Srinivasan SR, Berenson GS. Smoking, alcohol, and oral contraceptives. Effects on lipids during adolescence and young adulthood--Bogalusa Heart Study. Ann N Y Acad Sci. 1991;623:135-54. doi: 10.1111/j.1749-6632.1991.tb43725.x. No abstract available. PMID 2042822
- [Background] Webber LS, Srinivasan SR, Wattigney WA, Berenson GS. Tracking of serum lipids and lipoproteins from childhood to adulthood. The Bogalusa Heart Study. Am J Epidemiol. 1991 May 1;133(9):884-99. doi: 10.1093/oxfordjournals.aje.a115968. PMID 2028978
- [Background] Vijayagopal P, Srinivasan SR, Radhakrishnamurthy B, Berenson GS. Factors regulating the metabolism of low-density lipoprotein-proteoglycan complex in macrophages. Biochim Biophys Acta. 1990 Feb 6;1042(2):204-9. doi: 10.1016/0005-2760(90)90009-m. PMID 2302422
- [Background] Nicklas TA, Arbeit ML, Srinivasan SR, Berenson GS. Cardiovascular risk factors in children and prevention of adult atherosclerosis. Bol Asoc Med P R. 1991 Nov;83(11):502-4. No abstract available. PMID 1811600
- [Background] Mott DS, Virgilio SJ, Warren BL, Berenson GS. Effectiveness of a personalized fitness module on knowledge, attitude, and cardiovascular endurance of fifth-grade students: "heart smart". Percept Mot Skills. 1991 Dec;73(3 Pt 1):847-58. doi: 10.2466/pms.1991.73.3.847. PMID 1792133
- [Background] Nicklas TA, Arbeit ML, Berenson GS. Dietary studies in children: cardiovascular disease prevention: the Bogalusa Heart Study. Compr Ther. 1991 Oct;17(10):8-15. No abstract available. PMID 1764895
- [Background] Johnson CC, Nicklas TA, Arbeit ML, Harsha DW, Mott DS, Hunter SM, Wattigney W, Berenson GS. Cardiovascular intervention for high-risk families: the Heart Smart Program. South Med J. 1991 Nov;84(11):1305-12. doi: 10.1097/00007611-199111000-00004. PMID 1948212
- [Background] Nicklas TA, Webber LS, Berenson GS. Studies of consistency of dietary intake during the first four years of life in a prospective analysis: Bogalusa Heart Study. J Am Coll Nutr. 1991 Jun;10(3):234-41. doi: 10.1080/07315724.1991.10718150. PMID 1894881
- [Background] Berenson GS, Arbeit ML, Hunter SM, Johnson CC, Nicklas TA. Cardiovascular health promotion for elementary school children. The Heart Smart Program. Ann N Y Acad Sci. 1991;623:299-313. doi: 10.1111/j.1749-6632.1991.tb43739.x. PMID 2042838
- [Background] Nicklas TA, Forcier JE, Webber LS, Berenson GS. School lunch assessment to improve accuracy of 24-hour dietary recall for children. J Am Diet Assoc. 1991 Jun;91(6):711-3. No abstract available. PMID 2040787
- [Background] Webber LS, Harsha DW, Phillips GT, Srinivasan SR, Simpson JW, Berenson GS. Cardiovascular risk factors in Hispanic, white, and black children: the Brooks County and Bogalusa Heart studies. Am J Epidemiol. 1991 Apr 1;133(7):704-14. doi: 10.1093/oxfordjournals.aje.a115945. PMID 2018025
- [Background] Amos CI, Elston RC, Bonney GE, Keats BJ, Berenson GS. A multivariate method for detecting genetic linkage, with application to a pedigree with an adverse lipoprotein phenotype. Am J Hum Genet. 1990 Aug;47(2):247-54. PMID 2378349
- [Background] Tracy RE, Berenson G, Wattigney W, Barrett TJ. The evolution of benign arterionephrosclerosis from age 6 to 70 years. Am J Pathol. 1990 Feb;136(2):429-39. PMID 2305836
- [Background] Jiang X, Srinivasan SR, Urbina E, Berenson GS. Hyperdynamic circulation and cardiovascular risk in children and adolescents. The Bogalusa Heart Study. Circulation. 1995 Feb 15;91(4):1101-6. doi: 10.1161/01.cir.91.4.1101. PMID 7850947
- [Background] Jiang X, Srinivasan SR, Radhakrishnamurthy B, Dalferes ER Jr, Bao W, Berenson GS. Microalbuminuria in young adults related to blood pressure in a biracial (black-white) population. The Bogalusa Heart Study. Am J Hypertens. 1994 Sep;7(9 Pt 1):794-800. doi: 10.1093/ajh/7.9.794. PMID 7811437
- [Background] Jiang X, Srinivasan SR, Webber LS, Wattigney WA, Berenson GS. Association of fasting insulin level with serum lipid and lipoprotein levels in children, adolescents, and young adults: the Bogalusa Heart Study. Arch Intern Med. 1995 Jan 23;155(2):190-6. PMID 7811129
- [Background] Bao W, Srinivasan SR, Wattigney WA, Berenson GS. The relation of parental cardiovascular disease to risk factors in children and young adults. The Bogalusa Heart Study. Circulation. 1995 Jan 15;91(2):365-71. doi: 10.1161/01.cir.91.2.365. PMID 7805239
- [Background] Bao W, Srinivasan SR, Wattigney WA, Berenson GS. Persistence of multiple cardiovascular risk clustering related to syndrome X from childhood to young adulthood. The Bogalusa Heart Study. Arch Intern Med. 1994 Aug 22;154(16):1842-7. PMID 8053753
- [Background] Srinivasan SR, Bao W, Berenson GS. The amount of cholesterol relative to apolipoprotein B in low-density lipoproteins relates primarily to high-density lipoprotein cholesterol in children: the Bogalusa Heart Study. Metabolism. 1994 Aug;43(8):1042-6. doi: 10.1016/0026-0495(94)90187-2. PMID 8052145
- [Background] Srinivasan SR, Ehnholm C, Wattigney WA, Berenson GS. Relationship between obesity and serum lipoproteins in children with different apolipoprotein E phenotypes: the Bogalusa Heart Study. Metabolism. 1994 Apr;43(4):470-5. doi: 10.1016/0026-0495(94)90079-5. PMID 8159106
- [Background] Freedman DS, Wattigney WA, Srinivasan S, Newman WP 3rd, Tracy RE, Byers T, Berenson GS. The relation of atherosclerotic lesions to antemortem and postmortem lipid levels: the Bogalusa Heart Study. Atherosclerosis. 1993 Dec;104(1-2):37-46. doi: 10.1016/0021-9150(93)90174-s. PMID 8141849
- [Background] Jiang X, Srinivasan SR, Bao W, Berenson GS. Association of fasting insulin with longitudinal changes in blood pressure in children and adolescents. The Bogalusa Heart Study. Am J Hypertens. 1993 Jul;6(7 Pt 1):564-9. doi: 10.1093/ajh/6.7.564. PMID 8397996
- [Background] Bao W, Srinivasan SR, Berenson GS. Tracking of serum apolipoproteins A-I and B in children and young adults: the Bogalusa Heart Study. J Clin Epidemiol. 1993 Jul;46(7):609-16. doi: 10.1016/0895-4356(93)90033-w. PMID 8326345
- [Background] Berenson GS, Dalferes E Jr, Savage D, Webber LS, Bao W. Ambulatory blood pressure measurements in children and young adults selected by high and low casual blood pressure levels and parental history of hypertension: the Bogalusa Heart Study. Am J Med Sci. 1993 Jun;305(6):374-82. doi: 10.1097/00000441-199306000-00004. PMID 8506897
- [Background] Srinivasan SR, Ehnholm C, Wattigney W, Berenson GS. Apolipoprotein E polymorphism and its association with serum lipoprotein concentrations in black versus white children: the Bogalusa Heart Study. Metabolism. 1993 Mar;42(3):381-6. doi: 10.1016/0026-0495(93)90091-2. PMID 8487659
- [Background] Rautaharju PM, Zhou SH, Wong S, Calhoun HP, Berenson GS, Prineas R, Davignon A. Sex differences in the evolution of the electrocardiographic QT interval with age. Can J Cardiol. 1992 Sep;8(7):690-5. PMID 1422988
- [Background] Richards RJ, Svec F, Bao W, Srinivasan SR, Berenson GS. Steroid hormones during puberty: racial (black-white) differences in androstenedione and estradiol--the Bogalusa Heart Study. J Clin Endocrinol Metab. 1992 Aug;75(2):624-31. doi: 10.1210/jcem.75.2.1639961.
- [Background] Ciolino HP, Vijayagopal P, Radhakrishnamurthy B, Berenson GS. Heparin stimulates proteoglycan synthesis by vascular smooth muscle cells while suppressing cellular proliferation. Atherosclerosis. 1992 Jun;94(2-3):135-46. doi: 10.1016/0021-9150(92)90238-c. PMID 1632867
- [Background] Kikuchi DA, Srinivasan SR, Harsha DW, Webber LS, Sellers TA, Berenson GS. Relation of serum lipoprotein lipids and apolipoproteins to obesity in children: the Bogalusa Heart Study. Prev Med. 1992 Mar;21(2):177-90. doi: 10.1016/0091-7435(92)90017-c. PMID 1579553
- [Background] Svec F, Nastasi K, Hilton C, Bao W, Srinivasan SR, Berenson GS. Black-white contrasts in insulin levels during pubertal development. The Bogalusa Heart Study. Diabetes. 1992 Mar;41(3):313-7. doi: 10.2337/diab.41.3.313. PMID 1551490
- [Background] Williams DP, Going SB, Lohman TG, Harsha DW, Srinivasan SR, Webber LS, Berenson GS. Body fatness and risk for elevated blood pressure, total cholesterol, and serum lipoprotein ratios in children and adolescents. Am J Public Health. 1992 Mar;82(3):358-63. doi: 10.2105/ajph.82.3.358. PMID 1536350
- [Background] Nicklas TA, Farris RP, Myers L, Berenson GS. Impact of meat consumption on nutritional quality and cardiovascular risk factors in young adults: the Bogalusa Heart Study. J Am Diet Assoc. 1995 Aug;95(8):887-92. doi: 10.1016/S0002-8223(95)00246-4. PMID 7636079
- [Background] Johnson CC, Myers L, Webber LS, Hunter SM, Srinivasan SR, Berenson GS. Alcohol consumption among adolescents and young adults: the Bogalusa Heart Study, 1981 to 1991. Am J Public Health. 1995 Jul;85(7):979-82. doi: 10.2105/ajph.85.7.979. PMID 7604924
- [Background] Urbina EM, Gidding SS, Bao W, Pickoff AS, Berdusis K, Berenson GS. Effect of body size, ponderosity, and blood pressure on left ventricular growth in children and young adults in the Bogalusa Heart Study. Circulation. 1995 May 1;91(9):2400-6. doi: 10.1161/01.cir.91.9.2400. PMID 7729027
- [Background] Nicklas TA, Farris RP, Myers L, Berenson GS. Dietary fiber intake of children and young adults: the Bogalusa Heart Study. J Am Diet Assoc. 1995 Feb;95(2):209-14. doi: 10.1016/S0002-8223(95)00049-6. PMID 7852687
- [Background] Srinivasan SR, Berenson GS. Serum apolipoproteins A-I and B as markers of coronary artery disease risk in early life: the Bogalusa Heart Study. Clin Chem. 1995 Jan;41(1):159-64. PMID 7813072
- [Background] Laing AE, Amos CI, DeMeester C, Diep A, Xia YR, Elston RC, Srinivasan SR, Berenson GS, Lusis AJ. Linkage between the APOB gene and serum ApoB levels in a large pedigree from the Bogalusa Heart Study. Genet Epidemiol. 1994;11(1):29-40. doi: 10.1002/gepi.1370110104. PMID 7912214
- [Background] Berenson GS, Wattigney WA, Bao W, Nicklas TA, Jiang X, Rush JA. Epidemiology of early primary hypertension and implications for prevention: the Bogalusa Heart Study. J Hum Hypertens. 1994 May;8(5):303-11. PMID 8064774
- [Background] Nicklas TA, Myers L, Berenson GS. Impact of ready-to-eat cereal consumption on total dietary intake of children: the Bogalusa Heart Study. J Am Diet Assoc. 1994 Mar;94(3):316-8. doi: 10.1016/0002-8223(94)90377-8. No abstract available. PMID 8120300
- [Background] Bao W, Dalferes ER Jr, Srinivasan SR, Webber LS, Berenson GS. Normative distribution of complete blood count from early childhood through adolescence: the Bogalusa Heart Study. Prev Med. 1993 Nov;22(6):825-37. doi: 10.1006/pmed.1993.1075. PMID 8115341
- [Background] Heiba IM, DeMeester CA, Xia YR, Diep A, George VT, Amos CI, Srinivasan SR, Berenson GS, Elston RC, Lusis AJ. Genetic contributions to quantitative lipoprotein traits associated with coronary artery disease: analysis of a large pedigree from the Bogalusa Heart Study. Am J Med Genet. 1993 Nov 1;47(6):875-83. doi: 10.1002/ajmg.1320470615. PMID 8279486
- [Background] Nicklas TA, Bao W, Webber LS, Berenson GS. Breakfast consumption affects adequacy of total daily intake in children. J Am Diet Assoc. 1993 Aug;93(8):886-91. doi: 10.1016/0002-8223(93)91527-w. PMID 8335868
- [Background] Nicklas TA, Webber LS, Srinivasan SR, Berenson GS. Secular trends in dietary intakes and cardiovascular risk factors of 10-y-old children: the Bogalusa Heart Study (1973-1988). Am J Clin Nutr. 1993 Jun;57(6):930-7. doi: 10.1093/ajcn/57.6.930. PMID 8503364
- [Background] Srinivasan SR, Powers CR, Webber LS, Berenson GS. Serum lipids and lipoprotein profiles of military personnel and their families: Fort Polk Heart Smart Program. Mil Med. 1993 May;158(5):323-6. PMID 8502396
- [Background] Johnson CC, Harsha DW, Powers CR, Webber LS, Berenson GS. Fort Polk Heart Smart Program. Part IV: Lifestyles of military personnel and their families. Mil Med. 1993 May;158(5):317-22. PMID 8502395
- [Background] Nicklas TA, Webber LS, Kern SL, Powers CR, Harsha DW, Berenson GS. Fort Polk Heart Smart Program. Part III: Assessment of dietary intake of military wives. Mil Med. 1993 May;158(5):312-6. PMID 8502394
- [Background] Webber LS, Srinivasan SR, Harsha DW, Powers CR, Berenson GS. Fort Polk Heart Smart Program. Part II: Cardiovascular risk factor assessment. Mil Med. 1993 May;158(5):308-11. PMID 8502393
- [Background] Berenson GS, Schnakenberg D, Harsha DW, Webber LS, Johnson CC, Nicklas TA, Srinivasan SR. Fort Polk Heart Smart Program. Part I: Background design and significance. Mil Med. 1993 May;158(5):304-8. PMID 8502392
- [Background] Bao W, Srinivasan SR, Berenson GS. Plasma fibrinogen and its correlates in children from a biracial community: the Bogalusa Heart Study. Pediatr Res. 1993 Apr;33(4 Pt 1):323-6. doi: 10.1203/00006450-199304000-00003. PMID 8479809
- [Background] Rautaharju PM, Zhou SH, Wong S, Prineas R, Berenson GS. Functional characteristics of QT prediction formulas. The concepts of QTmax and QT rate sensitivity. Comput Biomed Res. 1993 Apr;26(2):188-204. doi: 10.1006/cbmr.1993.1012. PMID 8477589
- [Background] Radhakrishnamurthy B, Jeansonne N, Tracy RE, Berenson GS. A monoclonal antibody that recognizes hyaluronic acid binding region of aorta proteoglycans. Atherosclerosis. 1993 Jan 25;98(2):179-92. doi: 10.1016/0021-9150(93)90127-g. PMID 7681290
- [Background] Berenson GS. Cholesterol. Myth vs reality in pediatric practice. Am J Dis Child. 1993 Apr;147(4):371-3. doi: 10.1001/archpedi.1993.02160280021010. No abstract available. PMID 8456789
- [Background] Jiang X, Srinivasan SR, Bao W, Berenson GS. Association of fasting insulin with blood pressure in young individuals. The Bogalusa Heart Study. Arch Intern Med. 1993 Feb 8;153(3):323-8. PMID 8427537
- [Background] Berenson GS, Wattigney WA, Tracy RE, Newman WP 3rd, Srinivasan SR, Webber LS, Dalferes ER Jr, Strong JP. Atherosclerosis of the aorta and coronary arteries and cardiovascular risk factors in persons aged 6 to 30 years and studied at necropsy (The Bogalusa Heart Study). Am J Cardiol. 1992 Oct 1;70(9):851-8. doi: 10.1016/0002-9149(92)90726-f. PMID 1529936
- [Background] Farris RP, Nicklas TA, Webber LS, Berenson GS. Nutrient contribution of the school lunch program: implications for healthy people 2000. J Sch Health. 1992 May;62(5):180-4. doi: 10.1111/j.1746-1561.1992.tb06038.x. PMID 1522699
- [Background] Tracy RE, Berenson GS, Cueto-Garcia L, Wattigney WA, Barrett TJ. Nephrosclerosis and aortic atherosclerosis from age 6 to 70 years in the United States and Mexico. Virchows Arch A Pathol Anat Histopathol. 1992;420(6):479-88. doi: 10.1007/BF01600252. PMID 1609508
- [Background] Arbeit ML, Nicklas TA, Berenson GS. Considerations of dietary sodium/potassium/energy ratios of selected foods. J Am Coll Nutr. 1992 Apr;11(2):210-22. PMID 1578099
- [Background] Srinivasan SR, Berenson GS. Serum lipids and lipoproteins in children. Pediatr Ann. 1992 Apr;21(4):220-3. doi: 10.3928/0090-4481-19920401-10. No abstract available. PMID 1561001
- [Background] Johnson CC, Nicklas TA, Arbeit ML, Webber LS, Berenson GS. Behavioral counseling and contracting as methods for promoting cardiovascular health in families. J Am Diet Assoc. 1992 Apr;92(4):479-81. No abstract available. PMID 1556350
- [Background] Frank GC, Nicklas TA, Webber LS, Major C, Miller JF, Berenson GS. A food frequency questionnaire for adolescents: defining eating patterns. J Am Diet Assoc. 1992 Mar;92(3):313-8. PMID 1552130
- [Background] Vijayagopal P, Srinivasan SR, Radhakrishnamurthy B, Berenson GS. Lipoprotein-proteoglycan complexes from atherosclerotic lesions promote cholesteryl ester accumulation in human monocytes/macrophages. Arterioscler Thromb. 1992 Feb;12(2):237-49. doi: 10.1161/01.atv.12.2.237. PMID 1543697
- [Background] Arbeit ML, Johnson CC, Mott DS, Harsha DW, Nicklas TA, Webber LS, Berenson GS. The Heart Smart cardiovascular school health promotion: behavior correlates of risk factor change. Prev Med. 1992 Jan;21(1):18-32. doi: 10.1016/0091-7435(92)90003-z. PMID 1738766
- [Background] Nicklas TA, Webber LS, Koschak M, Berenson GS. Nutrient adequacy of low fat intakes for children: the Bogalusa Heart Study. Pediatrics. 1992 Feb;89(2):221-8. PMID 1734388
- [Background] Srinivasan SR, Ehnholm C, Wattigney WA, Bao W, Berenson GS. The relation of apolipoprotein E polymorphism to multiple cardiovascular risk in children: the Bogalusa Heart Study. Atherosclerosis. 1996 Jun;123(1-2):33-42. doi: 10.1016/0021-9150(95)05762-5. PMID 8782835
- [Background] Jiang X, Srinivasan SR, Berenson GS. Relation of obesity to insulin secretion and clearance in adolescents: the Bogalusa Heart Study. Int J Obes Relat Metab Disord. 1996 Oct;20(10):951-6. PMID 8910101
- [Background] Edupuganti S, Svec F, Bao W, Srinivasan SR, Berenson GS. Thyroid function in children with different lipoprotein profiles: observations in a biracial (black/white) population--the Bogalusa Heart Study. Am J Med Sci. 1997 Feb;313(2):80-4. doi: 10.1097/00000441-199702000-00002. PMID 9030672
- [Background] Donker GA, Labarthe DR, Harrist RB, Selwyn BJ, Wattigney W, Berenson GS. Low birth weight and blood pressure at age 7-11 years in a biracial sample. Am J Epidemiol. 1997 Mar 1;145(5):387-97. doi: 10.1093/oxfordjournals.aje.a009120. PMID 9048512
- [Background] Gustat J, Elkasabany A, Srinivasan S, Berenson GS. Relation of abdominal height to cardiovascular risk factors in young adults: the Bogalusa heart study. Am J Epidemiol. 2000 May 1;151(9):885-91. doi: 10.1093/oxfordjournals.aje.a010292. PMID 10791561
- [Background] Freedman DS, Kettel-Khan L, Srinivasan SR, Berenson GS. Black/white differences in relative weight and obesity among girls: the Bogalusa Heart Study. Prev Med. 2000 Mar;30(3):234-43. doi: 10.1006/pmed.1999.0611. PMID 10684747
- [Background] Freedman DS, Khan LK, Serdula MK, Srinivasan SR, Berenson GS. Secular trends in height among children during 2 decades: The Bogalusa Heart Study. Arch Pediatr Adolesc Med. 2000 Feb;154(2):155-61. doi: 10.1001/archpedi.154.2.155. PMID 10665602
- [Background] Chen W, Srinivasan SR, Elkasabany A, Berenson GS. Cardiovascular risk factors clustering features of insulin resistance syndrome (Syndrome X) in a biracial (Black-White) population of children, adolescents, and young adults: the Bogalusa Heart Study. Am J Epidemiol. 1999 Oct 1;150(7):667-74. doi: 10.1093/oxfordjournals.aje.a010069. PMID 10512420
- [Background] Chen W, Srinivasan SR, Elkasabany A, Berenson GS. The association of cardiovascular risk factor clustering related to insulin resistance syndrome (Syndrome X) between young parents and their offspring: the Bogalusa Heart Study. Atherosclerosis. 1999 Jul;145(1):197-205. doi: 10.1016/s0021-9150(99)00025-8. PMID 10428311
- [Background] Srinivasan SR, Myers L, Berenson GS. Temporal association between obesity and hyperinsulinemia in children, adolescents, and young adults: the Bogalusa Heart Study. Metabolism. 1999 Jul;48(7):928-34. doi: 10.1016/s0026-0495(99)90231-7. PMID 10421238
- [Background] Wattigney WA, Srinivasan SR, Chen W, Greenlund KJ, Berenson GS. Secular trend of earlier onset of menarche with increasing obesity in black and white girls: the Bogalusa Heart Study. Ethn Dis. 1999 Spring-Summer;9(2):181-9. PMID 10421080
- [Background] Urbina EM, Gidding SS, Bao W, Elkasabany A, Berenson GS. Association of fasting blood sugar level, insulin level, and obesity with left ventricular mass in healthy children and adolescents: The Bogalusa Heart Study. Am Heart J. 1999 Jul;138(1 Pt 1):122-7. doi: 10.1016/s0002-8703(99)70256-5. PMID 10385774
- [Background] Freedman DS, Dietz WH, Srinivasan SR, Berenson GS. The relation of overweight to cardiovascular risk factors among children and adolescents: the Bogalusa Heart Study. Pediatrics. 1999 Jun;103(6 Pt 1):1175-82. doi: 10.1542/peds.103.6.1175. PMID 10353925
- [Background] Hunter SM, Webber LS, Elkasabany A, Berenson GS. Are some children and adolescents in Louisiana addicted to tobacco? The Bogalusa Heart Study. J La State Med Soc. 1999 Apr;151(4):177-81. PMID 10234892
- [Background] Greenlund KJ, Srinivasan SR, Xu JH, Dalferes E Jr, Myers L, Pickoff A, Berenson GS. Plasma homocysteine distribution and its association with parental history of coronary artery disease in black and white children: the Bogalusa Heart Study. Circulation. 1999 Apr 27;99(16):2144-9. doi: 10.1161/01.cir.99.16.2144. PMID 10217655
- [Background] Srinivasan SR, Ehnholm C, Elkasabany A, Berenson G. Influence of apolipoprotein E polymorphism on serum lipids and lipoprotein changes from childhood to adulthood: the Bogalusa Heart Study. Atherosclerosis. 1999 Apr;143(2):435-43. doi: 10.1016/s0021-9150(98)00304-9. PMID 10217374
- [Background] Freedman DS, Serdula MK, Srinivasan SR, Berenson GS. Relation of circumferences and skinfold thicknesses to lipid and insulin concentrations in children and adolescents: the Bogalusa Heart Study. Am J Clin Nutr. 1999 Feb;69(2):308-17. doi: 10.1093/ajcn/69.2.308. PMID 9989697
- [Background] Berenson GS, Srinivasan SR, Nicklas TA. Atherosclerosis: a nutritional disease of childhood. Am J Cardiol. 1998 Nov 26;82(10B):22T-29T. doi: 10.1016/s0002-9149(98)00719-x. PMID 9860370
- [Background] Farris RP, Nicklas TA, Myers L, Berenson GS. Nutrient intake and food group consumption of 10-year-olds by sugar intake level: the Bogalusa Heart Study. J Am Coll Nutr. 1998 Dec;17(6):579-85. doi: 10.1080/07315724.1998.10718806. PMID 9853537
- [Background] Srinivasan SR, Elkasabani A, Dalferes ER Jr, Bao W, Berenson GS. Characteristics of young offspring of type 2 diabetic parents in a biracial (black-white) community-based sample: the Bogalusa Heart Study. Metabolism. 1998 Aug;47(8):998-1004. doi: 10.1016/s0026-0495(98)90358-4. PMID 9711999
- [Background] Srinivasan SR, Elkasabany A, Berenson GS. Distribution and correlates of serum high-density lipoprotein subclasses (LpA-I and LpA-I:A-II) in children from a biracial community. The Bogalusa Heart Study. Metabolism. 1998 Jun;47(6):757-63. doi: 10.1016/s0026-0495(98)90042-7. PMID 9627378
- [Background] Berenson GS, Srinivasan SR, Bao W, Newman WP 3rd, Tracy RE, Wattigney WA. Association between multiple cardiovascular risk factors and atherosclerosis in children and young adults. The Bogalusa Heart Study. N Engl J Med. 1998 Jun 4;338(23):1650-6. doi: 10.1056/NEJM199806043382302. PMID 9614255
- [Background] Elkasabany AM, Urbina EM, Daniels SR, Berenson GS. Prediction of adult hypertension by K4 and K5 diastolic blood pressure in children: the Bogalusa Heart Study. J Pediatr. 1998 Apr;132(4):687-92. doi: 10.1016/s0022-3476(98)70361-0. PMID 9580771
- [Background] Nicklas TA, O'Neil CE, Berenson GS. Nutrient contribution of breakfast, secular trends, and the role of ready-to-eat cereals: a review of data from the Bogalusa Heart Study. Am J Clin Nutr. 1998 Apr;67(4):757S-763S. doi: 10.1093/ajcn/67.4.757S. PMID 9537625
- [Background] Urbina EM, Bao W, Pickoff AS, Berenson GS. Ethnic (black-white) contrasts in heart rate variability during cardiovascular reactivity testing in male adolescents with high and low blood pressure: the Bogalusa Heart Study. Am J Hypertens. 1998 Feb;11(2):196-202. doi: 10.1016/s0895-7061(97)00314-2. PMID 9524048
- [Background] Batten LA, Urbina EM, Berenson GS. Interobserver reproducibility of heart rate variability in children (the Bogalusa Heart Study). Am J Cardiol. 2000 Dec 1;86(11):1264-6, A9. doi: 10.1016/s0002-9149(00)01217-0. PMID 11090806
- [Background] Freedman DS, Bowman BA, Otvos JD, Srinivasan SR, Berenson GS. Levels and correlates of LDL and VLDL particle sizes among children: the Bogalusa heart study. Atherosclerosis. 2000 Oct;152(2):441-9. doi: 10.1016/s0021-9150(99)00495-5. PMID 10998473
- [Background] Youssef AA, Srinivasan SR, Elkasabany A, Cruickshank JK, Berenson GS. Temporal relation between blood pressure and serum creatinine in young adults from a biracial community: the Bogalusa Heart Study. Am J Hypertens. 2000 Jul;13(7):770-5. doi: 10.1016/s0895-7061(00)00233-8. PMID 10933568
- [Background] McClain MR, Srinivasan SR, Chen W, Steinmann WC, Berenson GS. Risk of type 2 diabetes mellitus in young adults from a biracial community: the Bogalusa Heart Study. Prev Med. 2000 Jul;31(1):1-7. doi: 10.1006/pmed.2000.0682. PMID 10896837
- [Background] Chen W, Bao W, Begum S, Elkasabany A, Srinivasan SR, Berenson GS. Age-related patterns of the clustering of cardiovascular risk variables of syndrome X from childhood to young adulthood in a population made up of black and white subjects: the Bogalusa Heart Study. Diabetes. 2000 Jun;49(6):1042-8. doi: 10.2337/diabetes.49.6.1042. PMID 10866058
- [Background] Srinivasan SR, Myers L, Berenson GS. Risk variables of insulin resistance syndrome in African-American and Caucasian young adults with microalbuminuria: the Bogalusa Heart Study. Am J Hypertens. 2000 Dec;13(12):1274-9. doi: 10.1016/s0895-7061(00)01220-6. PMID 11130771
- [Background] Srinivasan SR, Myers L, Berenson GS. Rate of change in adiposity and its relationship to concomitant changes in cardiovascular risk variables among biracial (black-white) children and young adults: The Bogalusa Heart Study. Metabolism. 2001 Mar;50(3):299-305. doi: 10.1053/meta.2001.21019. PMID 11230782
- [Background] Frontini MG, Srinivasan SR, Elkasabany A, Berenson GS. Distribution and cardiovascular risk correlates of serum triglycerides in young adults from a biracial community: the Bogalusa Heart Study. Atherosclerosis. 2001 Mar;155(1):201-9. doi: 10.1016/s0021-9150(00)00538-4. PMID 11223443
- [Background] Chen W, Srinivasan SR, Berenson GS. Plasma renin activity and insulin resistance in African American and white children: the Bogalusa Heart Study. Am J Hypertens. 2001 Mar;14(3):212-7. doi: 10.1016/s0895-7061(00)01274-7. PMID 11281231
- [Background] Frontini MG, Bao W, Elkasabany A, Srinivasan SR, Berenson G. Comparison of weight-for-height indices as a measure of adiposity and cardiovascular risk from childhood to young adulthood: the Bogalusa heart study. J Clin Epidemiol. 2001 Aug;54(8):817-22. doi: 10.1016/s0895-4356(01)00343-2. PMID 11470391
- [Background] Hallman DM, Srinivasan SR, Elkasabany A, Boerwinkle E, Berenson GS. The Ser(447)-Stop polymorphism of lipoprotein lipase is associated with variation in longitudinal serum high-density lipoprotein-cholesterol profiles: the Bogalusa Heart Study. Metabolism. 2001 Aug;50(8):894-904. doi: 10.1053/meta.2001.24918. PMID 11474476
- [Background] Srinivasan SR, Ehnholm C, Elkasabany A, Berenson GS. Apolipoprotein E polymorphism modulates the association between obesity and dyslipidemias during young adulthood: The Bogalusa Heart Study. Metabolism. 2001 Jun;50(6):696-702. doi: 10.1053/meta.2001.23299. PMID 11398147
- [Background] Nicklas TA, Elkasabany A, Srinivasan SR, Berenson G. Trends in nutrient intake of 10-year-old children over two decades (1973-1994) : the Bogalusa Heart Study. Am J Epidemiol. 2001 May 15;153(10):969-77. doi: 10.1093/aje/153.10.969. PMID 11384953
- [Background] Freedman DS, Kettel Khan L, Serdula MK, Srinivasan SR, Berenson GS. BMI rebound, childhood height and obesity among adults: the Bogalusa Heart Study. Int J Obes Relat Metab Disord. 2001 Apr;25(4):543-9. doi: 10.1038/sj.ijo.0801581. PMID 11319660
- [Background] Freedman DS, Khan LK, Dietz WH, Srinivasan SR, Berenson GS. Relationship of childhood obesity to coronary heart disease risk factors in adulthood: the Bogalusa Heart Study. Pediatrics. 2001 Sep;108(3):712-8. doi: 10.1542/peds.108.3.712. PMID 11533341
- [Background] Berenson GS; Bogalusa Heart Study Investigators. Bogalusa Heart Study: a long-term community study of a rural biracial (Black/White) population. Am J Med Sci. 2001 Nov;322(5):293-300. PMID 11876192
- [Background] Berenson GS, Srinivasan SR. Emergence of obesity and cardiovascular risk for coronary artery disease: the Bogalusa Heart Study. Prev Cardiol. 2001 Summer;4(3):116-121. doi: 10.1111/j.1520-037x.2001.00537.x. PMID 11828187
- [Background] Freedman DS, Khan LK, Mei Z, Dietz WH, Srinivasan SR, Berenson GS. Relation of childhood height to obesity among adults: the Bogalusa Heart Study. Pediatrics. 2002 Feb;109(2):E23. doi: 10.1542/peds.109.2.e23. PMID 11826233
- [Background] Srinivasan SR, Myers L, Berenson GS. Predictability of childhood adiposity and insulin for developing insulin resistance syndrome (syndrome X) in young adulthood: the Bogalusa Heart Study. Diabetes. 2002 Jan;51(1):204-9. doi: 10.2337/diabetes.51.1.204. PMID 11756342
- [Background] Youssef AA, Srinivasan SR, Elkasabany A, Chen W, Berenson GS. Trends of lipoprotein variables from childhood to adulthood in offspring of parents with coronary heart disease: the Bogalusa Heart Study. Metabolism. 2001 Dec;50(12):1441-6. doi: 10.1053/meta.2001.28076. PMID 11735090
- [Background] Srinivasan SR, Segrest JP, Elkasabany AM, Berenson GS. Distribution and correlates of lipoproteins and their subclasses in black and white young adults. The Bogalusa Heart Study. Atherosclerosis. 2001 Dec;159(2):391-7. doi: 10.1016/s0021-9150(01)00514-7. PMID 11730819
- [Background] Chen W, Srinivasan SR, Elkasabany A, Ellsworth DL, Boerwinkle E, Berenson GS. Influence of lipoprotein lipase serine 447 stop polymorphism on tracking of triglycerides and HDL cholesterol from childhood to adulthood and familial risk of coronary artery disease: the Bogalusa heart study. Atherosclerosis. 2001 Dec;159(2):367-73. doi: 10.1016/s0021-9150(01)00508-1. PMID 11730816
- [Background] Chen W, Srinivasan SR, Elkasabany A, Ellsworth DL, Boerwinkle E, Berenson GS. Combined effects of endothelial nitric oxide synthase gene polymorphism (G894T) and insulin resistance status on blood pressure and familial risk of hypertension in young adults: the Bogalusa Heart Study. Am J Hypertens. 2001 Oct;14(10):1046-52. doi: 10.1016/s0895-7061(01)02192-6. PMID 11710784
- [Background] Chen W, Srinivasan SR, Bao W, Berenson GS. The magnitude of familial associations of cardiovascular risk factor variables between parents and offspring are influenced by age: the Bogalusa Heart Study. Ann Epidemiol. 2001 Nov;11(8):522-8. doi: 10.1016/s1047-2797(01)00228-9. PMID 11709270
- [Background] Urbina EM, Brinton TJ, Elkasabany A, Berenson GS. Brachial artery distensibility and relation to cardiovascular risk factors in healthy young adults (The Bogalusa Heart Study). Am J Cardiol. 2002 Apr 15;89(8):946-51. doi: 10.1016/s0002-9149(02)02244-0. PMID 11950433
- [Background] Nicklas TA, von Duvillard SP, Berenson GS. Tracking of serum lipids and lipoproteins from childhood to dyslipidemia in adults: the Bogalusa Heart Study. Int J Sports Med. 2002 May;23 Suppl 1:S39-43. doi: 10.1055/s-2002-28460. PMID 12012261
- [Background] Freedman DS, Bowman BA, Otvos JD, Srinivasan SR, Berenson GS. Differences in the relation of obesity to serum triacylglycerol and VLDL subclass concentrations between black and white children: the Bogalusa Heart Study. Am J Clin Nutr. 2002 May;75(5):827-33. doi: 10.1093/ajcn/75.5.827. PMID 11976155
- [Background] Srinivasan SR, Myers L, Berenson GS. Distribution and correlates of non-high-density lipoprotein cholesterol in children: the Bogalusa Heart Study. Pediatrics. 2002 Sep;110(3):e29. doi: 10.1542/peds.110.3.e29. PMID 12205279
- [Background] Ellsworth DL, Coady SA, Chen W, Srinivasan SR, Elkasabany A, Gustat J, Boerwinkle E, Berenson GS. Influence of the beta2-adrenergic receptor Arg16Gly polymorphism on longitudinal changes in obesity from childhood through young adulthood in a biracial cohort: the Bogalusa Heart Study. Int J Obes Relat Metab Disord. 2002 Jul;26(7):928-37. doi: 10.1038/sj.ijo.0802020. PMID 12080445
- [Background] Tershakovec AM, Jawad AF, Stouffer NO, Elkasabany A, Srinivasan SR, Berenson GS. Persistent hypercholesterolemia is associated with the development of obesity among girls: the Bogalusa Heart Study. Am J Clin Nutr. 2002 Oct;76(4):730-5. doi: 10.1093/ajcn/76.4.730. PMID 12324284
- [Background] Urbina EM, Srinivasan SR, Tang R, Bond MG, Kieltyka L, Berenson GS; Bogalusa Heart Study. Impact of multiple coronary risk factors on the intima-media thickness of different segments of carotid artery in healthy young adults (The Bogalusa Heart Study). Am J Cardiol. 2002 Nov 1;90(9):953-8. doi: 10.1016/s0002-9149(02)02660-7. PMID 12398961
- [Background] Freedman DS, Khan LK, Serdula MK, Dietz WH, Srinivasan SR, Berenson GS. Relation of age at menarche to race, time period, and anthropometric dimensions: the Bogalusa Heart Study. Pediatrics. 2002 Oct;110(4):e43. doi: 10.1542/peds.110.4.e43. PMID 12359816
- [Background] Youssef AA, Valdez R, Elkasabany A, Srinivasan SR, Berenson GS. Time-course of adiposity and fasting insulin from childhood to young adulthood in offspring of parents with coronary artery disease: the Bogalusa Heart Study. Ann Epidemiol. 2002 Nov;12(8):553-9. doi: 10.1016/s1047-2797(01)00286-1. PMID 12495828
- [Background] Gustat J, Srinivasan SR, Elkasabany A, Berenson GS. Relation of self-rated measures of physical activity to multiple risk factors of insulin resistance syndrome in young adults: the Bogalusa Heart Study. J Clin Epidemiol. 2002 Oct;55(10):997-1006. doi: 10.1016/s0895-4356(02)00427-4. PMID 12464376
- [Background] Hoq S, Chen W, Srinivasan SR, Berenson GS. Childhood blood pressure predicts adult microalbuminuria in African Americans, but not in whites: the Bogalusa Heart Study. Am J Hypertens. 2002 Dec;15(12):1036-41. doi: 10.1016/s0895-7061(02)03066-2. PMID 12460698
- [Background] Freedman DS, Khan LK, Serdula MK, Dietz WH, Srinivasan SR, Berenson GS; Bogalusa heart study. The relation of menarcheal age to obesity in childhood and adulthood: the Bogalusa heart study. BMC Pediatr. 2003 Apr 30;3:3. doi: 10.1186/1471-2431-3-3. Epub 2003 Apr 30. PMID 12723990
- [Background] Li S, Chen W, Srinivasan SR, Boerwinkle E, Berenson GS; Bogalusa Heart Study. The peroxisome proliferator-activated receptor-gamma2 gene polymorphism (Pro12Ala) beneficially influences insulin resistance and its tracking from childhood to adulthood: the Bogalusa Heart Study. Diabetes. 2003 May;52(5):1265-9. doi: 10.2337/diabetes.52.5.1265. PMID 12716762
- [Background] Srinivasan SR, Frontini MG, Berenson GS; Bogalusa Heart Study. Longitudinal changes in risk variables of insulin resistance syndrome from childhood to young adulthood in offspring of parents with type 2 diabetes: the Bogalusa Heart Study. Metabolism. 2003 Apr;52(4):443-50; discussion 451-3. doi: 10.1053/meta.2003.50065. PMID 12701056
- [Background] Frontini MG, Srinivasan SR, Elkasabany A, Berenson GS. Awareness of hypertension and dyslipidemia in a semirural population of young adults: the Bogalusa Heart Study. Prev Med. 2003 Apr;36(4):398-402. doi: 10.1016/s0091-7435(02)00045-2. PMID 12649047
- [Background] Chen W, Srinivasan SR, Boerwinkle E, Berenson GS; Bogalusa Heart Study. Hepatic lipase promoter C-514T polymorphism influences serial changes in HDL cholesterol levels since childhood: the Bogalusa Heart Study. Atherosclerosis. 2003 Jul;169(1):175-82. doi: 10.1016/s0021-9150(03)00162-x. PMID 12860265
- [Background] Nicklas TA, Yang SJ, Baranowski T, Zakeri I, Berenson G. Eating patterns and obesity in children. The Bogalusa Heart Study. Am J Prev Med. 2003 Jul;25(1):9-16. doi: 10.1016/s0749-3797(03)00098-9. PMID 12818304
- [Background] Srinivasan SR, Li S, Chen W, Boerwinkle E, Berenson GS. R219K polymorphism of the ABCA1 gene and its modulation of the variations in serum high-density lipoprotein cholesterol and triglycerides related to age and adiposity in white versus black young adults. The Bogalusa heart study. Metabolism. 2003 Jul;52(7):930-4. doi: 10.1016/s0026-0495(03)00076-3. PMID 12870173
- [Background] Olshan AF, Li R, Pankow JS, Bray M, Tyroler HA, Chambless LE, Boerwinkle E, Pittman GS, Bell DA. Risk of atherosclerosis: interaction of smoking and glutathione S-transferase genes. Epidemiology. 2003 May;14(3):321-7. PMID 12859033
- [Background] Bhuiyan AR, Gustat J, Srinivasan SR, Berenson GS. Differences in body shape representations among young adults from a biracial (Black-White), semirural community: the Bogalusa Heart Study. Am J Epidemiol. 2003 Oct 15;158(8):792-7. doi: 10.1093/aje/kwg218. PMID 14561669
- [Background] Frontini MG, Srinivasan SR, Berenson GS. Longitudinal changes in risk variables underlying metabolic Syndrome X from childhood to young adulthood in female subjects with a history of early menarche: the Bogalusa Heart Study. Int J Obes Relat Metab Disord. 2003 Nov;27(11):1398-404. doi: 10.1038/sj.ijo.0802422. PMID 14574352
- [Background] Xin X, Srinivasan SR, Chen W, Boerwinkle E, Berenson GS. Interaction effect of Serine447Stop variant of the lipoprotein lipase gene and C-514T variant of the hepatic lipase gene on serum triglyceride levels in young adults: the Bogalusa Heart Study. Metabolism. 2003 Oct;52(10):1337-42. doi: 10.1016/s0026-0495(03)00280-4. PMID 14564687
- [Background] Kieltyka L, Urbina EM, Tang R, Bond MG, Srinivasan SR, Berenson GS. Framingham risk score is related to carotid artery intima-media thickness in both white and black young adults: the Bogalusa Heart Study. Atherosclerosis. 2003 Sep;170(1):125-30. doi: 10.1016/s0021-9150(03)00244-2. PMID 12957690
- [Background] Krishnan P, Balamurugan A, Urbina E, Srinivasan SR, Bond G, Tang R, Berenson GS. Cardiovascular risk profile of asymptomatic healthy young adults with increased carotid artery intima-media thickness: the Bogalusa Heart Study. J La State Med Soc. 2003 May-Jun;155(3):165-9. PMID 12873105
- [Background] Li S, Chen W, Srinivasan SR, Bond MG, Tang R, Urbina EM, Berenson GS. Childhood cardiovascular risk factors and carotid vascular changes in adulthood: the Bogalusa Heart Study. JAMA. 2003 Nov 5;290(17):2271-6. doi: 10.1001/jama.290.17.2271. PMID 14600185
- [Background] Li S, Chen W, Srinivasan SR, Berenson GS. Childhood blood pressure as a predictor of arterial stiffness in young adults: the bogalusa heart study. Hypertension. 2004 Mar;43(3):541-6. doi: 10.1161/01.HYP.0000115922.98155.23. Epub 2004 Jan 26. PMID 14744922
- [Background] Freedman DS, Khan LK, Serdula MK, Dietz WH, Srinivasan SR, Berenson GS. Inter-relationships among childhood BMI, childhood height, and adult obesity: the Bogalusa Heart Study. Int J Obes Relat Metab Disord. 2004 Jan;28(1):10-6. doi: 10.1038/sj.ijo.0802544. PMID 14652621
- [Background] Eisenmann JC. Secular trends in variables associated with the metabolic syndrome of North American children and adolescents: a review and synthesis. Am J Hum Biol. 2003 Nov-Dec;15(6):786-94. doi: 10.1002/ajhb.10214. PMID 14595870
- [Background] Freedman DS, Dietz WH, Tang R, Mensah GA, Bond MG, Urbina EM, Srinivasan S, Berenson GS. The relation of obesity throughout life to carotid intima-media thickness in adulthood: the Bogalusa Heart Study. Int J Obes Relat Metab Disord. 2004 Jan;28(1):159-66. doi: 10.1038/sj.ijo.0802515. PMID 14581934
- [Background] Nicklas TA, Morales M, Linares A, Yang SJ, Baranowski T, De Moor C, Berenson G. Children's meal patterns have changed over a 21-year period: the Bogalusa Heart Study. J Am Diet Assoc. 2004 May;104(5):753-61. doi: 10.1016/j.jada.2004.02.030. PMID 15127060
- [Background] Mzayek F, Sherwin R, Fonseca V, Valdez R, Srinivasan SR, Cruickshank JK, Berenson GS. Differential association of birth weight with cardiovascular risk variables in African-Americans and Whites: the Bogalusa heart study. Ann Epidemiol. 2004 Apr;14(4):258-64. doi: 10.1016/j.annepidem.2003.09.014. PMID 15066605
- [Background] Chen W, Li S, Cook NR, Rosner BA, Srinivasan SR, Boerwinkle E, Berenson GS. An autosomal genome scan for loci influencing longitudinal burden of body mass index from childhood to young adulthood in white sibships: The Bogalusa Heart Study. Int J Obes Relat Metab Disord. 2004 Apr;28(4):462-9. doi: 10.1038/sj.ijo.0802610. PMID 14993914
- [Background] Chen W, Srinivasan SR, Bond MG, Tang R, Urbina EM, Li S, Boerwinkle E, Berenson GS. Nitric oxide synthase gene polymorphism (G894T) influences arterial stiffness in adults: The Bogalusa Heart Study. Am J Hypertens. 2004 Jul;17(7):553-9. doi: 10.1016/j.amjhyper.2004.02.021. PMID 15233973
- [Background] Nicklas TA, Demory-Luce D, Yang SJ, Baranowski T, Zakeri I, Berenson G. Children's food consumption patterns have changed over two decades (1973-1994): The Bogalusa heart study. J Am Diet Assoc. 2004 Jul;104(7):1127-40. doi: 10.1016/j.jada.2004.04.029. PMID 15215772
- [Background] Yoo S, Nicklas T, Baranowski T, Zakeri IF, Yang SJ, Srinivasan SR, Berenson GS. Comparison of dietary intakes associated with metabolic syndrome risk factors in young adults: the Bogalusa Heart Study. Am J Clin Nutr. 2004 Oct;80(4):841-8. doi: 10.1093/ajcn/80.4.841. PMID 15447888
- [Background] Demory-Luce D, Morales M, Nicklas T, Baranowski T, Zakeri I, Berenson G. Changes in food group consumption patterns from childhood to young adulthood: the Bogalusa Heart Study. J Am Diet Assoc. 2004 Nov;104(11):1684-91. doi: 10.1016/j.jada.2004.07.026. PMID 15499355
- [Background] Alper AB Jr, Chen W, Yau L, Srinivasan SR, Berenson GS, Hamm LL. Childhood uric acid predicts adult blood pressure: the Bogalusa Heart Study. Hypertension. 2005 Jan;45(1):34-8. doi: 10.1161/01.HYP.0000150783.79172.bb. Epub 2004 Nov 29. PMID 15569853
- [Background] Frontini MG, Srinivasan SR, Xu J, Berenson GS. Low birth weight and longitudinal trends of cardiovascular risk factor variables from childhood to adolescence: the bogalusa heart study. BMC Pediatr. 2004 Nov 3;4(1):22. doi: 10.1186/1471-2431-4-22. PMID 15527498
- [Background] Stein JH, Douglas PS, Srinivasan SR, Bond MG, Tang R, Li S, Chen W, Berenson GS. Distribution and cross-sectional age-related increases of carotid artery intima-media thickness in young adults: the Bogalusa Heart Study. Stroke. 2004 Dec;35(12):2782-7. doi: 10.1161/01.STR.0000147719.27237.14. Epub 2004 Oct 28. PMID 15514185
- [Background] Srinivasan SR, Li S, Chen W, Tang R, Bond MG, Boerwinkle E, Berenson GS. Q192R polymorphism of the paraoxanase 1 gene and its association with serum lipoprotein variables and carotid artery intima-media thickness in young adults from a biracial community. The Bogalusa Heart Study. Atherosclerosis. 2004 Nov;177(1):167-74. doi: 10.1016/j.atherosclerosis.2004.06.013. PMID 15488880
- [Background] Chen W, Srinivasan SR, Li S, Boerwinkle E, Berenson GS. Gender-specific influence of NO synthase gene on blood pressure since childhood: the Bogalusa Heart Study. Hypertension. 2004 Nov;44(5):668-73. doi: 10.1161/01.HYP.0000145474.23750.2b. Epub 2004 Oct 4. PMID 15466663
- [Background] Hallman DM, Srinivasan SR, Chen W, Boerwinkle E, Berenson GS. The beta(2)-adrenergic receptor Arg16-gly polymorphism and interactions involving beta(2)- and beta(3)-adrenergic receptor polymorphisms are associated with variations in longitudinal serum lipid profiles: the Bogalusa Heart Study. Metabolism. 2004 Sep;53(9):1184-91. doi: 10.1016/j.metabol.2004.03.019. PMID 15334382
- [Background] Rajeshwari R, Nicklas TA, Yang SJ, Berenson GS. Longitudinal changes in intake and food sources of calcium from childhood to young adulthood: the bogalusa heart study. J Am Coll Nutr. 2004 Aug;23(4):341-50. doi: 10.1080/07315724.2004.10719377. PMID 15310738
- [Background] Urbina EM, Srinivasan SR, Kieltyka RL, Tang R, Bond MG, Chen W, Berenson GS. Correlates of carotid artery stiffness in young adults: The Bogalusa Heart Study. Atherosclerosis. 2004 Sep;176(1):157-64. doi: 10.1016/j.atherosclerosis.2004.04.023. PMID 15306189
- [Background] Katzmarzyk PT, Srinivasan SR, Chen W, Malina RM, Bouchard C, Berenson GS. Body mass index, waist circumference, and clustering of cardiovascular disease risk factors in a biracial sample of children and adolescents. Pediatrics. 2004 Aug;114(2):e198-205. doi: 10.1542/peds.114.2.e198. PMID 15286257
- [Background] Chen W, Srinivasan SR, Li S, Xu J, Berenson GS. Metabolic syndrome variables at low levels in childhood are beneficially associated with adulthood cardiovascular risk: the Bogalusa Heart Study. Diabetes Care. 2005 Jan;28(1):126-31. doi: 10.2337/diacare.28.1.126. PMID 15616245
- [Background] Cook NR, Rosner BA, Chen W, Srinivasan SR, Berenson GS. Using the area under the curve to reduce measurement error in predicting young adult blood pressure from childhood measures. Stat Med. 2004 Nov 30;23(22):3421-35. doi: 10.1002/sim.1921. PMID 15505884
- [Background] Rajeshwari R, Yang SJ, Nicklas TA, Berenson GS. Secular trends in children's sweetened-beverage consumption (1973 to 1994): the Bogalusa Heart Study. J Am Diet Assoc. 2005 Feb;105(2):208-14. doi: 10.1016/j.jada.2004.11.026. PMID 15668676
- [Background] Berenson GS, Srnivasan SR; Bogalusa Heart Study Group. Cardiovascular risk factors in youth with implications for aging: the Bogalusa Heart Study. Neurobiol Aging. 2005 Mar;26(3):303-7. doi: 10.1016/j.neurobiolaging.2004.05.009. PMID 15639307
- [Background] Freedman DS, Khan LK, Serdula MK, Dietz WH, Srinivasan SR, Berenson GS. The relation of childhood BMI to adult adiposity: the Bogalusa Heart Study. Pediatrics. 2005 Jan;115(1):22-7. doi: 10.1542/peds.2004-0220. PMID 15629977
- [Background] Paul TK, Srinivasan SR, Chen W, Li S, Bond MG, Tang R, Berenson GS. Impact of multiple cardiovascular risk factors on femoral artery intima-media thickness in asymptomatic young adults (the Bogalusa Heart Study). Am J Cardiol. 2005 Feb 15;95(4):469-73. doi: 10.1016/j.amjcard.2004.10.013. PMID 15695130
- [Background] Cruickshank JK, Mzayek F, Liu L, Kieltyka L, Sherwin R, Webber LS, Srinavasan SR, Berenson GS. Origins of the "black/white" difference in blood pressure: roles of birth weight, postnatal growth, early blood pressure, and adolescent body size: the Bogalusa heart study. Circulation. 2005 Apr 19;111(15):1932-7. doi: 10.1161/01.CIR.0000161960.78745.33. PMID 15837946
- [Background] Chen W, Li S, Srinivasan SR, Boerwinkle E, Berenson GS. Autosomal genome scan for loci linked to blood pressure levels and trends since childhood: the Bogalusa Heart Study. Hypertension. 2005 May;45(5):954-9. doi: 10.1161/01.HYP.0000161881.02361.11. Epub 2005 Apr 4. PMID 15809362
- [Background] Li H, Srinivasan SR, Chen W, Xu JH, Li S, Berenson GS. Vascular abnormalities in asymptomatic, healthy young adult smokers without other major cardiovascular risk factors: the Bogalusa Heart Study. Am J Hypertens. 2005 Mar;18(3):319-24. doi: 10.1016/j.amjhyper.2004.10.005. PMID 15797647
- [Background] Bhuiyan AR, Li S, Li H, Chen W, Srinivasan SR, Berenson GS. Distribution and correlates of arterial compliance measures in asymptomatic young adults: the Bogalusa Heart Study. Am J Hypertens. 2005 May;18(5 Pt 1):684-91. doi: 10.1016/j.amjhyper.2004.11.039. PMID 15882552
- [Background] Tzou WS, Douglas PS, Srinivasan SR, Chen W, Berenson G, Stein JH. Advanced lipoprotein testing does not improve identification of subclinical atherosclerosis in young adults: the Bogalusa Heart Study. Ann Intern Med. 2005 May 3;142(9):742-50. doi: 10.7326/0003-4819-142-9-200505030-00009. PMID 15867406
- [Background] Gardner JP, Li S, Srinivasan SR, Chen W, Kimura M, Lu X, Berenson GS, Aviv A. Rise in insulin resistance is associated with escalated telomere attrition. Circulation. 2005 May 3;111(17):2171-7. doi: 10.1161/01.CIR.0000163550.70487.0B. Epub 2005 Apr 25. PMID 15851602
- [Background] Janssen I, Katzmarzyk PT, Srinivasan SR, Chen W, Malina RM, Bouchard C, Berenson GS. Combined influence of body mass index and waist circumference on coronary artery disease risk factors among children and adolescents. Pediatrics. 2005 Jun;115(6):1623-30. doi: 10.1542/peds.2004-2588. PMID 15930225
- [Background] Urbina EM, Kieltkya L, Tsai J, Srinivasan SR, Berenson GS. Impact of multiple cardiovascular risk factors on brachial artery distensibility in young adults: the Bogalusa Heart Study. Am J Hypertens. 2005 Jun;18(6):767-71. doi: 10.1016/j.amjhyper.2004.12.017. PMID 15925733
- [Background] Tzou WS, Douglas PS, Srinivasan SR, Bond MG, Tang R, Chen W, Berenson GS, Stein JH. Increased subclinical atherosclerosis in young adults with metabolic syndrome: the Bogalusa Heart Study. J Am Coll Cardiol. 2005 Aug 2;46(3):457-63. doi: 10.1016/j.jacc.2005.04.046. PMID 16053958
- [Background] Patel DA, Li S, Chen W, Srinivasan SR, Boerwinkle E, Berenson GS; Bogalusa Heart Study. G-6A polymorphism of the angiotensinogen gene and its association with left ventricular mass in asymptomatic young adults from a biethnic community: the Bogalusa Heart Study. Am J Hypertens. 2005 Nov;18(11):1437-41. doi: 10.1016/j.amjhyper.2005.05.031. PMID 16280278
- [Background] Berenson GS. Obesity--a critical issue in preventive cardiology: the Bogalusa Heart Study. Prev Cardiol. 2005 Fall;8(4):234-41; quiz 242-3. doi: 10.1111/j.0197-3118.2005.04485.x. PMID 16230878
- [Background] Paul TK, Srinivasan SR, Wei C, Li S, Bhuiyan AR, Bond MG, Tang R, Berenson GS. Cardiovascular risk profile of asymptomatic healthy young adults with increased femoral artery intima-media thickness: The Bogalusa Heart Study. Am J Med Sci. 2005 Sep;330(3):105-10. doi: 10.1097/00000441-200509000-00001. PMID 16174993
- [Background] Deshmukh-Taskar P, Nicklas TA, Morales M, Yang SJ, Zakeri I, Berenson GS. Tracking of overweight status from childhood to young adulthood: the Bogalusa Heart Study. Eur J Clin Nutr. 2006 Jan;60(1):48-57. doi: 10.1038/sj.ejcn.1602266. PMID 16132057
- [Background] Ranganathan R, Nicklas TA, Yang SJ, Berenson GS. The nutritional impact of dairy product consumption on dietary intakes of adults (1995-1996): the Bogalusa Heart Study. J Am Diet Assoc. 2005 Sep;105(9):1391-400. doi: 10.1016/j.jada.2005.06.024. PMID 16129080
- [Background] Agirbasli M, Ciliv G, Cakir S, Srinivasan S, Berenson GS, Ozme S. Body mass index and lipid levels in children from Ankara, Turkey versus Bogalusa, Louisiana. Prev Med. 2005 Nov-Dec;41(5-6):843-5. doi: 10.1016/j.ypmed.2005.08.001. Epub 2005 Sep 16. PMID 16169068
- [Background] Li S, Chen W, Srinivasan SR, Boerwinkle E, Berenson GS. Influence of lipoprotein lipase gene Ser447Stop and beta1-adrenergic receptor gene Arg389Gly polymorphisms and their interaction on obesity from childhood to adulthood: the Bogalusa Heart Study. Int J Obes (Lond). 2006 Aug;30(8):1183-8. doi: 10.1038/sj.ijo.0803281. Epub 2006 Mar 14. PMID 16534528
- [Background] Bhuiyan AR, Srinivasan SR, Chen W, Paul TK, Berenson GS. Correlates of vascular structure and function measures in asymptomatic young adults: the Bogalusa Heart Study. Atherosclerosis. 2006 Nov;189(1):1-7. doi: 10.1016/j.atherosclerosis.2006.02.011. Epub 2006 Mar 29. PMID 16569409
- [Background] Chen W, Li S, Srinivasan SR, Boerwinkle E, Berenson GS. A genome scan for loci influencing levels and trends of lipoprotein lipid-related traits since childhood: The Bogalusa Heart Study. Atherosclerosis. 2007 Feb;190(2):248-55. doi: 10.1016/j.atherosclerosis.2006.03.006. Epub 2006 May 6. PMID 16678832
- [Background] Chen W, Srinivasan SR, Li S, Berenson GS. Different effects of atherogenic lipoproteins and blood pressure on arterial structure and function: the Bogalusa Heart Study. J Clin Hypertens (Greenwich). 2006 May;8(5):323-9. doi: 10.1111/j.1524-6175.2005.04875.x. PMID 16687940
- [Background] Patel DA, Srinivasan SR, Xu JH, Li S, Chen W, Berenson GS. Distribution and metabolic syndrome correlates of plasma C-reactive protein in biracial (black-white) younger adults: the Bogalusa Heart Study. Metabolism. 2006 Jun;55(6):699-705. doi: 10.1016/j.metabol.2005.07.015. PMID 16713426
- [Background] Kabir AA, Whelton PK, Khan MM, Gustat J, Chen W. Association of symptoms of depression and obesity with hypertension: the Bogalusa Heart Study. Am J Hypertens. 2006 Jun;19(6):639-45. doi: 10.1016/j.amjhyper.2005.10.026. PMID 16733239
- [Background] Srinivasan SR, Myers L, Berenson GS. Changes in metabolic syndrome variables since childhood in prehypertensive and hypertensive subjects: the Bogalusa Heart Study. Hypertension. 2006 Jul;48(1):33-9. doi: 10.1161/01.HYP.0000226410.11198.f4. Epub 2006 Jun 12. PMID 16769996
- [Background] Srinivasan SR, Frontini MG, Xu J, Berenson GS. Utility of childhood non-high-density lipoprotein cholesterol levels in predicting adult dyslipidemia and other cardiovascular risks: the Bogalusa Heart Study. Pediatrics. 2006 Jul;118(1):201-6. doi: 10.1542/peds.2005-1856. PMID 16818566
- [Background] Berenson G, Srinivasan S, Chen W, Li S, Patel D; Bogalusa Heart Study Group. Racial (black-white) contrasts of risk for hypertensive disease in youth have implications for preventive care: the Bogalusa Heart Study. Ethn Dis. 2006 Summer;16(3 Suppl 4):S4-2-9. PMID 16937775
- [Background] Li H, Srinivasan SR, Berenson GS. Comparison of the measures of pulsatile arterial function between asymptomatic younger adult smokers and former smokers: the Bogalusa Heart Study. Am J Hypertens. 2006 Sep;19(9):897-901. doi: 10.1016/j.amjhyper.2006.02.004. PMID 16942930
- [Background] Patel DA, Srinivasan SR, Xu JH, Chen W, Berenson GS. Adiponectin and its correlates of cardiovascular risk in young adults: the Bogalusa Heart Study. Metabolism. 2006 Nov;55(11):1551-7. doi: 10.1016/j.metabol.2006.06.028. PMID 17046560
- [Background] Haji SA, Ulusoy RE, Patel DA, Srinivasan SR, Chen W, Delafontaine P, Berenson GS. Predictors of left ventricular dilatation in young adults (from the Bogalusa Heart Study). Am J Cardiol. 2006 Nov 1;98(9):1234-7. doi: 10.1016/j.amjcard.2006.05.054. Epub 2006 Sep 7. PMID 17056336
- [Background] Li S, Chen W, Srinivasan SR, Tang R, Bond MG, Berenson GS. Race (black-white) and gender divergences in the relationship of childhood cardiovascular risk factors to carotid artery intima-media thickness in adulthood: the Bogalusa Heart Study. Atherosclerosis. 2007 Oct;194(2):421-5. doi: 10.1016/j.atherosclerosis.2006.08.026. Epub 2006 Nov 22. PMID 17123535
- [Background] Hallman DM, Srinivasan SR, Chen W, Boerwinkle E, Berenson GS. Longitudinal analysis of haplotypes and polymorphisms of the APOA5 and APOC3 genes associated with variation in serum triglyceride levels: the Bogalusa Heart Study. Metabolism. 2006 Dec;55(12):1574-81. doi: 10.1016/j.metabol.2006.07.018. PMID 17142127
- [Background] Freedman DS, Mei Z, Srinivasan SR, Berenson GS, Dietz WH. Cardiovascular risk factors and excess adiposity among overweight children and adolescents: the Bogalusa Heart Study. J Pediatr. 2007 Jan;150(1):12-17.e2. doi: 10.1016/j.jpeds.2006.08.042. PMID 17188605
- [Background] Brooks BM, Rajeshwari R, Nicklas TA, Yang SJ, Berenson GS. Association of calcium intake, dairy product consumption with overweight status in young adults (1995-1996): the Bogalusa Heart Study. J Am Coll Nutr. 2006 Dec;25(6):523-32. doi: 10.1080/07315724.2006.10719568. PMID 17229900
- [Background] Deshmukh-Taskar P, Nicklas TA, Yang SJ, Berenson GS. Does food group consumption vary by differences in socioeconomic, demographic, and lifestyle factors in young adults? The Bogalusa Heart Study. J Am Diet Assoc. 2007 Feb;107(2):223-34. doi: 10.1016/j.jada.2006.11.004. PMID 17258958
- [Background] Johnson HM, Douglas PS, Srinivasan SR, Bond MG, Tang R, Li S, Chen W, Berenson GS, Stein JH. Predictors of carotid intima-media thickness progression in young adults: the Bogalusa Heart Study. Stroke. 2007 Mar;38(3):900-5. doi: 10.1161/01.STR.0000258003.31194.0a. Epub 2007 Feb 1. PMID 17272779
- [Background] Patel DA, Srinivasan SR, Xu JH, Chen W, Berenson GS. Persistent elevation of liver function enzymes within the reference range is associated with increased cardiovascular risk in young adults: the Bogalusa Heart Study. Metabolism. 2007 Jun;56(6):792-8. doi: 10.1016/j.metabol.2007.01.010. PMID 17512312
- [Background] Mzayek F, Hassig S, Sherwin R, Hughes J, Chen W, Srinivasan S, Berenson G. The association of birth weight with developmental trends in blood pressure from childhood through mid-adulthood: the Bogalusa Heart study. Am J Epidemiol. 2007 Aug 15;166(4):413-20. doi: 10.1093/aje/kwm098. Epub 2007 May 24. PMID 17525085
- [Background] Chen W, Srinivasan SR, Li S, Xu J, Berenson GS. Clustering of long-term trends in metabolic syndrome variables from childhood to adulthood in Blacks and Whites: the Bogalusa Heart Study. Am J Epidemiol. 2007 Sep 1;166(5):527-33. doi: 10.1093/aje/kwm105. Epub 2007 Jun 14. PMID 17573336
- [Background] Frontini MG, Srinivasan SR, Xu JH, Tang R, Bond MG, Berenson G. Utility of non-high-density lipoprotein cholesterol versus other lipoprotein measures in detecting subclinical atherosclerosis in young adults (The Bogalusa Heart Study). Am J Cardiol. 2007 Jul 1;100(1):64-8. doi: 10.1016/j.amjcard.2007.01.071. Epub 2007 May 11. PMID 17599442
- [Background] Hallman DM, Srinivasan SR, Chen W, Boerwinkle E, Berenson GS. Relation of PCSK9 mutations to serum low-density lipoprotein cholesterol in childhood and adulthood (from The Bogalusa Heart Study). Am J Cardiol. 2007 Jul 1;100(1):69-72. doi: 10.1016/j.amjcard.2007.02.057. Epub 2007 May 11. PMID 17599443
- [Background] Freedman DS, Kahn HS, Mei Z, Grummer-Strawn LM, Dietz WH, Srinivasan SR, Berenson GS. Relation of body mass index and waist-to-height ratio to cardiovascular disease risk factors in children and adolescents: the Bogalusa Heart Study. Am J Clin Nutr. 2007 Jul;86(1):33-40. doi: 10.1093/ajcn/86.1.33. PMID 17616760
- [Background] Bhuiyan AR, Chen W, Srinivasan SR, Rice J, Mock N, Tang R, Bond MG, Boerwinkle E, Berenson GS. Influence of nitric oxide synthase gene polymorphism (G894T) on carotid artery intima-media thickness in adults: the Bogalusa Heart Study. J Am Soc Hypertens. 2007 Sep-Oct;1(5):362-8. doi: 10.1016/j.jash.2007.06.006. PMID 20409867
- [Background] Bhuiyan AR, Chen W, Srinivasan SR, Rice J, Mock N, Tang R, Bond MG, Boerwinkle E, Berenson GS. G-6A polymorphism of angiotensinogen gene modulates the effect of blood pressure on carotid intima-media thickness. The Bogalusa Heart Study. Am J Hypertens. 2007 Oct;20(10):1073-8. doi: 10.1016/j.amjhyper.2007.06.001. PMID 17903690
- [Background] Tzou WS, Douglas PS, Srinivasan SR, Bond MG, Tang R, Li S, Chen W, Berenson GS, Stein JH. Distribution and predictors of carotid intima-media thickness in young adults. Prev Cardiol. 2007 Fall;10(4):181-9. doi: 10.1111/j.1520-037x.2007.06450.x. PMID 17917514
- [Background] Ortega FB, Ruiz JR, Sjostrom M. Physical activity, overweight and central adiposity in Swedish children and adolescents: the European Youth Heart Study. Int J Behav Nutr Phys Act. 2007 Nov 19;4:61. doi: 10.1186/1479-5868-4-61. PMID 18021444
- [Background] Chen W, Srinivasan SR, Boerwinkle E, Berenson GS. Beta-adrenergic receptor genes are associated with arterial stiffness in black and white adults: the Bogalusa Heart Study. Am J Hypertens. 2007 Dec;20(12):1251-7. doi: 10.1016/j.amjhyper.2007.09.002. PMID 18047913
- [Background] Magnussen CG, Raitakari OT, Thomson R, Juonala M, Patel DA, Viikari JS, Marniemi J, Srinivasan SR, Berenson GS, Dwyer T, Venn A. Utility of currently recommended pediatric dyslipidemia classifications in predicting dyslipidemia in adulthood: evidence from the Childhood Determinants of Adult Health (CDAH) study, Cardiovascular Risk in Young Finns Study, and Bogalusa Heart Study. Circulation. 2008 Jan 1;117(1):32-42. doi: 10.1161/CIRCULATIONAHA.107.718981. Epub 2007 Dec 10. PMID 18071074
- [Background] Chen W, Srinivasan SR, Berenson GS. Path analysis of metabolic syndrome components in black versus white children, adolescents, and adults: the Bogalusa Heart Study. Ann Epidemiol. 2008 Feb;18(2):85-91. doi: 10.1016/j.annepidem.2007.07.090. PMID 18191760
- [Background] Freedman DS, Patel DA, Srinivasan SR, Chen W, Tang R, Bond MG, Berenson GS. The contribution of childhood obesity to adult carotid intima-media thickness: the Bogalusa Heart Study. Int J Obes (Lond). 2008 May;32(5):749-56. doi: 10.1038/sj.ijo.0803798. Epub 2008 Jan 29. PMID 18227845
- [Background] Nguyen QM, Srinivasan SR, Xu JH, Chen W, Berenson GS. Racial (black-white) divergence in the association between adiponectin and arterial stiffness in asymptomatic young adults: the Bogalusa heart study. Am J Hypertens. 2008 May;21(5):553-7. doi: 10.1038/ajh.2008.14. Epub 2008 Feb 21. PMID 18292758
- [Background] Berenson GS, Patel DA, Wang H, Srinivasan SR, Chen W. Pressure-heart rate product changes from childhood to adulthood in a biracial population - a crossover phenomenon: the Bogalusa Heart Study. J Am Soc Hypertens. 2008 Mar-Apr;2(2):80-7. doi: 10.1016/j.jash.2007.08.007. PMID 20409889
- [Background] Bhuiyan AR, Srinivasan SR, Chen W, Sultana A, Berenson GS. Association of serum bilirubin with pulsatile arterial function in asymptomatic young adults: the Bogalusa Heart Study. Metabolism. 2008 May;57(5):612-6. doi: 10.1016/j.metabol.2007.12.003. PMID 18442622
- [Background] Chen W, Srinivasan SR, Berenson GS. Differential impact of heart rate on arterial wall stiffness and thickness in young adults: The Bogalusa Heart Study. J Am Soc Hypertens. 2008 May-Jun;2(3):152-7. doi: 10.1016/j.jash.2007.10.008. PMID 20409897
- [Background] Frontini MG, Srinivasan SR, Xu J, Tang R, Bond MG, Berenson GS. Usefulness of childhood non-high density lipoprotein cholesterol levels versus other lipoprotein measures in predicting adult subclinical atherosclerosis: the Bogalusa Heart Study. Pediatrics. 2008 May;121(5):924-9. doi: 10.1542/peds.2007-1472. PMID 18450895
- [Background] Hunt SC, Chen W, Gardner JP, Kimura M, Srinivasan SR, Eckfeldt JH, Berenson GS, Aviv A. Leukocyte telomeres are longer in African Americans than in whites: the National Heart, Lung, and Blood Institute Family Heart Study and the Bogalusa Heart Study. Aging Cell. 2008 Aug;7(4):451-8. doi: 10.1111/j.1474-9726.2008.00397.x. Epub 2008 May 2. PMID 18462274
- [Background] Muntner P, Srinivasan S, Menke A, Patel DA, Chen W, Berenson G. Impact of childhood metabolic syndrome components on the risk of elevated uric acid in adulthood: the Bogalusa Heart Study. Am J Med Sci. 2008 May;335(5):332-7. doi: 10.1097/MAJ.0b013e31815574a4. PMID 18480647
- [Background] Toprak A, Wang H, Chen W, Paul T, Srinivasan S, Berenson G. Relation of childhood risk factors to left ventricular hypertrophy (eccentric or concentric) in relatively young adulthood (from the Bogalusa Heart Study). Am J Cardiol. 2008 Jun 1;101(11):1621-5. doi: 10.1016/j.amjcard.2008.01.045. Epub 2008 Apr 2. PMID 18489940
- [Background] Bhuiyan AR, Chen W, Srinivasan SR, Rice JC, Mock NB, Tang R, Gene Bond M, Boerwinkle E, Berenson GS. Interaction of G-protein beta3 subunit and nitric oxide synthase gene polymorphisms on carotid artery intima-media thickness in young adults: the Bogalusa Heart Study. Am J Hypertens. 2008 Aug;21(8):917-21. doi: 10.1038/ajh.2008.188. Epub 2008 Jun 12. PMID 18551105
- [Background] Chen W, Srinivasan SR, Xu J, Berenson GS. Effect of parental coronary artery disease on adverse effects of the metabolic syndrome and aging on carotid artery intima-media thickness (from the Bogalusa Heart Study). Am J Cardiol. 2008 Jul 15;102(2):180-3. doi: 10.1016/j.amjcard.2008.03.035. Epub 2008 May 28. PMID 18602517
- [Background] Nguyen QM, Srinivasan SR, Xu JH, Chen W, Berenson GS. Changes in risk variables of metabolic syndrome since childhood in pre-diabetic and type 2 diabetic subjects: the Bogalusa Heart Study. Diabetes Care. 2008 Oct;31(10):2044-9. doi: 10.2337/dc08-0898. Epub 2008 Jul 15. PMID 18628566
- [Background] Nguyen QM, Srinivasan SR, Xu JH, Chen W, Berenson GS. Distribution and cardiovascular risk correlates of hemoglobin A(1c) in nondiabetic younger adults: the Bogalusa Heart Study. Metabolism. 2008 Nov;57(11):1487-92. doi: 10.1016/j.metabol.2008.04.011. PMID 18940383
- [Background] Aviv A, Chen W, Gardner JP, Kimura M, Brimacombe M, Cao X, Srinivasan SR, Berenson GS. Leukocyte telomere dynamics: longitudinal findings among young adults in the Bogalusa Heart Study. Am J Epidemiol. 2009 Feb 1;169(3):323-9. doi: 10.1093/aje/kwn338. Epub 2008 Dec 4. PMID 19056834
- [Background] Chen W, Srinivasan SR, Berenson GS. Influence of birth weight on white blood cell count in biracial (black-white) children, adolescents, and young adults: the Bogalusa Heart Study. Am J Epidemiol. 2009 Jan 15;169(2):214-8. doi: 10.1093/aje/kwn341. Epub 2008 Dec 8. PMID 19064646
- [Background] Ruan L, Chen W, Srinivasan SR, Sun M, Wang H, Toprak A, Berenson GS. Correlates of common carotid artery lumen diameter in black and white younger adults: the Bogalusa Heart Study. Stroke. 2009 Mar;40(3):702-7. doi: 10.1161/STROKEAHA.108.531608. Epub 2009 Jan 8. PMID 19131651
- [Background] Toprak A, Wang H, Chen W, Paul T, Ruan L, Srinivasan S, Berenson G. Prehypertension and black-white contrasts in cardiovascular risk in young adults: Bogalusa Heart Study. J Hypertens. 2009 Feb;27(2):243-50. doi: 10.1097/hjh.0b013e32831aeee3. PMID 19226697
- [Background] Freedman DS, Dietz WH, Srinivasan SR, Berenson GS. Risk factors and adult body mass index among overweight children: the Bogalusa Heart Study. Pediatrics. 2009 Mar;123(3):750-7. doi: 10.1542/peds.2008-1284. PMID 19254998
- [Background] Magnussen CG, Venn A, Thomson R, Juonala M, Srinivasan SR, Viikari JS, Berenson GS, Dwyer T, Raitakari OT. The association of pediatric low- and high-density lipoprotein cholesterol dyslipidemia classifications and change in dyslipidemia status with carotid intima-media thickness in adulthood evidence from the cardiovascular risk in Young Finns study, the Bogalusa Heart study, and the CDAH (Childhood Determinants of Adult Health) study. J Am Coll Cardiol. 2009 Mar 10;53(10):860-9. doi: 10.1016/j.jacc.2008.09.061. PMID 19264243
- [Background] Toprak A, Reddy J, Chen W, Srinivasan S, Berenson G. Relation of pulse pressure and arterial stiffness to concentric left ventricular hypertrophy in young men (from the Bogalusa Heart Study). Am J Cardiol. 2009 Apr 1;103(7):978-84. doi: 10.1016/j.amjcard.2008.12.011. PMID 19327426
- [Background] Ruan L, Chen W, Srinivasan SR, Xu J, Sun M, Toprak A, Berenson GS. Relation of plasma homocysteine to arterial stiffness in black and white young adults (from the Bogalusa Heart Study). Am J Cardiol. 2009 Apr 1;103(7):985-8. doi: 10.1016/j.amjcard.2008.12.012. PMID 19327427
- [Background] Sisson SB, Katzmarzyk PT, Srinivasan SR, Chen W, Freedman DS, Bouchard C, Berenson GS. Ethnic differences in subcutaneous adiposity and waist girth in children and adolescents. Obesity (Silver Spring). 2009 Nov;17(11):2075-81. doi: 10.1038/oby.2009.132. Epub 2009 Apr 23. PMID 19390519
- [Background] Ruan L, Chen W, Srinivasan SR, Xu J, Toprak A, Berenson GS. Plasma homocysteine is adversely associated with glomerular filtration rate in asymptomatic black and white young adults: the Bogalusa heart study. Eur J Epidemiol. 2009;24(6):315-9. doi: 10.1007/s10654-009-9340-0. Epub 2009 Apr 25. PMID 19396552
- [Background] Freedman DS, Katzmarzyk PT, Dietz WH, Srinivasan SR, Berenson GS. Relation of body mass index and skinfold thicknesses to cardiovascular disease risk factors in children: the Bogalusa Heart Study. Am J Clin Nutr. 2009 Jul;90(1):210-6. doi: 10.3945/ajcn.2009.27525. Epub 2009 May 6. PMID 19420092
- [Background] Mzayek F, Sherwin R, Hughes J, Hassig S, Srinivasan S, Chen W, Berenson GS. The association of birth weight with arterial stiffness at mid-adulthood: the Bogalusa Heart Study. J Epidemiol Community Health. 2009 Sep;63(9):729-33. doi: 10.1136/jech.2008.084475. Epub 2009 May 7. PMID 19429574
- [Background] Mohindra NA, Nicklas TA, O'neil CE, Yang SJ, Berenson GS. Eating patterns and overweight status in young adults: the Bogalusa Heart Study. Int J Food Sci Nutr. 2009;60 Suppl 3(Suppl 3):14-25. doi: 10.1080/09637480802322095. Epub 2009 May 21. PMID 19462322
- [Background] Patel DA, Srinivasan SR, Chen W, Berenson GS. Influence of the metabolic syndrome versus the sum of its individual components on left ventricular geometry in young adults (from the Bogalusa Heart Study). Am J Cardiol. 2009 Jul 1;104(1):69-73. doi: 10.1016/j.amjcard.2009.02.063. PMID 19576323
- [Background] Nguyen QM, Srinivasan SR, Xu JH, Chen W, Berenson GS. Influence of childhood parental history of type 2 diabetes on the pre-diabetic and diabetic status in adulthood: the Bogalusa Heart Study. Eur J Epidemiol. 2009;24(9):537-9. doi: 10.1007/s10654-009-9372-5. Epub 2009 Jul 19. PMID 19618280
- [Background] Srinivasan SR, Wang R, Chen W, Wei CY, Xu J, Berenson GS. Utility of waist-to-height ratio in detecting central obesity and related adverse cardiovascular risk profile among normal weight younger adults (from the Bogalusa Heart Study). Am J Cardiol. 2009 Sep 1;104(5):721-4. doi: 10.1016/j.amjcard.2009.04.037. Epub 2009 Jun 24. PMID 19699351
- [Background] Deshmukh-Taskar PR, O'Neil CE, Nicklas TA, Yang SJ, Liu Y, Gustat J, Berenson GS. Dietary patterns associated with metabolic syndrome, sociodemographic and lifestyle factors in young adults: the Bogalusa Heart Study. Public Health Nutr. 2009 Dec;12(12):2493-503. doi: 10.1017/S1368980009991261. Epub 2009 Sep 11. PMID 19744354
- [Background] Bhuiyan AR, Chen W, Srinivasan SR, Azevedo MJ, Berenson GS. Relationship of low birth weight to pulsatile arterial function in asymptomatic younger adults: the Bogalusa Heart Study. Am J Hypertens. 2010 Feb;23(2):168-73. doi: 10.1038/ajh.2009.218. Epub 2009 Nov 26. PMID 19942864
- [Background] Muntner P, Arshad A, Morse SA, Patel DA, Manapatra PD, Reisin E, Aguilar EA, Chen W, Srinivasan S, Berenson GS. End-stage renal disease in young black males in a black-white population: longitudinal analysis of the Bogalusa Heart Study. BMC Nephrol. 2009 Dec 2;10:40. doi: 10.1186/1471-2369-10-40. PMID 19954521
- [Background] Kabir AA, Srinivasan SR, Sultana A, Chen W, Wei CY, Berenson GS. Association between depression and intima-media thickness of carotid bulb in asymptomatic young adults. Am J Med. 2009 Dec;122(12):1151.e1-8. doi: 10.1016/j.amjmed.2009.07.016. PMID 19958896
- [Background] Nguyen QM, Srinivasan SR, Xu JH, Chen W, Berenson GS. Distribution and cardiovascular risk correlates of plasma soluble intercellular adhesion molecule-1 levels in asymptomatic young adults from a biracial community: the Bogalusa Heart Study. Ann Epidemiol. 2010 Jan;20(1):53-9. doi: 10.1016/j.annepidem.2009.10.001. PMID 20006276
- [Background] Nguyen QM, Srinivasan SR, Xu JH, Chen W, Kieltyka L, Berenson GS. Utility of childhood glucose homeostasis variables in predicting adult diabetes and related cardiometabolic risk factors: the Bogalusa Heart Study. Diabetes Care. 2010 Mar;33(3):670-5. doi: 10.2337/dc09-1635. Epub 2009 Dec 15. PMID 20009096
- [Background] Berenson GS. Cardiovascular health promotion for children: a model for a Parish (County)-wide program (implementation and preliminary results). Prev Cardiol. 2010 Winter;13(1):23-8. doi: 10.1111/j.1751-7141.2009.00049.x. PMID 20021623
- [Background] Nguyen QM, Srinivasan SR, Xu JH, Chen W, Berenson GS. Fasting plasma glucose levels within the normoglycemic range in childhood as a predictor of prediabetes and type 2 diabetes in adulthood: the Bogalusa Heart Study. Arch Pediatr Adolesc Med. 2010 Feb;164(2):124-8. doi: 10.1001/archpediatrics.2009.268. PMID 20124140
- [Background] Camhi SM, Katzmarzyk PT, Broyles S, Srinivasan SR, Chen W, Bouchard C, Berenson GS. Predicting adult body mass index-specific metabolic risk from childhood. Metab Syndr Relat Disord. 2010 Apr;8(2):165-72. doi: 10.1089/met.2009.0063. PMID 20156071
- [Background] Toprak D, Toprak A, Chen W, Xu JH, Srinivasan S, Berenson GS. Adiposity in childhood is related to C-reactive protein and adiponectin in young adulthood: from the Bogalusa Heart Study. Obesity (Silver Spring). 2011 Jan;19(1):185-90. doi: 10.1038/oby.2010.75. Epub 2010 Apr 1. PMID 20360758
- [Background] Broyles S, Katzmarzyk PT, Srinivasan SR, Chen W, Bouchard C, Freedman DS, Berenson GS. The pediatric obesity epidemic continues unabated in Bogalusa, Louisiana. Pediatrics. 2010 May;125(5):900-5. doi: 10.1542/peds.2009-2748. Epub 2010 Apr 5. PMID 20368311
- [Background] Kobori H, Urushihara M, Xu JH, Berenson GS, Navar LG. Urinary angiotensinogen is correlated with blood pressure in men (Bogalusa Heart Study). J Hypertens. 2010 Jul;28(7):1422-8. doi: 10.1097/HJH.0b013e3283392673. PMID 20375906
- [Background] Freedman DS, Katzmarzyk PT, Dietz WH, Srinivasan SR, Berenson GS. The relation of BMI and skinfold thicknesses to risk factors among young and middle-aged adults: the Bogalusa Heart Study. Ann Hum Biol. 2010 Nov;37(6):726-37. doi: 10.3109/03014461003641849. Epub 2010 May 7. PMID 20450389
- [Background] Chen W, Srinivasan SR, Hallman DM, Berenson GS. The relationship between birthweight and longitudinal changes of blood pressure is modulated by beta-adrenergic receptor genes: the Bogalusa Heart Study. J Biomed Biotechnol. 2010;2010:543514. doi: 10.1155/2010/543514. Epub 2010 May 11. PMID 20467565
- [Background] Chen W, Srinivasan SR, Berenson GS. Amplification of the association between birthweight and blood pressure with age: the Bogalusa Heart Study. J Hypertens. 2010 Oct;28(10):2046-52. doi: 10.1097/HJH.0b013e32833cd31f. PMID 20616754
- [Background] Freedman DS, Wang YC, Dietz WH, Xu JH, Srinivasan SR, Berenson GS. Changes and variability in high levels of low-density lipoprotein cholesterol among children. Pediatrics. 2010 Aug;126(2):266-73. doi: 10.1542/peds.2009-3454. Epub 2010 Jul 19. PMID 20643721
- [Background] Chen W, Srinivasan SR, Ruan L, Mei H, Berenson GS. Adult hypertension is associated with blood pressure variability in childhood in blacks and whites: the bogalusa heart study. Am J Hypertens. 2011 Jan;24(1):77-82. doi: 10.1038/ajh.2010.176. Epub 2010 Aug 19. PMID 20725054
- [Background] Chen W, Srinivasan SR, Xu J, Berenson GS. Black-white divergence in the relation of white blood cell count to metabolic syndrome in preadolescents, adolescents, and young adults: the Bogalusa Heart Study. Diabetes Care. 2010 Nov;33(11):2474-6. doi: 10.2337/dc10-0619. Epub 2010 Aug 26. PMID 20798336
- [Background] d'Annunzio G, Russo C, Lorini R. Utility of childhood glucose homeostasis variables in predicting adult diabetes and related cardiometabolic risk factors: the Bogalusa Heart Study: comment on Nguyen et Al. Diabetes Care. 2010 Sep;33(9):e123; author reply e124. doi: 10.2337/dc10-0827. No abstract available. PMID 20805265
- [Background] Ruan L, Chen W, Srinivasan SR, Xu J, Toprak A, Berenson GS. Relation of serum phosphorus levels to carotid intima-media thickness in asymptomatic young adults (from the Bogalusa Heart Study). Am J Cardiol. 2010 Sep 15;106(6):793-7. doi: 10.1016/j.amjcard.2010.05.004. Epub 2010 Aug 2. PMID 20816119
- [Background] Smith EN, Chen W, Kahonen M, Kettunen J, Lehtimaki T, Peltonen L, Raitakari OT, Salem RM, Schork NJ, Shaw M, Srinivasan SR, Topol EJ, Viikari JS, Berenson GS, Murray SS. Longitudinal genome-wide association of cardiovascular disease risk factors in the Bogalusa heart study. PLoS Genet. 2010 Sep 9;6(9):e1001094. doi: 10.1371/journal.pgen.1001094. PMID 20838585
- [Background] Magnussen CG, Koskinen J, Chen W, Thomson R, Schmidt MD, Srinivasan SR, Kivimaki M, Mattsson N, Kahonen M, Laitinen T, Taittonen L, Ronnemaa T, Viikari JS, Berenson GS, Juonala M, Raitakari OT. Pediatric metabolic syndrome predicts adulthood metabolic syndrome, subclinical atherosclerosis, and type 2 diabetes mellitus but is no better than body mass index alone: the Bogalusa Heart Study and the Cardiovascular Risk in Young Finns Study. Circulation. 2010 Oct 19;122(16):1604-11. doi: 10.1161/CIRCULATIONAHA.110.940809. Epub 2010 Oct 4. PMID 20921439
- [Background] Mokha JS, Srinivasan SR, Dasmahapatra P, Fernandez C, Chen W, Xu J, Berenson GS. Utility of waist-to-height ratio in assessing the status of central obesity and related cardiometabolic risk profile among normal weight and overweight/obese children: the Bogalusa Heart Study. BMC Pediatr. 2010 Oct 11;10:73. doi: 10.1186/1471-2431-10-73. PMID 20937123
- [Background] Paul TK, Chen W, Srinivasan SR, Rice J, Toprak A, He J, Berenson GS. Framingham risk score is associated with femoral artery intima-media thickness in asymptomatic young adults (the Bogalusa heart study). Atherosclerosis. 2010 Dec;213(2):627-31. doi: 10.1016/j.atherosclerosis.2010.09.026. Epub 2010 Oct 20. PMID 20970137
- [Background] Freedman DS, Fulton JE, Dietz WH, Pan L, Nihiser AJ, Srinivasan SR, Berenson GS. The identification of children with adverse risk factor levels by body mass index cutoffs from 2 classification systems: the Bogalusa Heart Study. Am J Clin Nutr. 2010 Dec;92(6):1298-305. doi: 10.3945/ajcn.2010.29758. Epub 2010 Oct 27. PMID 20980492
- [Background] Juonala M, Magnussen CG, Venn A, Dwyer T, Burns TL, Davis PH, Chen W, Srinivasan SR, Daniels SR, Kahonen M, Laitinen T, Taittonen L, Berenson GS, Viikari JS, Raitakari OT. Influence of age on associations between childhood risk factors and carotid intima-media thickness in adulthood: the Cardiovascular Risk in Young Finns Study, the Childhood Determinants of Adult Health Study, the Bogalusa Heart Study, and the Muscatine Study for the International Childhood Cardiovascular Cohort (i3C) Consortium. Circulation. 2010 Dec 14;122(24):2514-20. doi: 10.1161/CIRCULATIONAHA.110.966465. Epub 2010 Nov 29. PMID 21126976
- [Background] Camhi SM, Katzmarzyk PT, Broyles ST, Srinivasan SR, Chen W, Bouchard C, Berenson GS. Subclinical atherosclerosis and metabolic risk: role of body mass index and waist circumference. Metab Syndr Relat Disord. 2011 Apr;9(2):119-25. doi: 10.1089/met.2010.0079. Epub 2010 Dec 6. PMID 21133775
- [Background] Nguyen QM, Toprak A, Xu JH, Srinivasan SR, Chen W, Berenson GS. Progression of segment-specific carotid artery intima-media thickness in young adults (from the Bogalusa Heart Study). Am J Cardiol. 2011 Jan;107(1):114-9. doi: 10.1016/j.amjcard.2010.08.054. PMID 21146698
- [Background] Chio SS, Urbina EM, Lapointe J, Tsai J, Berenson GS. Korotkoff sound versus oscillometric cuff sphygmomanometers: comparison between auscultatory and DynaPulse blood pressure measurements. J Am Soc Hypertens. 2011 Jan-Feb;5(1):12-20. doi: 10.1016/j.jash.2010.10.005. Epub 2011 Jan 26. PMID 21269907
- [Background] Kolovou GD, Bilianou H, Mikhailidis DP. Postprandial lipemia in children and adolescents. Curr Vasc Pharmacol. 2011 May;9(3):318-20. doi: 10.2174/157016111795495521. PMID 21314624
- [Background] Wang J, Chen W, Ruan L, Toprak A, Srinivasan SR, Berenson GS. Differential effect of elevated blood pressure on left ventricular geometry types in black and white young adults in a community (from the Bogalusa Heart Study). Am J Cardiol. 2011 Mar 1;107(5):717-22. doi: 10.1016/j.amjcard.2010.10.053. PMID 21316506
- [Background] Paul TK, Chen W, Srinivasan SR, He J, Berenson GS. Contrast of the impact of multiple cardiovascular risk factors on the femoral and carotid intima-media thickness in asymptomatic young adults: the Bogalusa Heart Study. Atherosclerosis. 2011 Jun;216(2):359-64. doi: 10.1016/j.atherosclerosis.2011.02.023. Epub 2011 Feb 18. PMID 21376319
- [Background] Bazzano LA, Belame SN, Patel DA, Chen W, Srinivasan S, McIlwain E, Berenson GS. Obesity and left ventricular dilatation in young adulthood: the Bogalusa Heart Study. Clin Cardiol. 2011 Mar;34(3):153-9. doi: 10.1002/clc.20896. PMID 21400542
- [Background] Bhuiyan AR, Srinivasan SR, Chen W, Azevedo MJ, Berenson GS. Influence of low birth weight on C-reactive protein in asymptomatic younger adults: the bogalusa heart study. BMC Res Notes. 2011 Mar 21;4:71. doi: 10.1186/1756-0500-4-71. PMID 21418637
- [Background] Dasmahapatra P, Srinivasan SR, Mokha J, Fernandez C, Chen W, Xu J, Berenson GS. Subclinical atherosclerotic changes related to chronic kidney disease in asymptomatic black and white young adults: the Bogalusa heart study. Ann Epidemiol. 2011 May;21(5):311-7. doi: 10.1016/j.annepidem.2011.01.007. PMID 21458723
- [Background] Patel DA, Srinivasan SR, Chen W, Berenson GS. Serum alanine aminotransferase and its association with metabolic syndrome in children: the bogalusa heart study. Metab Syndr Relat Disord. 2011 Jun;9(3):211-6. doi: 10.1089/met.2010.0086. Epub 2011 Apr 8. PMID 21476865
- [Background] Berenson GS, Chen W, Dasmahapatra P, Fernandez C, Giles T, Xu J, Srinivasan SR. Stimulus response of blood pressure in black and white young individuals helps explain racial divergence in adult cardiovascular disease: the Bogalusa Heart Study. J Am Soc Hypertens. 2011 Jul-Aug;5(4):230-8. doi: 10.1016/j.jash.2011.02.006. Epub 2011 Apr 13. PMID 21493177
- [Background] Paul TK, Chen W, Srinivasan SR, Toprak A, He J, Berenson GS. Gender divergence on the impact of multiple cardiovascular risk factors on the femoral artery intima-media thickness in asymptomatic young adults: the Bogalusa Heart Study. Am J Med Sci. 2012 Jan;343(1):40-5. doi: 10.1097/MAJ.0b013e31821da9c0. PMID 21681071
- [Background] Nguyen QM, Srinivasan SR, Xu JH, Chen W, Hassig S, Rice J, Berenson GS. Elevated liver function enzymes are related to the development of prediabetes and type 2 diabetes in younger adults: the Bogalusa Heart Study. Diabetes Care. 2011 Dec;34(12):2603-7. doi: 10.2337/dc11-0919. Epub 2011 Sep 27. PMID 21953798
- [Background] Hallman DM, Friedel VC, Eissa MA, Boerwinkle E, Huber JC Jr, Harrist RB, Srinivasan SR, Chen W, Dai S, Labarthe DR, Berenson GS. The association of variants in the FTO gene with longitudinal body mass index profiles in non-Hispanic white children and adolescents. Int J Obes (Lond). 2012 Jan;36(1):61-8. doi: 10.1038/ijo.2011.190. Epub 2011 Oct 11. PMID 21986706
- [Background] Berenson GS; Bogalusa Heart Study group. Health consequences of obesity. Pediatr Blood Cancer. 2012 Jan;58(1):117-21. doi: 10.1002/pbc.23373. PMID 22076834
- [Background] Kelley RE, Dasmahapatra P, Wang J, Chen W, Srinivasan SR, Fernandez C, Xu J, Martin-Schild S, Berenson GS. Prevalence of atherosclerotic plaque in young and middle-aged asymptomatic individuals: the Bogalusa heart study. South Med J. 2011 Dec;104(12):803-8. doi: 10.1097/SMJ.0b013e318236c35c. PMID 22089358
- [Background] Toprak A, Kandavar R, Toprak D, Chen W, Srinivasan S, Xu JH, Anwar A, Berenson GS. C-reactive protein is an independent predictor for carotid artery intima-media thickness progression in asymptomatic younger adults (from the Bogalusa Heart Study). BMC Cardiovasc Disord. 2011 Dec 30;11:78. doi: 10.1186/1471-2261-11-78. PMID 22208681
- [Background] Hernesniemi JA, Seppala I, Lyytikainen LP, Mononen N, Oksala N, Hutri-Kahonen N, Juonala M, Taittonen L, Smith EN, Schork NJ, Chen W, Srinivasan SR, Berenson GS, Murray SS, Laitinen T, Jula A, Kettunen J, Ripatti S, Laaksonen R, Viikari J, Kahonen M, Raitakari OT, Lehtimaki T. Genetic profiling using genome-wide significant coronary artery disease risk variants does not improve the prediction of subclinical atherosclerosis: the Cardiovascular Risk in Young Finns Study, the Bogalusa Heart Study and the Health 2000 Survey--a meta-analysis of three independent studies. PLoS One. 2012;7(1):e28931. doi: 10.1371/journal.pone.0028931. Epub 2012 Jan 25. PMID 22295058
- [Background] Nguyen QM, Xu JH, Chen W, Srinivasan SR, Berenson GS. Correlates of age onset of type 2 diabetes among relatively young black and white adults in a community: the Bogalusa Heart Study. Diabetes Care. 2012 Jun;35(6):1341-6. doi: 10.2337/dc11-1818. Epub 2012 Mar 7. PMID 22399694
- [Background] Freedman DS, Goodman A, Contreras OA, DasMahapatra P, Srinivasan SR, Berenson GS. Secular trends in BMI and blood pressure among children and adolescents: the Bogalusa Heart Study. Pediatrics. 2012 Jul;130(1):e159-66. doi: 10.1542/peds.2011-3302. Epub 2012 Jun 4. PMID 22665416
- [Background] Freedman DS, Blanck HM, Dietz WH, DasMahapatra P, Srinivasan SR, Berenson GS. Is the body adiposity index (hip circumference/height(1.5)) more strongly related to skinfold thicknesses and risk factor levels than is BMI? The Bogalusa Heart Study. Br J Nutr. 2013 Jan 28;109(2):338-45. doi: 10.1017/S0007114512000979. Epub 2012 Apr 13. PMID 22716994
- [Background] Harville EW, Srinivasan S, Chen W, Berenson GS. Is the metabolic syndrome a "small baby" syndrome?: the bogalusa heart study. Metab Syndr Relat Disord. 2012 Dec;10(6):413-21. doi: 10.1089/met.2012.0031. Epub 2012 Jul 25. PMID 22831273
- [Background] Mei H, Chen W, Mills K, He J, Srinivasan SR, Schork N, Murray S, Berenson GS. Influences of FTO gene on onset age of adult overweight. Hum Genet. 2012 Dec;131(12):1851-9. doi: 10.1007/s00439-012-1204-0. Epub 2012 Jul 29. PMID 22842737
- [Background] Magnussen CG, Koskinen J, Juonala M, Chen W, Srinivasan SR, Sabin MA, Thomson R, Schmidt MD, Nguyen QM, Xu JH, Skilton MR, Kahonen M, Laitinen T, Taittonen L, Lehtimaki T, Ronnemaa T, Viikari JS, Berenson GS, Raitakari OT. A diagnosis of the metabolic syndrome in youth that resolves by adult life is associated with a normalization of high carotid intima-media thickness and type 2 diabetes mellitus risk: the Bogalusa heart and cardiovascular risk in young Finns studies. J Am Coll Cardiol. 2012 Oct 23;60(17):1631-9. doi: 10.1016/j.jacc.2012.05.056. Epub 2012 Sep 26. PMID 23021330
- [Background] Li S, Chen W, Srinivasan SR, Xu J, Berenson GS. Relation of childhood obesity/cardiometabolic phenotypes to adult cardiometabolic profile: the Bogalusa Heart Study. Am J Epidemiol. 2012 Oct 1;176 Suppl 7(Suppl 7):S142-9. doi: 10.1093/aje/kws236. PMID 23035138
- [Background] Chen W, Srinivasan SR, Yao L, Li S, Dasmahapatra P, Fernandez C, Xu J, Berenson GS. Low birth weight is associated with higher blood pressure variability from childhood to young adulthood: the Bogalusa Heart Study. Am J Epidemiol. 2012 Oct 1;176 Suppl 7(Suppl 7):S99-105. doi: 10.1093/aje/kws298. PMID 23035149
- [Background] Vassy JL, Dasmahapatra P, Meigs JB, Schork NJ, Magnussen CG, Chen W, Raitakari OT, Pencina MJ, Jamal SM, Berenson GS, Goodman E. Genotype prediction of adult type 2 diabetes from adolescence in a multiracial population. Pediatrics. 2012 Nov;130(5):e1235-42. doi: 10.1542/peds.2012-1132. Epub 2012 Oct 15. PMID 23071215
- [Background] Sharma D, DasMahapatra P, Fernandez C, Chen W, Srinivasan SR, Xu J, Berenson GS. The association of c-reactive protein with arterial compliance in asymptomatic young adults: the Bogalusa heart study. J Hum Hypertens. 2013 Apr;27(4):256-60. doi: 10.1038/jhh.2012.34. Epub 2012 Nov 15. PMID 23151748
- [Background] Wineinger NE, Harper A, Libiger O, Srinivasan SR, Chen W, Berenson GS, Schork NJ. Genomic risk models improve prediction of longitudinal lipid levels in children and young adults. Front Genet. 2013 May 21;4:86. doi: 10.3389/fgene.2013.00086. eCollection 2013. PMID 23734161
- [Background] Oikonen M, Laitinen TT, Magnussen CG, Steinberger J, Sinaiko AR, Dwyer T, Venn A, Smith KJ, Hutri-Kahonen N, Pahkala K, Mikkila V, Prineas R, Viikari JS, Morrison JA, Woo JG, Chen W, Nicklas T, Srinivasan SR, Berenson G, Juonala M, Raitakari OT. Ideal cardiovascular health in young adult populations from the United States, Finland, and Australia and its association with cIMT: the International Childhood Cardiovascular Cohort Consortium. J Am Heart Assoc. 2013 Jun 19;2(3):e000244. doi: 10.1161/JAHA.113.000244. PMID 23782922
- [Background] Chester R, Sander G, Fernandez C, Chen W, Berenson G, Giles T. Women have significantly greater difference between central and peripheral arterial pressure compared with men: the Bogalusa Heart Study. J Am Soc Hypertens. 2013 Sep-Oct;7(5):379-85. doi: 10.1016/j.jash.2013.05.007. Epub 2013 Jul 12. PMID 23850194
- [Background] Scott-Van Zeeland AA, Bloss CS, Tewhey R, Bansal V, Torkamani A, Libiger O, Duvvuri V, Wineinger N, Galvez L, Darst BF, Smith EN, Carson A, Pham P, Phillips T, Villarasa N, Tisch R, Zhang G, Levy S, Murray S, Chen W, Srinivasan S, Berenson G, Brandt H, Crawford S, Crow S, Fichter MM, Halmi KA, Johnson C, Kaplan AS, La Via M, Mitchell JE, Strober M, Rotondo A, Treasure J, Woodside DB, Bulik CM, Keel P, Klump KL, Lilenfeld L, Plotnicov K, Topol EJ, Shih PB, Magistretti P, Bergen AW, Berrettini W, Kaye W, Schork NJ. Evidence for the role of EPHX2 gene variants in anorexia nervosa. Mol Psychiatry. 2014 Jun;19(6):724-32. doi: 10.1038/mp.2013.91. Epub 2013 Sep 3. PMID 23999524
- [Background] Rosini N, Machado MJ, Webster IZ, Moura SA, Cavalcante Lda S, da Silva EL. Simultaneous prediction of hyperglycemia and dyslipidemia in school children in Santa Catarina State, Brazil based on waist circumference measurement. Clin Biochem. 2013 Dec;46(18):1837-41. doi: 10.1016/j.clinbiochem.2013.08.015. Epub 2013 Sep 4. PMID 24012695
- [Background] Wallace M, Harville E, Theall K, Webber L, Chen W, Berenson G. Preconception biomarkers of allostatic load and racial disparities in adverse birth outcomes: the Bogalusa Heart Study. Paediatr Perinat Epidemiol. 2013 Nov;27(6):587-97. doi: 10.1111/ppe.12091. Epub 2013 Oct 10. PMID 24117472
- [Background] Salz I, DasMahapatra P, Fernandez C, Ratard R, Srinivasan SR, Xu JH, Chen W, Wright M, Berenson GS. Public health perspective on causes of death among relatively young adults in a biracial (Black-white) semi-rural Louisiana community and implications for prevention: the Bogalusa Heart Study. J La State Med Soc. 2013 Jul-Aug;165(4):194-200. No abstract available. PMID 24133781
- [Background] Freedman DS, Horlick M, Berenson GS. A comparison of the Slaughter skinfold-thickness equations and BMI in predicting body fatness and cardiovascular disease risk factor levels in children. Am J Clin Nutr. 2013 Dec;98(6):1417-24. doi: 10.3945/ajcn.113.065961. Epub 2013 Oct 23. PMID 24153344
- [Background] Wallace M, Harville E, Theall K, Webber L, Chen W, Berenson G. Neighborhood poverty, allostatic load, and birth outcomes in African American and white women: findings from the Bogalusa Heart Study. Health Place. 2013 Nov;24:260-6. doi: 10.1016/j.healthplace.2013.10.002. Epub 2013 Oct 12. PMID 24184350
- [Background] O'Neil CE, Nicklas TA, Liu Y, Berenson GS. Candy consumption in childhood is not predictive of weight, adiposity measures or cardiovascular risk factors in young adults: the Bogalusa Heart Study. J Hum Nutr Diet. 2015 Feb;28 Suppl 2(0 2):59-69. doi: 10.1111/jhn.12200. Epub 2013 Dec 30. PMID 24382141
- [Background] Li S, Chen W, Yun M, Fernandez C, Krousel-Wood M, Webber L, Srinivasan SR, Berenson GS. Sex and race (black-white) differences in the relationship of childhood risk factors to adulthood arterial stiffness: the Bogalusa Heart Study. Am J Med Sci. 2014 Aug;348(2):101-7. doi: 10.1097/MAJ.0000000000000264. PMID 24762753
- [Background] Li S, Yun M, Fernandez C, Xu J, Srinivasan SR, Chen W, Berenson GS. Cigarette smoking exacerbates the adverse effects of age and metabolic syndrome on subclinical atherosclerosis: the Bogalusa Heart Study. PLoS One. 2014 May 2;9(5):e96368. doi: 10.1371/journal.pone.0096368. eCollection 2014. PMID 24789040
- [Background] Lai CC, Sun D, Cen R, Wang J, Li S, Fernandez-Alonso C, Chen W, Srinivasan SR, Berenson GS. Impact of long-term burden of excessive adiposity and elevated blood pressure from childhood on adulthood left ventricular remodeling patterns: the Bogalusa Heart Study. J Am Coll Cardiol. 2014 Oct 14;64(15):1580-7. doi: 10.1016/j.jacc.2014.05.072. PMID 25301461
- [Background] Sun D, Li S, Zhang X, Fernandez C, Chen W, Srinivasan SR, Berenson GS. Uric acid is associated with metabolic syndrome in children and adults in a community: the Bogalusa Heart Study. PLoS One. 2014 Oct 24;9(10):e89696. doi: 10.1371/journal.pone.0089696. eCollection 2014. PMID 25343690
- [Background] Yun M, Li S, Sun D, Ge S, Lai CC, Fernandez C, Chen W, Srinivasan SR, Berenson GS. Tobacco smoking strengthens the association of elevated blood pressure with arterial stiffness: the Bogalusa Heart Study. J Hypertens. 2015 Feb;33(2):266-74. doi: 10.1097/HJH.0000000000000410. PMID 25380147
- [Background] Hu T, Yao L, Gustat J, Chen W, Webber L, Bazzano L. Which measures of adiposity predict subsequent left ventricular geometry? Evidence from the Bogalusa Heart Study. Nutr Metab Cardiovasc Dis. 2015 Mar;25(3):319-26. doi: 10.1016/j.numecd.2014.11.001. Epub 2014 Nov 17. PMID 25534865
- [Background] Li C, Chen W, Jiang F, Simino J, Srinivasan SR, Berenson GS, Mei H. Genetic association and gene-smoking interaction study of carotid intima-media thickness at five GWAS-indicated genes: the Bogalusa Heart Study. Gene. 2015 May 15;562(2):226-31. doi: 10.1016/j.gene.2015.02.078. Epub 2015 Mar 6. PMID 25746325
- [Background] Bhuiyan AR, Srinivasan SR, Chen W, Fernandez C, Xu JH, Berenson GS. Timing of menarche related to carotid artery intima-media thickness in black and white young adult women: the Bogalusa Heart Study. Ann Epidemiol. 2015 Jun;25(6):414-9. doi: 10.1016/j.annepidem.2015.02.001. Epub 2015 Feb 14. PMID 25840807
- [Background] Chen W, Yun M, Fernandez C, Li S, Sun D, Lai CC, Hua Y, Wang F, Zhang T, Srinivasan SR, Johnson CC, Berenson GS. Secondhand smoke exposure is associated with increased carotid artery intima-media thickness: the Bogalusa Heart Study. Atherosclerosis. 2015 Jun;240(2):374-9. doi: 10.1016/j.atherosclerosis.2015.04.002. Epub 2015 Apr 7. PMID 25875389
- [Background] Li S, Chen W, Sun D, Fernandez C, Li J, Kelly T, He J, Krousel-Wood M, Whelton PK. Variability and rapid increase in body mass index during childhood are associated with adult obesity. Int J Epidemiol. 2015 Dec;44(6):1943-50. doi: 10.1093/ije/dyv202. Epub 2015 Oct 8. PMID 26452389
- [Background] Zhang T, Zhang H, Li S, Li Y, Liu Y, Fernandez C, Harville E, Bazzano L, He J, Chen W. Impact of Adiposity on Incident Hypertension Is Modified by Insulin Resistance in Adults: Longitudinal Observation From the Bogalusa Heart Study. Hypertension. 2016 Jan;67(1):56-62. doi: 10.1161/HYPERTENSIONAHA.115.06509. Epub 2015 Nov 16. PMID 26573703
- [Background] Agirbasli M, Tanrikulu AM, Berenson GS. Metabolic Syndrome: Bridging the Gap from Childhood to Adulthood. Cardiovasc Ther. 2016 Feb;34(1):30-6. doi: 10.1111/1755-5922.12165. PMID 26588351
- [Background] Zhang H, Zhang T, Li S, Li Y, Hussain A, Fernandez C, Harville E, Bazzano LA, He J, Chen W. Long-term Impact of Childhood Adiposity on Adult Metabolic Syndrome Is Modified by Insulin Resistance: The Bogalusa Heart Study. Sci Rep. 2015 Dec 7;5:17885. doi: 10.1038/srep17885. PMID 26640243
- [Background] Bazzano LA, Hu T, Bertisch SM, Yao L, Harville EW, Gustat J, Chen W, Webber LS, Shu T, Redline S. Childhood obesity patterns and relation to middle-age sleep apnoea risk: the Bogalusa Heart Study. Pediatr Obes. 2016 Dec;11(6):535-542. doi: 10.1111/ijpo.12103. Epub 2016 Jan 19. PMID 26780975
- [Background] Das M, Sha J, Hidalgo B, Aslibekyan S, Do AN, Zhi D, Sun D, Zhang T, Li S, Chen W, Srinivasan SR, Tiwari HK, Absher D, Ordovas JM, Berenson GS, Arnett DK, Irvin MR. Association of DNA Methylation at CPT1A Locus with Metabolic Syndrome in the Genetics of Lipid Lowering Drugs and Diet Network (GOLDN) Study. PLoS One. 2016 Jan 25;11(1):e0145789. doi: 10.1371/journal.pone.0145789. eCollection 2016. PMID 26808626
- [Background] Jacobs MB, Harville EW, Kelly TN, Bazzano LA, Chen W. Maternal apolipoprotein E genotype as a potential risk factor for poor birth outcomes: The Bogalusa Heart Study. J Perinatol. 2016 Jun;36(6):432-8. doi: 10.1038/jp.2016.4. Epub 2016 Feb 18. PMID 26890557
- [Background] Chen W, Li S, Fernandez C, Sun D, Lai CC, Zhang T, Bazzano L, Urbina EM, Deng HW. Temporal Relationship Between Elevated Blood Pressure and Arterial Stiffening Among Middle-Aged Black and White Adults: The Bogalusa Heart Study. Am J Epidemiol. 2016 Apr 1;183(7):599-608. doi: 10.1093/aje/kwv274. Epub 2016 Mar 8. PMID 26960706
- [Background] Hu T, Guralnik JM, Yao L, Gustat J, Harville EW, Webber LS, Chen W, He J, Whelton PK, Bazzano LA. Postural hand tremor and incident hypertension in young to middle-aged adults: the Bogalusa heart study. J Hypertens. 2016 Jul;34(7):1273-8. doi: 10.1097/HJH.0000000000000963. PMID 27136316
- [Background] Li S, Xiong X, Harville E, Zhang T, Sun D, Fernandez C, Krousel-Wood M, Chen W, Whelton PK. Childhood Risk Factors and Pregnancy-Induced Hypertension: The Bogalusa Heart Study. Am J Hypertens. 2016 Oct;29(10):1206-11. doi: 10.1093/ajh/hpw057. Epub 2016 Jun 1. PMID 27251339
- [Background] Jacobs MB, Bazzano LA, Pridjian G, Harville EW. Childhood adiposity and fertility difficulties: the Bogalusa Heart Study. Pediatr Obes. 2017 Dec;12(6):477-484. doi: 10.1111/ijpo.12168. Epub 2016 Jun 28. PMID 27350648
- [Background] Zhang T, Zhang H, Li Y, Sun D, Li S, Fernandez C, Qi L, Harville E, Bazzano L, He J, Xue F, Chen W. Temporal Relationship Between Childhood Body Mass Index and Insulin and Its Impact on Adult Hypertension: The Bogalusa Heart Study. Hypertension. 2016 Sep;68(3):818-23. doi: 10.1161/HYPERTENSIONAHA.116.07991. Epub 2016 Jul 18. PMID 27432860
- [Background] Hua Y, Wang F, Zhang T, Zhang H, Chen W, Shen W, Fernandez C, Harville E, Bazzano L, He J, Li S. Relation of Birth Weight to Heart Rate in Childhood, Adolescence, and Adulthood (from the Bogalusa Heart Study). Am J Cardiol. 2016 Sep 15;118(6):828-832. doi: 10.1016/j.amjcard.2016.06.046. Epub 2016 Jun 28. PMID 27453510
- [Background] Pollock BD, Hu T, Chen W, Harville EW, Li S, Webber LS, Fonseca V, Bazzano LA. Utility of existing diabetes risk prediction tools for young black and white adults: Evidence from the Bogalusa Heart Study. J Diabetes Complications. 2017 Jan;31(1):86-93. doi: 10.1016/j.jdiacomp.2016.07.025. Epub 2016 Jul 27. PMID 27503406
- [Background] Kelly TN, Bazzano LA, Ajami NJ, He H, Zhao J, Petrosino JF, Correa A, He J. Gut Microbiome Associates With Lifetime Cardiovascular Disease Risk Profile Among Bogalusa Heart Study Participants. Circ Res. 2016 Sep 30;119(8):956-64. doi: 10.1161/CIRCRESAHA.116.309219. Epub 2016 Aug 9. PMID 27507222
- [Background] Mzayek F, Cruickshank JK, Amoah D, Srinivasan S, Chen W, Berenson GS. Birth weight was longitudinally associated with cardiometabolic risk markers in mid-adulthood. Ann Epidemiol. 2016 Sep;26(9):643-7. doi: 10.1016/j.annepidem.2016.07.013. Epub 2016 Aug 10. PMID 27664850
- [Background] Zhang T, Li Y, Zhang H, Sun D, Li S, Fernandez C, Harville E, Bazzano L, He J, Chen W. Insulin-sensitive adiposity is associated with a relatively lower risk of diabetes than insulin-resistant adiposity: the Bogalusa Heart Study. Endocrine. 2016 Oct;54(1):93-100. doi: 10.1007/s12020-016-0948-z. Epub 2016 Apr 8. PMID 27060004
- [Background] Harville EW, Jacobs MB, Qi L, Chen W, Bazzano LA. Multigenerational Cardiometabolic Risk as a Predictor of Birth Outcomes: The Bogalusa Heart Study. J Pediatr. 2017 Feb;181:154-162.e1. doi: 10.1016/j.jpeds.2016.10.031. Epub 2016 Nov 7. PMID 27832834
- [Background] Tanrikulu MA, Agirbasli M, Berenson G. Primordial Prevention of Cardiometabolic Risk in Childhood. Adv Exp Med Biol. 2017;956:489-496. doi: 10.1007/5584_2016_172. PMID 27864799
- [Background] Berenson GS, Srinivasan SR, Xu JH, Chen W. Adiposity and Cardiovascular Risk Factor Variables in Childhood Are Associated With Premature Death From Coronary Heart Disease in Adults: The Bogalusa Heart Study. Am J Med Sci. 2016 Nov;352(5):448-454. doi: 10.1016/j.amjms.2016.08.006. Epub 2016 Aug 11. PMID 27865291
- [Background] Fernandez C, Hsu R, Sander G, Hussain A, Barshop R, Li S, Shu T, Zhang T, Galazka P, Chen W, Bazzano L, Giles TD. Methodological evaluation of the noninvasive estimation of central systolic blood pressure in nontreated patients: the Bogalusa Heart Study. Blood Press Monit. 2017 Apr;22(2):95-100. doi: 10.1097/MBP.0000000000000224. PMID 27902495
- [Background] Harville EW, Chen W, Bazzano L, Oikonen M, Hutri-Kahonen N, Raitakari O. Indicators of fetal growth and adult liver enzymes: the Bogalusa Heart Study and the Cardiovascular Risk in Young Finns Study. J Dev Orig Health Dis. 2017 Apr;8(2):226-235. doi: 10.1017/S2040174416000635. Epub 2016 Dec 6. PMID 27919310
- [Background] Pollock BD, Chen W, Harville EW, Bazzano LA. Associations between Hunter Type A/B Personality and Cardiovascular Risk Factors from Adolescence through Young Adulthood. Int J Behav Med. 2017 Aug;24(4):593-601. doi: 10.1007/s12529-017-9636-5. PMID 28127708
- [Background] Aslibekyan S, Do AN, Xu H, Li S, Irvin MR, Zhi D, Tiwari HK, Absher DM, Shuldiner AR, Zhang T, Chen W, Tanner K, Hong C, Mitchell BD, Berenson G, Arnett DK. CPT1A methylation is associated with plasma adiponectin. Nutr Metab Cardiovasc Dis. 2017 Mar;27(3):225-233. doi: 10.1016/j.numecd.2016.11.004. Epub 2016 Nov 23. PMID 28139377
- [Background] Xi B, Zhang T, Li S, Harville E, Bazzano L, He J, Chen W. Can Pediatric Hypertension Criteria Be Simplified? A Prediction Analysis of Subclinical Cardiovascular Outcomes From the Bogalusa Heart Study. Hypertension. 2017 Apr;69(4):691-696. doi: 10.1161/HYPERTENSIONAHA.116.08782. Epub 2017 Feb 21. PMID 28223474
- [Background] Zhang T, Zhang H, Li Y, Li S, Fernandez C, Bazzano L, He J, Xue F, Chen W. Long-term Impact of Temporal Sequence from Childhood Obesity to Hyperinsulinemia on Adult Metabolic Syndrome and Diabetes: The Bogalusa Heart Study. Sci Rep. 2017 Feb 23;7:43422. doi: 10.1038/srep43422. PMID 28230104
- [Background] Zhang H, Zhang T, Li S, Guo Y, Shen W, Fernandez C, Harville E, Bazzano LA, Urbina EM, He J, Chen W. Long-Term Excessive Body Weight and Adult Left Ventricular Hypertrophy Are Linked Through Later-Life Body Size and Blood Pressure: The Bogalusa Heart Study. Circ Res. 2017 May 12;120(10):1614-1621. doi: 10.1161/CIRCRESAHA.116.310421. Epub 2017 Feb 23. PMID 28232594
- [Background] Pollock BD, Chen W, Harville EW, Shu T, Fonseca V, Mauvais-Jarvis F, Kelly TN, Bazzano LA. Differential sex effects of systolic blood pressure and low-density lipoprotein cholesterol on type 2 diabetes: Life course data from the Bogalusa Heart Study. J Diabetes. 2018 Jun;10(6):449-457. doi: 10.1111/1753-0407.12543. Epub 2017 Apr 6. PMID 28239958
- [Background] Shen W, Zhang T, Li S, Zhang H, Xi B, Shen H, Fernandez C, Bazzano L, He J, Chen W. Race and Sex Differences of Long-Term Blood Pressure Profiles From Childhood and Adult Hypertension: The Bogalusa Heart Study. Hypertension. 2017 Jul;70(1):66-74. doi: 10.1161/HYPERTENSIONAHA.117.09537. Epub 2017 May 22. PMID 28533330
- [Background] Cicero AFG, Fogacci F, Borghi C. Letter by Cicero et al Regarding Article, "Long-Term Excessive Body Weight and Adult Left Ventricular Hypertrophy Are Linked Through Later-Life Body Size and Blood Pressure: The Bogalusa Heart Study". Circ Res. 2017 May 26;120(11):e50. doi: 10.1161/CIRCRESAHA.117.311186. No abstract available. PMID 28546362
- [Background] Seyednasrollah F, Makela J, Pitkanen N, Juonala M, Hutri-Kahonen N, Lehtimaki T, Viikari J, Kelly T, Li C, Bazzano L, Elo LL, Raitakari OT. Prediction of Adulthood Obesity Using Genetic and Childhood Clinical Risk Factors in the Cardiovascular Risk in Young Finns Study. Circ Cardiovasc Genet. 2017 Jun;10(3):e001554. doi: 10.1161/CIRCGENETICS.116.001554. PMID 28620069
- [Background] Sun D, Wang T, Heianza Y, Lv J, Han L, Rabito F, Kelly T, Li S, He J, Bazzano L, Chen W, Qi L. A History of Asthma From Childhood and Left Ventricular Mass in Asymptomatic Young Adults: The Bogalusa Heart Study. JACC Heart Fail. 2017 Jul;5(7):497-504. doi: 10.1016/j.jchf.2017.03.009. Epub 2017 Jun 26. PMID 28662937
- [Background] Wang F, Hua Y, Whelton PK, Zhang T, Fernandez CA, Zhang H, Bazzano L, He J, Chen W, Li S. Relationship Between Birth Weight and the Double Product in Childhood, Adolescence, and Adulthood (from the Bogalusa Heart Study). Am J Cardiol. 2017 Sep 15;120(6):1016-1019. doi: 10.1016/j.amjcard.2017.06.037. Epub 2017 Jun 28. PMID 28739035
- [Background] Wallace M, Bazzano L, Chen W, Harville E. Maternal childhood cardiometabolic risk factors and pregnancy complications. Ann Epidemiol. 2017 Jul;27(7):429-434. doi: 10.1016/j.annepidem.2017.06.002. Epub 2017 Jun 29. PMID 28789774
- [Background] Freedman DS, Berenson GS. Tracking of BMI z Scores for Severe Obesity. Pediatrics. 2017 Sep;140(3):e20171072. doi: 10.1542/peds.2017-1072. Epub 2017 Aug 22. PMID 28830920
- [Background] Koskinen J, Magnussen CG, Sinaiko A, Woo J, Urbina E, Jacobs DR Jr, Steinberger J, Prineas R, Sabin MA, Burns T, Berenson G, Bazzano L, Venn A, Viikari JSA, Hutri-Kahonen N, Raitakari O, Dwyer T, Juonala M. Childhood Age and Associations Between Childhood Metabolic Syndrome and Adult Risk for Metabolic Syndrome, Type 2 Diabetes Mellitus and Carotid Intima Media Thickness: The International Childhood Cardiovascular Cohort Consortium. J Am Heart Assoc. 2017 Aug 16;6(8):e005632. doi: 10.1161/JAHA.117.005632. PMID 28862940
- [Background] Chen BH, Carty CL, Kimura M, Kark JD, Chen W, Li S, Zhang T, Kooperberg C, Levy D, Assimes T, Absher D, Horvath S, Reiner AP, Aviv A. Leukocyte telomere length, T cell composition and DNA methylation age. Aging (Albany NY). 2017 Sep 20;9(9):1983-1995. doi: 10.18632/aging.101293. PMID 28930701
- [Background] Koskinen J, Juonala M, Dwyer T, Venn A, Thomson R, Bazzano L, Berenson GS, Sabin MA, Burns TL, Viikari JSA, Woo JG, Urbina EM, Prineas R, Hutri-Kahonen N, Sinaiko A, Jacobs D, Steinberger J, Daniels S, Raitakari OT, Magnussen CG. Impact of Lipid Measurements in Youth in Addition to Conventional Clinic-Based Risk Factors on Predicting Preclinical Atherosclerosis in Adulthood: International Childhood Cardiovascular Cohort Consortium. Circulation. 2018 Mar 20;137(12):1246-1255. doi: 10.1161/CIRCULATIONAHA.117.029726. Epub 2017 Nov 23. PMID 29170152
- [Background] Du Y, Zhang T, Sun D, Li C, Bazzano L, Qi L, Krousel-Wood M, He J, Whelton PK, Chen W, Li S. Effect of Serum Adiponectin Levels on the Association Between Childhood Body Mass Index and Adulthood Carotid Intima-Media Thickness. Am J Cardiol. 2018 Mar 1;121(5):579-583. doi: 10.1016/j.amjcard.2017.11.029. Epub 2017 Dec 12. PMID 29329827
- [Background] Wallace ME, Bazzano L, Zhang C, Harville E. Fasting glucose concentrations and associations with reproductive history over 40 years of follow-up. Gynecol Endocrinol. 2018 Aug;34(8):724-727. doi: 10.1080/09513590.2018.1431771. Epub 2018 Jan 24. PMID 29366358
- [Background] Pollock BD, Harville EW, Mills KT, Tang W, Chen W, Bazzano LA. Cardiovascular Risk and the American Dream: Life Course Observations From the BHS (Bogalusa Heart Study). J Am Heart Assoc. 2018 Feb 6;7(3):e007693. doi: 10.1161/JAHA.117.007693. PMID 29432134
- [Background] Harville EW, Jacobs M, Shu T, Breckner D, Wallace M. Feasibility of Linking Long-Term Cardiovascular Cohort Data to Offspring Birth Records: The Bogalusa Heart Study. Matern Child Health J. 2018 Jun;22(6):858-865. doi: 10.1007/s10995-018-2460-y. PMID 29435783
- [Background] Li Y, Zhang T, Han T, Li S, Bazzano L, He J, Chen W. Impact of cigarette smoking on the relationship between body mass index and insulin: Longitudinal observation from the Bogalusa Heart Study. Diabetes Obes Metab. 2018 Jul;20(7):1578-1584. doi: 10.1111/dom.13259. Epub 2018 Mar 11. PMID 29446554
- [Background] Harville EW, Chen W, Guralnik J, Bazzano LA. Reproductive history and physical functioning in midlife: The Bogalusa Heart Study. Maturitas. 2018 Mar;109:26-31. doi: 10.1016/j.maturitas.2017.12.006. Epub 2017 Dec 8. PMID 29452778
- [Background] Wang LX, Filipp SL, Urbina EM, Gurka MJ, DeBoer MD. Longitudinal Associations of Metabolic Syndrome Severity Between Childhood and Young Adulthood: The Bogalusa Heart Study. Metab Syndr Relat Disord. 2018 Jun;16(5):208-214. doi: 10.1089/met.2017.0160. Epub 2018 Mar 27. PMID 29584578
- [Background] Sun D, Li X, Heianza Y, Nisa H, Shang X, Rabito F, Kelly T, Harville E, Li S, He J, Bazzano L, Chen W, Qi L. History of Asthma From Childhood and Arterial Stiffness in Asymptomatic Young Adults: The Bogalusa Heart Study. Hypertension. 2018 May;71(5):928-936. doi: 10.1161/HYPERTENSIONAHA.118.10916. PMID 29632104